Official Title: MULTICENTER, INTERNATIONAL, DOUBLE-BLIND, TWO-ARM,

RANDOMIZED, PLACEBO-CONTROLLED PHASE II TRIAL OF

PIRFENIDONE IN PATIENTS WITH UNCLASSIFIABLE

PROGRESSIVE FIBROSING ILD

NCT Number: NCT03099187

**Document Date:** SAP Version 3: 20-July-2020

#### STATISTICAL ANALYSIS PLAN

TITLE: MULTICENTER, INTERNATIONAL, DOUBLE-

BLIND, TWO-ARM, RANDOMIZED, PLACEBO-CONTROLLED PHASE II TRIAL OF PIRFENIDONE

IN PATIENTS WITH UNCLASSIFIABLE

**PROGRESSIVE FIBROSING ILD** 

PROTOCOL NUMBER: MA39189

STUDY DRUG: Pirfenidone (RO0220912)

VERSION NUMBER: Version 3.0 17-July-2020

IND NUMBER: 67284

**PLAN PREPARED BY:** 

**Eudract Number:** 2016-002744-17

SPONSOR: F. Hoffmann-La Roche Ltd

(Clinipace) (Clinipace)

(F. Hoffmann-La Roche Ltd)

**DATE FINAL:** 17 July 2020

Date and Time(UTC) Reason for Signing Name

20-Jul-2020 08:57:11 Company Signatory

# STATISTICAL ANALYSIS PLAN AMENDMENT RATIONALE

The following changes were made compared to the first version of the SAP:

| | | | <u> </u> |
|---|---|---|---|
| Version | Date | Change number | Change description |
| 2 | 08-Oct-2018 | 1 | Clarification related to the aim and timeline of the primary analysis and final analysis of the study are included under section Outcome Measures. |
| 2 | 08-Oct-2018 | 2 | Week 28 is included in all descriptive efficacy tables. |
| 2 | 08-Oct-2018 | 3 | The safety follow-up period definition is changed as stated in section On-treatment Assessments (12-Month Safety Follow-up Period). |
| 2 | 08-Oct-2018 | 4 | Disposition is updated in section <u>Patient Disposition</u> . |
| 2 | 08-Oct-2018 | 5 | Details were added in order to analyze valid daily spirometry data in section <u>Demographic and Baseline Characteristics</u> . |
| 2 | 08-Oct-2018 | 6 | Additional analyses needed in the safety follow-up period based on safety follow-up population are presented under section <u>Safety Follow-up analyses</u> . |
| 2 | 08-Oct-2018 | 7 | Safety follow-up visits were included under section <u>Visit Windows</u> . |
| 2 | 08-Oct-2018 | 8 | Listings of stratification factors, separated types of adverse events and pregnancy data were removed from the corresponding sections. |
| 3 | 18-Jun-2020 | 9 | Categorical change of 5% and 10% for home FVC measurements deleted because of implausible data collected |
| 3 | 18-Jun-2020 | 10 | Restrict analysis of oxygen requirements to patients who had oxygen requirements |
| 3 | 18-Jun-2020 | 11 | Add information about sensitivity analyses performed for home FVC measurements in section Sensitivity Analyses |
| 3 | 18-Jun-2020 | 12 | Add correlation analysis for home FVC and site FVC measurements (Additional analyses after FDA feedback), see <a href="Exploratory Efficacy Endpoints">Exploratory Efficacy Endpoints</a> |
| 3 | 18-Jun-2020 | 13 | Mixed model analysis added for home spirometry and site spirometry as sensitivity analysis in section Sensitivity Analyses |

Pirfenidone — F. Hoffmann-La Roche Ltd

| 3 | 18-Jun-2020 | 14 | Subgroup analysis for biopsy taken before randomization (yes/no) added |
|---|---|---|---|
| 3 | 18-Jun-2020 | 15 | Tipping point analysis added for various assumptions to impute missing values in section <u>Sensitivity Analyses for missing data</u> |
| 3 | 18-Jun-2020 | 16 | Safety tables added to compare study data with phase III studies in section Adverse events |

Pirfenidone — F. Hoffmann-La Roche Ltd

## **TABLE OF CONTENTS**

| 1. | BACKGRO | UND | 11 |
|---|---|---|---|
| 2. | STUDY DE | SIGN | 11 |
| | 2.1 | Protocol Synopsis | 12 |
| | 2.2 | Outcome Measures | 12 |
| | 2.2.1 | Primary Efficacy Outcome Measures | 13 |
| | 2.2.2 | Secondary Efficacy Outcome Measures | 13 |
| | 2.2.3 | Exploratory Efficacy Outcome Measures | 14 |
| | 2.2.4 | Safety Outcome Measures | 14 |
| | 2.3 | Determination of Sample Size | 14 |
| | 2.4 | Interim Analysis | 15 |
| 3. | STUDY CO | NDUCT | 15 |
| | 3.1 | Randomization, BLINDING AND UNBLINDING PROCEDURES | 15 |
| | 3.2 | Independent Review Facility | 15 |
| | 3.3 | Data Monitoring | 16 |
| 4. | STATISTIC | AL METHODS | 16 |
| | 4.1 | Analysis Populations | 16 |
| | 4.1.1 | Intent-to-treat Population | 16 |
| | 4.1.2 | Per Protocol Population | 16 |
| | 4.1.3 | Safety Population | 16 |
| | 4.1.4 | Safety Follow-up Population | 17 |
| | 4.2 | Trial Periods, Observation and analysis times | 17 |
| | 4.2.1 | Study Days | 17 |
| | 4.2.2 | Baseline and Screening Observations | 18 |
| | 4.2.3<br>(Double-b | On-treatment Assessments for Efficacy Analyses plind Treatment Period) | 18 |
| | 4.2.4<br>(Double-b | On-treatment Assessments for Safety Analyses blind Treatment Period) | 18 |

Pirfenidone — F. Hoffmann-La Roche Ltd

| 4.2 | 2.5 | On-treatment Assessments (12-Month Safety | |
|---|---|---|---|
| Fo | llow-up I | Period) | 18 |
| 4.2 | 2.6 | Cut-off points | 19 |
| 4.3 | | Analysis of Treatment arm Comparability | 19 |
| 4.4 | | Analysis of Study Conduct | 19 |
| 4.4 | 4.1 | Patient Disposition | 19 |
| 4.4 | 4.2 | Major Protocol Deviations | 21 |
| 4.4 | 4.3 | Demographic and Baseline Characteristics | 21 |
| 4.4 | 4.4 | Previous and Concomitant Medication | 24 |
| 4.4 | 4.5 | Daily Spirometry (Handheld Device) | 25 |
| 4.4 | 4.6 | Compliance | 25 |
| 4.5 | | Efficacy Analysis | 25 |
| 4. | 5.1 | Primary Efficacy Endpoints | 26 |
| 4. | 5.2 | Reassessment of quality of home spirometry | 27 |
| 4. | 5.3 | Secondary Efficacy Endpoints | 27 |
| 4. | 5.4 | Exploratory Efficacy Endpoints | 30 |
| 4. | 5.5 | Analyses of Patient-Reported Outcomes | 31 |
| 4. | 5.6 | Sensitivity Analyses | 33 |
| 4. | 5.7 | Subgroup Analyses | 34 |
| 4. | 5.8 | Sensitivity Analyses for missing data | 34 |
| | 4.5.8.1 | Fixed missing imputation based on Placebo | 0.4 |
| | | tion | 34 |
| | | Fixed missing imputation between Q1 and Q3 of distribution | 35 |
| | 4.5.8.3 | Tipping point analysis with shifts | 36 |
| 4.6 | | Safety Analyses | 37 |
| 4.0 | 6.1 | Exposure of Study Medication | 38 |
| | 4.6.1.1 | Treatment duration | 38 |
| | 4.6.1.2 | Doses and Dose modifications or interruptions | 38 |
| 11 | 6.2 | Adverse Events | 30 |

Pirfenidone — F. Hoffmann-La Roche Ltd

| 4.6.3 | Deaths | 42 |
|------------|---------------------------|----|
| 4.6.4 | Laboratory Data | 43 |
| 4.6.5 | Vital Signs | 44 |
| 4.6.6 | ECG | 44 |
| 4.7 | Safety Follow-up analyses | 44 |
| 4.8 | Missing Data | 45 |
| 4.9 | Visit Windows | 47 |
| 4.10 | Interim Analyses | 48 |
| 4.11 | Biomarker Analyses | 48 |
| REFERENCES | | 50 |

Pirfenidone — F. Hoffmann-La Roche Ltd

## LIST OF TABLES

| Table 1 | Definition of Baseline and Screening Observations | 18 |
|------------|---------------------------------------------------|----|
| Table 2 | Visit Windows | 47 |
| | LIST OF APPENDICES | |
| APPENDIX 1 | PROTOCOL SYNOPSIS | 51 |
| APPENDIX 2 | SCHEDULE OF ASSESSMENTS | 59 |
| APPENDIX 3 | PRO QUESTIONNAIRES | 67 |

Pirfenidone — F. Hoffmann-La Roche Ltd

## **LIST OF ABBREVIATIONS**

| Abbreviation | Definition |
|--------------|----------------------------------------------------------|
| 6MWD | 6-minute walk distance |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| AST | aspartate aminotransferase |
| BID | two times daily |
| BTPS | body temperature and pressure saturated with water vapor |
| BP | blood pressure |
| BUN | blood urea nitrogen |
| CAPACITY | Clinical Studies Assessing Pirfenidone in idiopathic |
| | pulmonary fibrosis: Research of Efficacy and Safety |
| | Outcomes |
| cHP | chronic hypersensitivity pneumonitis |
| CI | confidence interval |
| CRO | contract research organization |
| CSP | clinical study protocol |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTD | connective tissue disease |
| CYP | cytochrome P450 |
| DLco | diffusing capacity of the lung for carbon monoxide |
| DNA | deoxyribonucleic acid |
| DSMB | Data and Safety Monitoring Board |
| EC | Ethics Committee |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| EEA | European Economic Area |
| ERA | endothelin receptor antagonist |
| FDA | Food and Drug Administration |
| FEV1 | forced expiratory volume in 1 second |
| FVC | forced vital capacity |
| GCP | Good Clinical Practice |
| GERD | gastroesophageal reflux disease |
| HIPAA | Health Insurance Portability and Accountability Act |
| HRCT | high-resolution computed tomography |
| ICH | International Conference on Harmonisation |
| iDMC | independent Data Monitoring Committee |
| IL | interleukin |

Pirfenidone — F. Hoffmann-La Roche Ltd

| ILD | interstitial lung disease |
|--------|---------------------------------------------------------------|
| IMP | investigational medicinal product |
| IND | · |
| IPAF | investigational New Drug |
| | interstitial pneumonia with autoimmune features |
| IPF | idiopathic pulmonary fibrosis<br>Institutional Review Board |
| IRB | |
| ITT | intent-to-treat |
| IxRS | interactive voice or web-based response system |
| LDH | lactate dehydrogenase |
| LFT | liver function test |
| LOTUSS | An open-Label, randOmized, Phase 2 sTUdy of the safety |
| | and tolerability of pirfenidone when administered to patients |
| LDL)/ | with Systemic Sclerosis-related interstitial lung disease |
| LPLV | last patient, last visit |
| MDT | multidisciplinary team |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMF | mycophenolate mofetil/sodium or mycophenolate acid |
| NAC | N-acetyl-cysteine |
| NCI | National Cancer Institute |
| NGS | next-generation sequencing |
| NSIP | nonspecific interstitial pneumonia |
| PDGF | platelet-derived growth factor |
| PDMS | protocol deviation management system |
| PFS | progression-free survival |
| PFTs | pulmonary function tests |
| PRO | patient-reported outcome |
| QTcF | QT interval corrected using Fridericia's formula |
| RBC | red blood cells |
| RBR | Research Biosample Repository |
| RNA | ribonucleic acid |
| RoW | Rest of the World |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SBP | systolic blood pressure |
| SGRQ | St. George's Respiratory Questionnaire |
| SOBQ | Shortness of Breath Questionnaire |
| SOC | System Organ Class |
| SOP | standard operating procedure |
| SpO2 | oxyhemoglobin saturation at rest |
| SQRT | Square root |

Pirfenidone — F. Hoffmann-La Roche Ltd

| SSc | systemic sclerosis |
|------|-------------------------------------|
| TEAE | treatment-emergent adverse event |
| TGF | transforming growth factor |
| TID | three times daily |
| UCSD | University of California, San Diego |
| UIP | usual interstitial pneumonia |
| ULN | upper limit of normal |
| US | United States |
| VAS | Visual Analogue Scale |
| VC | vital capacity |
| WBC | white blood cells |
| WGS | whole genome sequencing |

Pirfenidone — F. Hoffmann-La Roche Ltd

## 1. <u>BACKGROUND</u>

As described in section 1.3 of Clinical Study Protocol (CSP) version 2.0 dated 3 March 2017, no approved treatments are available for the 15% of patients with interstitial lung disease (ILD) who have unclassifiable disease. Therapeutic management is based on the most probable diagnosis after multidisciplinary discussions and consideration of the expected disease behavior (Antoniou et al. 2014). The data for pirfenidone in idiopathic pulmonary fibrosis (IPF) are sufficiently encouraging to hypothesize that a beneficial clinical effect would also be observed with this agent in patients with unclassifiable fibrosing ILD.

There are several key areas for uncertainty in the assessment of the benefit-risk profile for pirfenidone (Esbriet®) in the unclassifiable ILD patient population. Fibrosing ILD might have a different natural history compared with IPF and the efficacy of pirfenidone treatment may be different in patients with unclassifiable ILD compared with patients with IPF.

Mycophenolate mofetil/sodium or mycophenolic acid (MMF) may have an effect on the disease course of patients with unclassifiable ILD, in particular patients with interstitial pneumonia with autoimmune features (IPAF). Patients may be receiving treatment with MMF as a concomitant therapy at the start of the trial and therefore the patient population in this trial will be stratified according to use of MMF. Patients receiving MMF concomitant therapy at the start of the trial are allowed to continue with this treatment throughout the study including the 24-week double-blind and 12-month safety follow-up periods. A similar approach had been used previously in a study of the safety and tolerability of pirfenidone in patients with systemic sclerosis-related ILD (SSc-ILD; an open-Label, randomized, Phase 2 sTUdy of the safety and tolerability of pirfenidone when administered to patients with Systemic Sclerosis-related interstitial lung disease [LOTUSS]) (Khanna et al. 2016). The results of this trial also include data concerning the use of MMF as concomitant treatment with pirfenidone. The conclusion from this trial was that MMF, which was taken concomitantly with pirfenidone by 63.5% of patients, did not appear to affect the tolerability of pirfenidone and no particular safety concerns were noted following the combined use of MMF and pirfenidone.

#### 2. STUDY DESIGN

This is a multicenter, international, double-blind, two-arm, randomized, placebo-controlled Phase II trial in patients with fibrosing ILD who cannot be classified with moderate or high confidence into any other category of fibrosing ILD by multidisciplinary team (MDT) review ("unclassifiable ILD"). Patients will be randomized in a 1:1 ratio, on a double-blind basis using a stratified algorithm, to receive either pirfenidone (801 mg TID) or placebo. The randomized patients will be stratified by concomitant MMF treatment (yes/no), the presence/absence of IPAF as defined by the MDT.

In total, approximately 90 clinical centers (sites) in Australia, Europe, the Middle East, and North America are expected to enroll approximately 250 patients. Patients who are withdrawn from the trial will not be replaced.

Pirfenidone — F. Hoffmann-La Roche Ltd

After discussing the risks and benefits of the trial with the investigator and providing informed consent, patients will be required to taper and/or discontinue all prohibited medications (Section 4.4.2 in the CSP) in the 28 days prior to the start of screening during the washout period. If a prohibited medication must be tapered, the process must start early enough so that the patient discontinues the medication in the 28 days prior to the start of screening. After completing the washout patients will enter screening, which lasts up to 21 days. During screening, patients will be evaluated for eligibility based on the inclusion and exclusion criteria. Patients not taking a prohibited medication will forgo the washout period and directly enter screening.

At the end of screening, patients will be randomized (Day 1) to receive either pirfenidone or placebo (1:1 ratio).

Following treatment initiation, the daily dosage will be titrated to the full dosage of nine capsules per day over a 14-day period. After the titration period, trial treatment will continue through Week 24 and monitoring will be conducted by site visits. Patients should remain on a stable maintenance dose for the duration of the treatment period unless the dose is reduced or dosing is interrupted to manage an adverse event (see CSP Section 5.1.1). Any patient with an actual or anticipated interruption of trial treatment for a period of ≥28 consecutive days will be reported by telephone to Roche's medical monitor or designee to discuss the circumstances of the case. A Follow-up Visit will occur 28 days after the end of the 24-week double-blind treatment period.

After completion of the double-blind treatment period and the Follow-up visit at Week 28, patients will be given the opportunity to receive open-label pirfenidone within a safety follow-up period of up to 12 months of the trial protocol. A final Follow-up visit will be performed at the end of the safety period, 28 days after the last open-label dose. During the safety follow-up period, the patients should be evaluated by the investigator initially at monthly visits during the first 6 months and subsequently at each visit occurring approximately every 3 months thereafter.

#### 2.1 PROTOCOL SYNOPSIS

The Protocol Synopsis is in <u>Appendix 1</u> and the Schedule of Assessments in <u>Appendix 2</u> For additional details, please see the CSP Version 3, 28 June 2018 (and its Appendices).

#### 2.2 OUTCOME MEASURES

This trial will evaluate the efficacy and safety of pirfenidone in patients with fibrosing interstitial lung disease (ILD) who cannot be classified with moderate or high confidence into any other category of fibrosing ILD by multidisciplinary team (MDT) review ("unclassifiable" ILD).

The primary analysis of the primary and secondary efficacy outcome measures of this study is planned to be performed when the last patient reached the date of the last follow-up visit after end of the double-blind treatment period.

Pirfenidone — F. Hoffmann-La Roche Ltd

## 2.2.1 <u>Primary Efficacy Outcome Measures</u>

The primary efficacy objective for this trial is to evaluate the effect of pirfenidone vs. placebo on lung function parameters on the basis of Forced Vital Capacity (FVC) measurements. FVC will be measured daily by the patients by use of a handheld spirometry.

The primary efficacy endpoint is defined as:

 rate of decline in FVC in mL measured by daily handheld spirometer over the 24week double-blind treatment period.

## 2.2.2 Secondary Efficacy Outcome Measures

The secondary efficacy objective for this trial is to evaluate the efficacy of pirfenidone compared with placebo from baseline until Week 24 on other functional parameters, outcomes, and patient reported outcomes (PROs).

The following endpoints will be analyzed:

- Change in percent predicted FVC and in mL measured by spirometry during clinic visits
- Categorical change in FVC of >5% (absolute change in percent predicted and relative change in mL), measured by spirometry during clinic visits
- Categorical change in FVC of >10% (absolute change in percent predicted and relative change in mL), measured by spirometry during clinic visits
- Change in percent predicted diffusing capacity of the lung for carbon monoxide (DLco)
- Change in (6-minute walk distance) 6MWD in meters
- Change in University of California, San Diego Shortness of Breath Questionnaire (UCSD-SOBQ) score
- Change in score in Leicester Cough Questionnaire
- Change in cough visual analog scale
- Change in total and sub-scores of the St. George's Respiratory Questionnaire (SGRQ)
- Non-elective hospitalization, both respiratory and all cause
- Incidence of, and time to first, investigator-reported acute exacerbations
- Progression free survival (PFS), defined as the time to the first occurrence of a >10% absolute decline in percent predicted FVC (measured during a clinic visit), a >50 m decline of 6MWD, or death
- PFS, alternatively defined as the time to the first occurrence of a >10% relative decline in FVC (measured during a clinic visit), non-elective respiratory hospitalization, or death
- Time to death from any cause

Pirfenidone — F. Hoffmann-La Roche Ltd

• Time to death from respiratory diseases

## 2.2.3 <u>Exploratory Efficacy Outcome Measures</u>

One exploratory objective for this trial is to evaluate the role of mycophenolate mofetil/sodium or mycophenolic acid (MMF) treatment in ILD and to evaluate potential biomarkers associated with fibrosis and ILD.

The exploratory endpoints associated are:

- Efficacy and safety data from subgroups of patients who did or did not receive MMF treatment
- Biomarker data from plasma, serum, and whole blood ribonucleic acid (RNA) and deoxyribonucleic acid (DNA) samples

## 2.2.4 Safety Outcome Measures

The safety objective for this trial is to evaluate the safety of pirfenidone vs. placebo by investigating the following endpoints:

- Nature, frequency, severity, and timing of treatment-emergent adverse events
- Dose reductions and treatment interruptions
- Clinical laboratory test results
- 12-lead ECGs
- Withdrawals from trial treatment or trial discontinuations

All analyses with regard to the safety outcome measures will be performed from the date of first randomized treatment intake until 28 days after the last positive dose during the double-blind randomized treatment period.

#### 2.3 DETERMINATION OF SAMPLE SIZE

The purpose of this trial is hypothesis generation regarding the efficacy of pirfenidone vs. placebo on lung function parameters on the basis of rate of decline in FVC, as measured by daily handheld spirometry.

A total sample size of approximately 250 patients is planned, and patients will be randomized in a 1:1 ratio. The randomization will be stratified by concomitant MMF treatment (yes/no), the presence/absence of IPAF as defined by the MDT.

The planned sample size is based on the statistical hypothesis of the primary endpoint and assumes 80% power and a two-sided significance level of 5% using a student's t-test. It is assumed, after inspection of historical data, that FVC decline in the placebo arm is 85 mL with a common standard deviation of 70 mL, which can be reduced to 60 mL with a common standard deviation of 70 mL in the pirfenidone arm. In this

Pirfenidone — F. Hoffmann-La Roche Ltd

scenario, 125 patients per treatment arm are needed to detect this treatment effect with 80% power.

These assumptions are based upon the following considerations: in IPF, the annual rate of decline of FVC is approximately 200 mL. Owing to the fact that patients with unclassifiable ILD have rates of disease progression in the range of patients with IPF, albeit with a lower mortality rate (Ryerson et al. 2013), a similar decline rate of 200 mL/year, equivalent to a 100 mL decline over a treatment period of 24 weeks, can be expected. However, a yet unknown proportion of patients in this trial will be treated concomitantly with MMF. In a previous study of CTD-ILD (Fischer et al. 2013), MMF was found to have beneficial effects on lung functions in these patients. While CTD-ILD is a distinct entity from the current trial population, both conditions may share some autoimmune features. Therefore, assuming a smaller FVC decline of 85 mL in the placebo arm compared with 60 mL in the pirfenidone arm over the 24-week double-blind treatment period appears justified. In addition, the potential confounding effect of concomitant MMF therapy in these patients justifies stratification to ensure equal distribution of patients who receive and do not receive treatment with MMF.

#### 2.4 INTERIM ANALYSIS

There are no planned interim efficacy analyses for this trial.

#### 3. STUDY CONDUCT

The study conduct is described in <u>Section 2</u>.

#### 3.1 RANDOMIZATION, BLINDING AND UNBLINDING PROCEDURES

Patients will be randomized 1:1 to receive either pirfenidone or placebo. The randomization process will be conducted using a validated interactive voice or webbased response system (IxRS). To guard against systematic selection bias and ensure comparability of treatment arm, the randomization will be stratified by concomitant MMF treatment (yes/no), the presence/absence of IPAF as defined by the MDT.

To maintain the double-blind nature of the trial, the pirfenidone and placebo treatments will be identical in appearance (see CSP Section 4.3.1.1).

The investigational site personnel and the patients will be blinded to treatment assignment following randomization. The iDMC and any personnel performing any interim analysis (as applicable) will be unblinded to the treatment throughout the trial.

#### 3.2 INDEPENDENT REVIEW FACILITY

An independent review of home spirometry date (FVC (mL)) took place after it was recognized that the data collected for the primary analysis of this study was jeopardized by incorrect readings of the device and implausible values were collected due to technical issues. A new data set is available now after doing the reread of the FVC data and will be analyzed together with the previous data set collected to investigate the impact of the new data on the statistical results of this endpoint.

Pirfenidone — F. Hoffmann-La Roche Ltd

More details are provided in section 4.5.2.

#### 3.3 DATA MONITORING

An independent Data Monitoring Committee (iDMC) will review safety data and advice on study conduct at least three times during the study. Efficacy data will only be provided if requested by the iDMC. A first meeting is planned 6 months after start of recruitment, and subsequently at 12 and 18 months. Details on procedures and safety review by the iDMC are described within an iDMC charter.

#### 4. STATISTICAL METHODS

Categorical data will be summarized using frequencies and percentages (including a category for missing, if appropriate). Percentages will be based on the number of patients in each treatment arm for the analysis population, if not otherwise specified.

Continuous endpoints will be summarized using descriptive statistics (mean, standard deviation, minimum, 25th and 75th quartiles, median, and maximum).

Where data will be summarized over time, the following timepoints will be presented as applicable: Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28 (if applicable) and early discontinuation visit.

Data analysis of data collected during the 12-month safety follow-up period will be described in section 4.7.

Where applicable other analysis methods will be specified below.

#### 4.1 ANALYSIS POPULATIONS

#### 4.1.1 Intent-to-treat Population

The intent-to-treat (ITT) population is defined as all randomized patients. Patients in the ITT population will be assigned to treatment arm as randomized (planned treatment). The ITT population is the primary analysis population for all efficacy analyses. The time period for all efficacy analyses is defined from date of randomization until the treatment completion date of the double-blind treatment period or the date of early discontinuation collected on the early treatment discontinuation eCRF page in case a patient does not complete the planned 24 weeks of double-blind treatment.

#### 4.1.2 Per Protocol Population

Not applicable.

#### 4.1.3 Safety Population

The safety population is defined as all patients with at least one intake of pirfenidone or placebo, i.e. at least one record in the drug-log of the double-blind period with a non-zero dose. Patients in the safety population will be assigned to treatment arm according to the actual treatment they received.

Pirfenidone — F. Hoffmann-La Roche Ltd

## 4.1.4 Safety Follow-up Population

For the 12-month safety follow-up period, the safety follow-up population will be defined as all patients who have received at least one dose of pirfenidone after the randomized treatment end plus 28 days.

Safety analyses for the 12-month follow-up period will be performed from the date of the first pirfenidone drug intake during safety follow-up period up to the study completion/discontinuation visit.

## 4.2 TRIAL PERIODS, OBSERVATION AND ANALYSIS TIMES

Where durations are to be calculated (e.g. treatment duration), these will be derived based on the interval in days (end date – start date + 1) and converted to months and years if needed, using 30.4375 and 365.25, respectively, as denominator if not otherwise specified.

For the investigational medicinal product (IMP) exposure, treatments administered from the date of first randomized pirfenidone/placebo treatment up to the date of completion of double-blind treatment or date of early treatment discontinuation, will be regarded.

For drug safety, analyses will be restricted to AEs or assessments that occurred from the first day of randomized treatment until the date of last positive dose of randomized treatment plus 28 days.

Safety analyses for the 12-month follow-up period will be performed using the time window from the safety follow-up period start up to the study completion/discontinuation visit.

## 4.2.1 Study Days

Study days will be defined as the number of days since randomization, and is calculated as:

- Study day = Assessment date randomization date + 1, for assessments on or after the randomization date.
- Study day = Assessment date randomization date, for assessments before the randomization date.

The day of randomization will be study day 1.

Pirfenidone — F. Hoffmann-La Roche Ltd

## 4.2.2 <u>Baseline and Screening Observations</u>

## Table 1 Definition of Baseline and Screening Observations

| | Definition |
|---|---|
| Baseline data | Baseline is defined as the last valid assessment prior to first intake of randomized study drug (pirfenidone/placebo). |
| | This may not be the same as the Day 1 (Week 1) visit as per eCRF. In case that Day 1 (Week 1) visit data is missing and the randomized treatment is given, data from the screening period will be used as baseline. In addition, if randomized treatment is not given then baseline will be defined as the last valid assessment collected either screening or day 1. |
| | Generally, it is assumed that measurements referring to the Day 1 (Week 1) visit have been performed before randomized study drug (pirfenidone/placebo) was given. |
| | Adverse events occurring on the date of first randomized pirfenidone/placebo treatment will not be considered baseline, but treatment-emergent. |
| Screening data | Screening measurements are all the measurements performed before the randomization date. |

# 4.2.3 <u>On-treatment Assessments for Efficacy Analyses (Double-blind Treatment Period)</u>

For efficacy analyses, on-treatment assessments will be the assessments performed on or after the randomization date until the double-blind treatment completion or discontinuation date.

## 4.2.4 <u>On-treatment Assessments for Safety Analyses (Double-blind Treatment Period)</u>

For safety analyses, on-treatment assessments will be the assessments performed on or after the first dose of randomized pirfenidone/placebo date until the last positive dose of randomized treatment plus 28 days.

## 4.2.5 On-treatment Assessments (12-Month Safety Follow-up Period)

Details of all data recorded during the 12-month safety follow-up period will be presented. This period starts on the day of the first positive dose of pirfenidone after the 28 days follow-up visit for patients who completed the double-blind treatment period without being discontinued the study. The safety follow-up period ends with the study completion/discontinuation visit, with a maximum duration of 12 months plus 28 days.

Pirfenidone — F. Hoffmann-La Roche Ltd

Safety follow-up analyses will be presented separately from double-blind treatment phase ones.

## 4.2.6 <u>Cut-off points</u>

The clinical cut-off for the primary analysis will occur when the last patient has completed the final safety Follow-up Visit, 28 days after the double-blind treatment period.

There will be a second cut-off for the final analysis when all patients have completed the 12-month safety follow-up period.

For each patient the total length of the trial is expected to be up to a maximum of 91 weeks. The trial duration includes the washout period of up to 4 weeks, the screening period of up to 3 weeks, the double-blind treatment period of 24 weeks, the follow-up period of 4 weeks, the open-label safety follow-up period up to 12 months (52 weeks) plus 28 days and a final safety Follow-up Visit 4 weeks after the last dose.

#### 4.3 ANALYSIS OF TREATMENT ARM COMPARABILITY

To ensure the comparability of the treatment arm, the randomization will be stratified by the availability of a previous MMF treatment (yes/no) and the presence/absence of IPAF as defined by MDT to ensure an equal distribution of patients.

These stratification factors will be included in the analysis of the primary endpoint as a sensitivity analysis. Please refer to the corresponding section 4.4.5 for further details.

Outputs for concordance between the stratification factors by eCRF and by IxRS will also be presented.

#### 4.4 ANALYSIS OF STUDY CONDUCT

Unless otherwise specified, all analyses described in this section will be performed on the ITT population, presenting data by treatment arm.

#### 4.4.1 Patient Disposition

An overview on patient disposition, showing number and percentages of patients enrolled, screened, failed screening, randomized, treated, completed or early discontinued the double-blind treatment period, patients entering the 12-month safety follow-up period and their current status (ongoing, completion, discontinued) in that period will be provided. For patients who have early discontinued the double-blind treatment period or the study, frequencies of reasons for early discontinuation will be provided. A listing with all the patient disposition data will be also presented.

The following definitions will be used:

 Patients randomized: All patients who have been randomized to receive either pirfenidone or placebo, i.e. have a randomization date.

Pirfenidone — F. Hoffmann-La Roche Ltd

- Patients randomized and not treated: all randomized patients who have not received at least one dose of the randomized treatment.
- Patients randomized and treated: all randomized patients who have received at least one dose of the randomized treatment.
- Patients randomized and treated with sufficient post-baseline efficacy data: all randomized patients who have received at least one dose of the randomized treatment and have at least one post-baseline assessment of FVC (mL).
- Completion of double-blind treatment period: eCRF question "Did the patient complete course of double-blind treatment?" is ticked "Yes" (eCRF form "Doubleblind treatment Completion/Early Discontinuation").
- Early discontinuation (non-completion) of double-blind treatment period: eCRF
  question "Did the patient complete course of double-blind treatment?" is ticked "No"
  (eCRF form "Double-blind treatment Completion/Early Discontinuation").
- Early discontinuation (non-completion) of study: eCRF question "Did the subject early discountinue from the study?" is ticked "Yes" (eCRF form "Study Completion/Early Discontinuation") for patients who discontinued double-blind treatment period.
- Status during the 12-month safety follow-up (entered, ongoing, completed).
   Completers are defined as those patients that have filled the study completion/discontinuation form. Otherwise, the patient is considered ongoing in the safety follow-up phase.
- Completion of study: eCRF question "Did the subject complete the study?" is ticked "Yes" (eCRF form "Study Completion/Early Discontinuation")
- Early discontinuation (non-completion) of study: eCRF question "Did the subject early discountinue from the study?" is ticked "Yes" (eCRF form "Study Completion/Early Discontinuation")

An overview on patients' enrolment will be provided based on the randomized subjects by country and center separately for the pirfenidone and placebo arm.

Kaplan-Meier (KM) plots for time to treatment discontinuation will be provided for all randomized patients and by randomized arm, based on the date subject completed or early discontinued from double-blind treatment period, as per eCRF. If the patient completed the treatment without treatment discontinuation, then it will be censored to the date of treatment completion.

In addition, KM plots for time to study discontinuation will be presented for all randomized patients by arm, based on the study discontinuation date. If the patient completed the study as planned per protocol, then the patient will be censored to the study completion date.

Pirfenidone — F. Hoffmann-La Roche Ltd

In addition, a consort diagram with some of the categories above will be presented.

#### 4.4.2 Major Protocol Deviations

Major protocol deviations and eligibility violations will be summarized by frequency tables and all patients with protocol deviations will be listed. Protocol deviations will be collected in the protocol deviation management system (PDMS), reviewed by the medical monitors. All deviations provided in that dataset will be considered as major protocol deviations.

## 4.4.3 Demographic and Baseline Characteristics

Baseline and disease characteristics such as demographics, medical history and tobacco use history will be summarized by descriptive statistics or frequency tables for each treatment arm.

#### **Demographics**

The following demographic characteristics will be summarized by treatment arm:

- Age (years): as entered in the eCRF at the screening visit.
- Age categories: <65, and ≥ 65.
- Age categories: <45, ≥45 to <65 years, ≥65 to <85 years, and ≥ 85 years.
- Gender: Male/Female.
- Race: White, American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, Unknown. In case that more than one race will be ticked, a concatenated variable, containing all races will be presented (e.g. Asian/White).
- Ethnicity: Hispanic or Latino, Not Hispanic or Latino, Not reported, Unknown.
- Weight (kg) at baseline
- Height (cm) at baseline
- BMI (kg/m2) at baseline. BMI will be calculated as: weight(kg) / (height(m))2
- Female reproductive status: childbearing potential without contraceptive protection, Childbearing potential with contraceptive protection, surgically sterilized, Postmenopausal, Pre-menarchal, Non childbearing potential.

Data on female reproductive status will be presented descriptively.

Demographic data will be also listed.

Pirfenidone — F. Hoffmann-La Roche Ltd

## **Medical History**

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), version 20.1 or higher and will be summarized presenting numbers and frequencies by primary System Organ Class (SOC) and Preferred Term (PT) by treatment arm. If patients have more than one disease within a SOC or PT they will be counted only once for the respective SOC or PT.

A listing with past and ongoing medical history data from the washout period will be presented.

## **Tobacco use history**

The history of tobacco use will be summarized by treatment arm with the following characteristics:

- Tobacco use history (never, current, previous)
- Nicotine exposure (pack-years), smokers only

Numbers and percentages of patients will be provided for tobacco use history. Nicotine exposure will be summarized descriptively.

#### Diagnosis and time from uILD Diagnosis

Frequencies and percentages will be presented for the uILD category collected into the eCRF page MDT/Diagnosis (Eligibility).

The time in months since the original uILD diagnosis will be calculated as

Date of randomization – Date of ILD diagnosis and will be summarized descriptively by randomized treatment arm. The number and percentage of patients with a historical high-resolution computed tomography and with a historical surgical lung biopsy will also be presented.

Descriptive statistics of the time from most recent historical high-resolution computed tomography (months) and historical surgical lung biopsy will be presented. As above, the date of randomization will be used as reference date for calculation of duration.

#### Stratification Factors

The number and percentage of patients that fall into each of the four groups based on the two stratification factors: Concomitant MMF treatment (yes/no), and the presence/absence of IPAF as defined by the MDT will be presented by treatment arm.

#### **Baseline Site Spirometry Test**

The values recorded for the baseline assessments of the site spirometry tests were the following:

Pirfenidone — F. Hoffmann-La Roche Ltd

- Forced vital capacity (FVC) (L and % predicted)
- Forced expiratory volume in 1 second (FEV1) (L and % predicted)
- FEV1 (L) / FVC (L) ratio (1)
- Carbon monoxide diffusing capacity (DLco) (% predicted)

Descriptive statistics will be provided for these parameters separately for treatment arm.

## **Historical Spirometry Test**

The number and percentage of patients who performed spirometry test (FVC, DLco, FEV1, and FEV1/FVC ratio) in the past will be provided. The most recent assessment before the Screening visit will be collected:

- Hemoglobin corrected DLco (mmol/min/kPa and %)
- DLco/Va (KCO) (mL/min/mmHg/L and % predicted)
- FVC (L and % predicted)
- FEV1 (L and % predicted)
- FEV1(L)/FVC(L) ratio (1)

These historical spirometry test parameters will be summarized using descriptive statistics by treatment arm. Both, absolute and percent predicted values will be presented. Frequencies and percentages will be presented for the high-resolution computed tomography and the surgical lung biopsy.

#### Baseline 6-minute walk distance (6MWD)

The 6MWD is used to evaluate the functional capacity of patients with lung disease. The 6MWD measures the distance a patient is able to walk quickly on a flat, hard surface in a period of 6 minutes.

The number and percentage of patients that

- Performed the 6-minute walking test (yes/no),
- Rested for at least 10 minutes (yes/no),
- Stopped the test before 6 minutes (yes/no),
- Required O2 (yes/no)

at the baseline visit will be summarized by randomized treatment group.

Pirfenidone — F. Hoffmann-La Roche Ltd

The values of the parameters recorded for the 6MWD test are:

- Vital signs (Heart rate (beats/min), systolic blood pressure (mmHg), diastolic pressure (mmHg)) (before the test, at the end of the test)
- Distance walked (m),
- Oxyhemoglobin saturation (SPO2) (before the test (at rest), at the end of the test),
- Oxygen (O2) requirements (L) for patients who received oxygen (at the end of the test)

will be summarized descriptively by treatment arm.

## 4.4.4 Previous and Concomitant Medication

Previous and concomitant medications will be presented based on the safety population. Post medications administrated during the safety follow-up period will be presented based on the safety follow-up population.

Previous and concomitant medications are non-study medications. Concomitant therapy includes any medication used by a patient from the washout period until 28 days after the last dose of trial treatment. The previous and concomitant medication will be coded using the Genentech (GNE) drug dictionary. This is a proprietary Roche Dictionary which is used to code concomitant medications in the Trial Management System (TMS) coding tool. The Standardized Medication Name (CMDECOD), which is the medication generic or combination generic as defined by the Drug Thesaurus (proprietary Genentech/Roche dictionary), and the Medication Class (CMCLAS), which is the primary medication class as defined by the Drug Thersaurus, will be used for the analyses.

Therapies will be classified as previous or concomitant as follows:

Previous: If the medication start date is prior to start of double-blind treatment,

Concomitant: If medication is taken at any time between the start of double-blind treatment and 28 days after last positive dose of randomized treatment.

Post (safety follow-up): If the medication is taken more than 28 days after the last positive dose of randomized treatment.

The number and frequency of previous and concomitant medications taken by patients in the two treatment arms will be presented by Medication Class and Standardized Medication Name. If patients receive more than one drug within a Medication Class or Standardized Medication Name they will be counted only once for the respective Medication Class or Standardized Medication Name.

Pirfenidone — F. Hoffmann-La Roche Ltd

A separated table will be presented for post medications during the safety follow-up period.

All medications will be listed identifying the previous/concomitant and post medications.

The missing imputation rules for the medication dates are described under Section 4.9..

## 4.4.5 <u>Daily Spirometry (Handheld Device)</u>

A handheld spirometry device will be used by the patient to measure daily FVC at home. Confirmatory site (trial center) based FVC measurements will be conducted every 4 weeks. The following blow categories will be collected:

| Quality description | Acceptable text |
|---------------------|-----------------|
| Accepted | YES |
| Rejected | NO |
| Borderline Accepted | BOR |

Only accepted blows will be considered for the analysis. If one patient has more than one measurement per day, the last measurement will be taken.

FVC (mL) will be measured daily with a handheld device.

After primary analysis of study data it was detected that FVC values from home spirometry were impacted by high variability and implausible values were accepted by the system. In order to evaluate the issue a re-read of home spirometry data will be performed and the new dataset with modified flagging of acceptable values will be analyzed in the same way as described below for the primary endpoint, see also 4.5.2.

#### 4.4.6 Compliance

With respect to the home-based daily measurements compliance of patients will be investigated. It will be analyzed if gaps of measurements occur over time. A gap is thereby defined as 7 or more than 7 consecutive days of missing measurements. A summary table displaying number of patients with gaps in daily measurements, number of gaps and duration of gaps will be provided by treatment arm for data from handheld spirometer.

#### 4.5 EFFICACY ANALYSIS

The primary and secondary efficacy analyses will include all patients in ITT population, with patients grouped according to their assigned treatment.

Pirfenidone — F. Hoffmann-La Roche Ltd

The primary analysis of the primary efficacy endpoint of this study is planned to be performed when the last patient reached the date of the last follow-up visit after end of the double-blind treatment period (clinical cut-off date).

#### 4.5.1 <u>Primary Efficacy Endpoints</u>

The primary efficacy objective for this trial is to evaluate the efficacy of pirfenidone vs. placebo on lung function parameters on the basis of rate of decline in FVC in mL measured by handheld spirometer over the 24-week double-blind treatment period.

The primary analysis will be based on the ITT population. Patients who discontinue treatment prematurely will be analyzed based on the available data. No imputation method will be applied for the primary endpoint.

The primary analysis of the primary endpoint will compare the mean FVC decline in each treatment arm using a student's t-test with a two-sided significance level  $\alpha$ =0.05. The mean FVC decline for each treatment arm will be calculated using the estimated FVC decline for each individual patient. The estimated FVC decline for individual patients will be obtained by applying a linear regression model to all data points collected during the 24-week double-blind treatment period:

$$X_{it} = \alpha_i + \beta_i D_{it} + u_{it}$$

where

 $X_{it}$  = the FVC measurements (mL) of patient i on day t, with i=1,...,N and t=1,...,T, being N the total number of patients randomized and T the total number of days with assessment.

 $D_{i*}$  = study day t of patient i

 $\alpha_i, \beta_i$  = intercept and slope of the individual linear regression of patient i

The time-adjusted decline for patient i is then obtained by estimating the patients' individual difference in predicted values between baseline and week 24 from the linear regression.

In a further step, the time-adjusted mean FVC decline is estimated by calculating the mean over all individual time-adjusted declines of all patients by treatment arm.

A summary table displaying the mean FVC decline together with two-sided 95% confidence intervals based on percentiles of the t-distribution will be provided by treatment arm. The mean FVC decline in each treatment arm will be compared using a student's t-test with a two-sided significance level  $\alpha$ =0.05. Additionally, a two sample Wilcoxon test will be used for treatment comparison. Results of this test are of descriptive nature only.

The same analyses will be done by restricting the FVC decline values:

- Including patients with at least 3 site spirometry measurements Pirfenidone — F. Hoffmann-La Roche Ltd

- excluding patients with a predicted FVC decline below -1000 mL
- or above 1000 mL
- excluding values with a difference +/-50% from corresponding baseline site spirometry

Mean FVC declines and results from Student's t-test by subgroups (for definition see 4.5.6) will be displayed in a forest plot.

As a sensitivity analysis to the primary analysis, the time-adjusted mean FVC decline will be estimated by a repeated measures mixed model with patient effects fitted as random and day of measurement and treatment fitted as fixed effects. Please refer to <a href="Section-4.5.6">Section 4.5.6</a> for further details.

A detailed description of SAS code to be used for the repeated measures mixed model is provided together with the respective table shell.

## 4.5.2 Reassessment of quality of home spirometry

Due to the nature of the home FVC measurements resulting in a highly skewed distribution with high unexpected variability and a number of measurements resulting in physiologically implausible values the home spirometry data was reassessed by an independent and blinded group of experts.

The reassessment of home spirometry data resulted in a flag with 2 categories:

130 = acceptable, 110 = not acceptable.

A comparison between the quality assessments before and after update will be presented by a concordance analysis. In this analysis old assessments with "BOR" are tabulated as non-acceptable quality.

The compliance of home spirometry data will also be assessed by analyzing the number of gaps in daily measurements.

## 4.5.3 Secondary Efficacy Endpoints

For secondary endpoints, all data from baseline until Week 24 will be taken into account for the statistical analysis. In a similar manner to the primary endpoint data, patients who discontinue early will be analyzed based on the data collected until date of withdrawal from treatment

The secondary efficacy objective for this trial is to evaluate the efficacy of pirfenidone compared with placebo on the basis of the following endpoints:

 Descriptive statistics for values and changes from baseline over time of all spirometry test parameters will be presented.

Pirfenidone — F. Hoffmann-La Roche Ltd

- The decline of FVC in mL measured by spirometry during site (clinic) visits will be compared between the treatment arms in the same fashion as described for the primary endpoint. A Wilcoxon tests was not planned for this endpoint.
- Mean FVC declines and results from Student's t-test by subgroups (for definition see 4.5.6) will be displayed in a forest plot.
- In addition the decline of FVC in mL measured by spirometry during site (clinic) visits will be compared between the treatment arms using a repeated measures mixed effects model. Please refer to <a href="Section 4.5.6">Section 4.5.6</a> for further details.
- The absolute change in percent predicted FVC measured by spirometry during site visits at week 24 will be compared between the treatment arms using a rank analysis of covariance (ANCOVA). Change from baseline will be used as an outcome variable and standardized rank baseline value will be used as a covariate
- Categorical changes in FVC (mL) measured during site (clinic) visits of >5% and >10% will be compared between the treatment arms using a Cochran-Mantel-Haenszel test stratified by concomitant MMF medication use (Yes/No), and the presence/absence of IPAF as defined by the MDT
- Absolute change from baseline to week 24 in percent predicted DLco will be compared between the treatment arms using a rank ANCOVA. Change from baseline to week 24 will be used as an outcome variable and standardized rank baseline value will be used as a covariate
  - A summary table presenting the values of DLco (%) and its change from baseline will be presented over time and by treatment arm.
- The absolute change in 6MWD will be analyzed using a rank ANCOVA model.
   The 6MWD recorded at 24 weeks will be used as an outcome variable and standardized rank baseline 6MWD will be used as a covariate
  - A summary table presenting the 6MWD parameters and their change from baseline will be presented over time and by treatment arm.
- The absolute change in UCSD-SOBQ total score will be analyzed using a rank ANCOVA model. The UCSD-SOBQ total score recorded at 24 weeks will be used as an outcome variable and standardized rank baseline UCSD-SOBQ score will be used as a covariate Please see Section 4.5.5 for further details.
- The absolute change in Leicester Cough Questionnaire total score will be analyzed using a rank ANCOVA model. The Leicester Cough Questionnaire total score recorded at 24 weeks will be used as the outcome variable and standardized rank baseline Leicester Cough Questionnaire total score will be used as a covariate. Please see <u>Section 4.5.5</u> for further details.

Pirfenidone — F. Hoffmann-La Roche Ltd

- The change in cough visual analog scale will be analyzed using a rank ANCOVA model. The result recorded at 24 weeks will be used as the outcome variable and the standardized rank baseline result will be used as a covariate. Please see Section 4.5.5 for further details.
- The change in total of the SGRQ will be analyzed using a rank ANCOVA model.
  The scores recorded at 24 weeks will be used as outcome variables and the
  standardized rank baseline scores will be used as covariates. Please see <u>Section</u>
  4.5.5 for further details.
- The time from randomization to the first occurrence of all-cause non-elective hospitalization and respiratory non-elective hospitalization will be analyzed using Kaplan-Meier (KM) techniques:
  - KM plots of time to first occurrence of the different events will be provided by treatment arm. Frequencies and percentages of patients with events and patients censored will be provided. Descriptive statistics of KM estimates of the time to first occurrence (weeks) will be presented.
  - Log-rank tests based on the time to the first event will be used to compare the two treatment arms.
  - Hazard ratios and corresponding 95% CI will be calculated by applying Cox-proportional hazard models in which the four groups from the two randomization stratification factors are included in the model.
- The incidence of investigator reported acute exacerbations in the two treatment arms will be compared with Fisher's exact test.
  - o Incidence of, and time to first, investigator-reported acute exacerbations
- Progression free survival (PFS), defined as the time to the first occurrence of a >10% absolute decline in percent predicted FVC, a >50 m decline of 6MWD, or death from any cause, will be analyzed using Kaplan-Meier techniques:
  - KM plots of time to first occurrence of the combined primary efficacy endpoint will be provided by treatment arm.
  - Frequencies and percentages of patients with events and patients censored will be provided. Descriptive statistics of KM estimates of PFS (weeks) will be presented.
  - The PFS of two randomized treatment arms will be compared with a logrank test.
  - Hazard ratios and corresponding 95% CI will be calculated by applying Cox-proportional hazard models.
- An alternative definition of PFS (also in weeks), namely the time to the first occurrence of a >10% relative decline in FVC, non-elective respiratory hospitalization, or death, will be analyzed using Kaplan-Meier techniques as Pirfenidone — F. Hoffmann-La Roche Ltd

- defined for the point above; and the two treatment arms will be compared with a log-rank test. In addition, hazard ratios and corresponding 95% CI will be calculated by applying Cox-proportional hazard models
- Time to death from any cause and time to death from respiratory diseases
  assessed by the SOC "Respiratory, thoracic and mediastinal disorders" (in weeks)
  will be analyzed using Kaplan-Meier techniques as defined above; and the two
  treatment arms will be compared with a log-rank test. In addition, hazard ratios
  and corresponding 95% CI will be calculated by applying Cox-proportional
  hazard models.

For all secondary endpoints p-values will be reported in a descriptive fashion. No multiplicity adjustments for statistical testing will be done.

#### 4.5.4 Exploratory Efficacy Endpoints

The exploratory objectives for this trial are to evaluate the role of MMF treatment in ILD and to investigate potential biomarkers associated with fibrosis and ILD.

For the MMF objective, primary and selected secondary endpoints will be investigated by means of a subgroup analyses that stratifies patients according to whether they received MMF treatment. In addition, the overall safety summary will be presented by this subgroup. The selected secondary endpoints are:

- Deaths from any cause and respiratory disease-related
- Hospitalizations from any cause and respiratory disease-related

The analysis of these exploratory efficacy endpoints by subgroup are defined under section <u>Section 4.5.6.</u>

The mean FVC decline in each treatment arm will be calculated as in the primary analysis for the subgroups of patients that received MMF treatment and compared using a student's t-test.

Other exploratory efficacy endpoints are discussed in the sensitivity and subgroup sections (see <u>Section 4.5.6</u> and <u>Section 4.5.7</u>, respectively).

Moreover, additional categorical analyses for the percent predicted DLco and 6MWD will be presented as exploratory:

- Categorical change of >15% absolute decline from baseline to week 24 in percent predicted DLco will be compared between the treatment arms using a logistic regression.
- Categorical change of >50% absolute decline from baseline to week 24 in 6MWD
   (m) will be compared between the treatment arms using a logistic regression.

Pirfenidone — F. Hoffmann-La Roche Ltd

For the biomarker objective, assessments of the exploratory biomarkers and their relationship with drug responses will be described in a separate analysis plan.

A correlation analysis of individual patient slopes estimated by linear regression models between those obtained for home spirometry and site spirometry were performed to assess the concordance of the data obtained by the two methods.

#### 4.5.5 Analyses of Patient-Reported Outcomes

Several PRO assessments will be conducted in this trial, including the UCSD-SOBQ, the Leicester Cough Questionnaire, the cough visual analog scale, and the SGRQ.

PRO data will be collected via questionnaires to document the treatment effect and to evaluate the benefit of pirfenidone. The questionnaires, translated into the local language as required, will be completed in their entirety at specified time points during the trial. To ensure instrument validity and that data standards meet health authority requirements, questionnaires will be self-administered before the patient receives any information on disease status and prior to the performance of non-PRO assessments, unless otherwise specified.

## St. George's Respiratory Questionnaire (SGRQ)

The St. George's Respiratory Questionnaire (SGRQ) is an index designed to measure and quantifies health-related health status in patients with chronic airflow limitations. The SGRQ is a 50-item questionnaire, addressing the frequency of respiratory symptoms (items 1-8), the patient's current state (sections 9-16). From the 50 items a total score, as well as three component scores (Symptoms, Activities, Impacts) will be derived. The total score ranges from 0, presenting the best possible health status to 100, presenting the worst possible health status.

The change in SGRQ total score will be of primary interest when assessing health-related quality of life (HRQoL).

The analysis of PROs assessed by SGRQ total score and by SGRQ component scores for symptoms, activity, and impacts will be analyzed as follows:

- The absolute score values and changes from baseline for the total and each subscore will be presented descriptively over time by treatment arm.
- Changes from baseline to week 24 or early discontinuation visit will be compared between the treatment arms using a rank ANCOVA with change from baseline as outcome variable and standardized rank baseline value as covariate. This analysis will be done only for the total score.

The SGRQ and the details for calculating the score can be found in Appendix 3.

Pirfenidone — F. Hoffmann-La Roche Ltd

## The University of California, San Diego-Shortness of Breath Questionnaire (UCSD-SOBQ)

The University of California, San Diego-Shortness of Breath Questionnaire (UCSD-SOBQ) is a symptom-specific, 24-item, patient-self-administered questionnaire that assesses shortness of breath while doing a variety of activities of daily living. Each of the 24 activities are rated on how dyspnea affects the activity on a 6-point scale: 0 = None at all to 5 = Maximal or unable to do because of breathlessness. The scores will be summarized to a total score, ranging from 0 - 120.

The total score of the UCSD SOBQ will be summarized as follows:

- The absolute total scores and changes from baseline will be presented descriptively over time by treatment arm.
- Changes from baseline to week 24 or early discontinuation visit will be compared between the treatment arms using a rank ANCOVA with change from baseline as outcome variable and standardized rank baseline value as covariate.

Additional details on the UCSD SOBQ can be found in Appendix 3

#### The Leicester Cough Questionnaire

The Leicester Cough Questionnaire is a patient-reported questionnaire evaluating the impact of cough on quality of life. The questionnaire comprises 19 items and takes 5 to 10 minutes to complete. Each item assesses symptoms, or the impact of symptoms, over the last 2 weeks on a seven-point Likert scale. Scores in three domains (physical, psychological and social) are calculated as a mean for each domain (range 1 to 7). A total score (range 3 to 21) is also calculated by adding the domain scores together. Higher scores indicate better quality of life.

The total score and the physical, psychological and social domain scores of the Leicester Cough Questionnaire will be analyzed as follows:

- The scores and changes from baseline will be presented descriptively over time by treatment arm.
- Changes from baseline to week 24 or early discontinuation visit will be compared between the treatment arms using a rank ANCOVA with change from baseline as outcome variable and standardized rank baseline value as covariate. This analysis will be done only for the total score.

Details on calculating the domain scores can be found in Appendix 3

## The Cough VAS

This visual analogue scale is designed to help us learn about the severity of your cough. This scale is 100mm (10cm) in length.

Pirfenidone — F. Hoffmann-La Roche Ltd

The cough VAS score will be summarized descriptively by visit and treatment arm. The change in cough VAS will be analyzed using a rank ANCOVA model. The change in VAS score for cough recorded at 24 weeks will be used as the outcome variable and the standardized rank baseline result will be used as a covariate. Please refer to <a href="Appendix 3">Appendix 3</a> for further details.

#### 4.5.6 Sensitivity Analyses

As a sensitivity analysis to the primary analysis, the time-adjusted mean FVC decline will be estimated a random slope and intercept linear regression model, with an absolute change in FVC (mL) as the outcome variable assuming linear decline in lung function over time. The model includes random coefficients for slope and intercept and fixed effect terms for treatment, and covariates to be selected as described below. The statistical model is defined as follows:

$$Y_{ijk} = (\alpha + a_i) + (\gamma + \beta_s T_k + g_i) t_{ij} + \beta_g Cov 1_i + \beta_a Cov 2_i + \epsilon_{ij}$$

- o Y<sub>ijk</sub> is the value measured for ith patient at time j in treatment group k
- o t<sub>ij</sub> is the time of measurements for ith patient at study day j
- $\circ$  T<sub>k</sub> =0 if patient in Placebo group and T<sub>k</sub>=1 is patient in Pirfenidone
- $\circ$   $\beta_s$  is the effect of Pirfenidone on the slope
- $\circ$   $\alpha$  and  $\gamma$  are elements of the intercept and slope respectively  $a_i$  and  $g_i$  are random specific components of the intercept and slope for the ith patient
- $\circ$   $\beta_g$ ,  $\beta_a$  are patient specific demographics' coefficients (strata)
- o Cov1<sub>i</sub>, Cov2<sub>i</sub> are covariates to be included for the ith patient
- ο ε<sub>ii</sub> is the random error for ith patient at time j
- o a<sub>i</sub> and g<sub>i</sub> are assumed to be normally distributed with mean 0 and arbitrary covariance matrix
- $\circ$  ε<sub>ij</sub> are assumed to be independent and normally distributed with mean 0 and variance  $\sigma$ ε<sup>2</sup>
- Within patient errors follow a random coefficient regression model with random effect for intercept and slope
- An unstructured variance-covariance structure will be used to model the within patient measurements
- The variance-covariance matrix, modeled to estimate the inter-individual variability is considered to have a Variance-Components structure

The model will be applied by adding the stratification factors MMF treatment and IPAF as covariates to the home spirometry data, once taking into account the old and once the new quality flag.

The same model with and without adding the stratification factors as covariates will be applied to the key secondary endpoint of site-measured FVC (mL).

Pirfenidone — F. Hoffmann-La Roche Ltd

#### 4.5.7 Subgroup Analyses

Subgroup analyses will be conducted for the exploratory endpoint, as described in Section 4.5.4. The following subgroups will be based on:

- The four groups resulting from combinations of the two stratification factors:
  - Concomitant MMF treatment (yes/no)
  - o Presence/absence of IPAF as defined by the MDT
- Gender: Male, Female
- Age (years): <65 years, ≥ 65 years
- Percent predicted FVC at Baseline: <65%, ≥65% to < 80%, ≥80%</li>
- Percent predicted DLco at Baseline: <35%, ≥35%</li>
- Body weight: <60 kg, ≥60 kg</li>
- Previous Biopsy (yes/no)

## 4.5.8 <u>Sensitivity Analyses for missing data</u>

The robustness of the primary method of estimation described above will be explored by a series of sensitivity estimators based on varying assumptions underlying the multiple imputation strategy.

As the primary analysis for this study was performed in March 2019 the number of patients with missing FVC values at week 24 are known. No data was collected after treatment discontinuation.

3 different approaches will be used to evaluate the robustness of the analysis of the secondary endpoint to the missing at random (MAR) assumption.

Due to the low number, deaths and other intercurrent events have not been considered in the multiple imputation analysis.

#### 4.5.8.1 Fixed missing imputation based on Placebo distribution

To evaluate the robustness of the analysis of the second endpoint to the missing at random (MAR) assumption missing data of both treatment groups will be imputed by descriptive statistics derived from the distribution of the placebo group. For each visit the following descriptive statistics of FVC (mL) will be calculated from the placebo group only: lower quartile, median, upper quartile.

Pirfenidone — F. Hoffmann-La Roche Ltd

For each of the 2 treatment groups 3 datasets with imputed missing values will be created:

- Missing values imputed by median of placebo group for the respective visit
- Missing values imputed by lower quartile of placebo group for the respective visit
- Missing values imputed by upper quartile of placebo group for the respective visit

Then, within each of the 9 possible combinations of datasets two analyses will be performed:

The mean FVC decline in the treatment arms will be compared using a student's t-test. The mean FVC decline for each treatment arm will be calculated using the estimated FVC decline for each individual patient, which will be obtained by applying a linear regression model to the data over time of the respective patient.

The decline in FVC (mL) at week 24 will be estimated from a random slope and intercept model. This model will include fixed effects for treatment, the stratifying variables concomitant use of MMF and presence/absence of IPAF and treatment-by time-interaction. Random effects will be included for both time and intercept.

The difference between treatment groups will be calculated together with the corresponding p-value.

A table will present the results from the two analyses: estimates for the placebo group, pirfenidone group and the comparison pirfenidone versus placebo together with the respective p-value for each of the 9 combinations of imputed values.

## 4.5.8.2 Fixed missing imputation between Q1 and Q3 of Placebo distribution

In another approach to evaluate the robustness of the analysis of the second endpoint to the missing at random (MAR) assumption a tipping point sensitivity analysis will be performed, where missing data of both treatment groups will be imputed by values derived from the range between lower and upper quartile (Q1 - Q3) in the Placebo group at each visit. The aim of the tipping point approach is to assess how severe departures from MAR could be in order to reverse conclusions from the analysis of secondary endpoint under different assumptions for the decline after withdrawal of the randomized treatment.

100 datasets with imputed values will be created for each treatment group. For the first dataset missing values in the respective treatment group will be imputed by the lower quartile (Q1) of placebo group within each visit. In the second dataset, the missing values will be imputed by Q1 plus the amount of  $0.01 \times (Q3 - Q1)$ . The value added to Q1 will be increased within each subsequent dataset by another amount of  $0.01 \times (Q3 - Q1)$ , so that in the last of the 100 dataset the amount of Q3 from the placebo group will be imputed for missing values.

Pirfenidone — F. Hoffmann-La Roche Ltd
Then, for each of the 10000 combinations of datasets the decline in FVC (mL) at week 24 will be estimated from a random slope model This model will include fixed effects for the stratifying variables concomitant use of MMF and presence/absence of IPAF and treatment-by time-interaction. Random effects will be included for both time and intercept.

The difference between treatment groups will be calculated together with the respective p-value.

A heat map displaying positive and negative outcome based on the p-values for the comparison pirfenidone versus placebo with green and red colors (green: < 0.05, red: > 0.05) will be provided to illustrate the outcome of this analysis graphically. The robustness of the results will be discussed based on the magnitude of deviations from MAR required to change the results.

# 4.5.8.3 Tipping point analysis with shifts

An additional approach is to evaluate the robustness of the analysis of the secondary endpoint to the missing at random (MAR) assumption by performing a tipping point sensitivity analysis using the Multiple Delta Adjustment Method.

As a first step non-monotone missing data will be imputed 100 times using MCMC (Markov Chain Monte Carlo) to generate 100 data sets of longitudinal spirometry data (FVC [mL]) with monotone missingness pattern (PROC MI). Such a missingness pattern is the pre-requisite for subsequently applying sequential imputation and means that once a patient has a missing FVC value at a particular time point, FVC values at all subsequent time points also have missing values. The seed in PROC MI number will be set to 1234.

Once the monotone missing pattern has been created, the tipping point analysis for the longitudinal FVC data will be based on the Multiple Delta Adjustment Method. Data in each of the 100 generated datasets with the monotone missingness pattern will be imputed once by using sequential regression. A delta adjustment will be added to each imputed value. The value of each delta adjustment will be given by shift parameters  $S_1$  and  $S_2$  for the 2 treatments.

For patients with more than one monotone missing visit, multiple adjustments must be applied and since the imputation method is sequential, the effect of the adjustments is cumulative. S1 and S2 therefore represent the slope of a linear adjustment over time. This step will be repeated for a variety of combinations of S1 and S2.

For each combination of shift values S1 and S2 the 100 complete data sets will be analyzed using the statistical model as described above. The estimate of treatment difference at week 24 will be derived. Rubin's rules (16) will be used to combine the results from the analyses for each pair of S1 and S2 (PROC MIIANALYZE). Point estimates for the comparison pirfenidone versus placebo and respective p-values will be reported for selected combinations of S1 and S2 in a cross-table.

The following combinations of S1 and S2 will be applied:

Pirfenidone — F. Hoffmann-La Roche Ltd

- S1 (Pirfenidone): -130, -125,-120,-115,-110,-105,-100,-95,-90,-85,-80,-75,-70,-65,-60,-55,-50,-45,-40,-35,-30,-25,-20,-15,-10,-5,0, 5, 10
- S2 (Placebo): -40,-35,-30,-25,-20,-15,-10,-5,0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 65, 70, 75, 80, 85, 90, 95, 100, 105, 110, 115, 120.

A heat map displaying positive and negative outcome based on the p-values for the comparison pirfenidone versus placebo with green and red colors (green: < 0.05, red: > 0.05) will be provided to illustrate the outcome of this analysis graphically. The robustness of the results will be discussed based on the magnitude of deviations from MAR required to change the results (Rubin, 1987). Pharmacokinetic and Pharmacodynamic Analyses

No pharmacokinetic or pharmacodynamic analyses are planned for this study.

#### 4.6 SAFETY ANALYSES

All safety analyses of data from the double-blind treatment period will be based on the safety population, i.e., the safety population will include all randomized patients who received at least one dose of trial treatment, with patients grouped according to treatment received. Safety data from the follow-up period will be summarized based on the safety follow-up population.

The safety objective for this trial is to evaluate the safety of pirfenidone vs. placebo.

No formal statistical testing will be performed for safety parameters.

Data collected during the 12-month safety follow-up will be analyzed separately (see section 4.7).

The safety analysis will involve investigating the nature, frequency, severity, and timing of treatment-emergent adverse events. The specific parameters that will be investigated include all adverse events, adverse events Grade ≥3 according to the NCI CTCAE version 4.03, adverse events of special interest, and serious adverse events. The primary interest in this trial will be adverse events Grade ≥3 related to pirfenidone or placebo.

Prior to the first administration, only serious adverse events caused by a protocol-mandated intervention will be recorded. These adverse events will be listed.

The incidence, type, and severity of adverse events will be summarized according to the primary System Organ Class (SOC) and within each SOC, by the Medical Dictionary for Regulatory Activities (MedDRA) version 20.1 or higher preferred term.

Adverse events Grade ≥3, adverse events of special interest, and serious adverse events will be analyzed in a similar way to all adverse events.

Pirfenidone — F. Hoffmann-La Roche Ltd

Descriptive statistics will be presented for dose modifications and treatment interruptions. Adverse events leading to treatment interruption or dose modification will also be summarized.

Laboratory parameters including hematology and the chemistry panel will be presented in shift tables of NCI-CTCAE version 4.03 grade at baseline vs. worst grade during treatment period. The laboratory parameters will be presented according to means, standard deviation, minimum, and maximum. Selected laboratory parameters will be also graphically presented over time. Liver abnormalities for the parameters total bilirubin, alkaline phosphatase, ALAT (SGPT) and ASAT (SGOT)) will be also presented.

The results from the 12-lead ECGs will be summarized and presented.

# 4.6.1 <u>Exposure of Study Medication</u>

All analyses described in this section refer to the data collected in the drug-log for the double-blind randomized treatment period. Unknown doses will be excluded from the exposure analyses.

#### 4.6.1.1 Treatment duration

Summaries of dosing, treatment duration, dose interruptions or reductions during the randomized double-blind treatment period will be provided for each treatment arm separately.

The overall treatment duration (weeks), including and excluding dose interruptions, will be summarized descriptively by treatment arm. The overall treatment duration including dose interruptions will be defined as follows:

[Date of last positive dose of randomized treatment received (pirfenidone/placebo) – date of first intake of randomized treatment) + 1)] / 7.

The overall treatment duration excluding dose interruptions will be derived from the treatment administration panels using the time windows described above, considering only days on treatment. i.e. positive dose.

Details on treatment administration, reductions or interruptions will be listed.

#### 4.6.1.2 Doses and Dose modifications or interruptions

The total dose (mg), the average daily dose (mg/d) and the last dose administered (mg/d) will be presented descriptively for each of the study treatments.

The average daily dose will be calculated by summing up the number of capsules taken, divided by the overall treatment duration including dose interruptions as defined above.

Numbers and proportions of patients with at least one dose modification, or drug interruption, will be presented for each treatment arm separately. Numbers and proportions of patients with 1, 2, 3 or more dose modifications, or treatment interruptions, will be given.

Pirfenidone — F. Hoffmann-La Roche Ltd

The total number of dose modifications, reductions or treatment interruptions, will be presented together with numbers and frequencies of reasons for dose modification, reduction or treatment interruption.

Dose modifications, reductions or treatment interruptions will be presented as given in the drug logs dose strength and number of capsules taken.

In addition, dose intensity will be analyzed descriptively by treatment arm over time. For calculation of dose intensities, the time from first administration of randomized treatment to the end date of randomized treatment will be considered. The following formula will be used for calculation:

Dose intensity (DI) = (total dose received / total dose planned)\*100.

# 4.6.2 Adverse Events

Verbatim descriptions of adverse events (AEs) will be mapped to a preferred term (PT) and system organ class (SOC) using the Medical Dictionary for Regulatory Agencies (MedDRA®). MedDRA version 20.1 or above and related SMQ lists will be used for coding.

AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03. For AEs of varying severity, the most severe grade as documented on the eCRF will be used in the summaries. An AE will be considered severe if the most extreme grade will be larger or equal to 3.

After informed consent has been obtained but prior to initiation of trial treatment, only serious adverse events caused by a protocol-mandated intervention (e.g. invasive procedures such as biopsies, discontinuation of medications) should be reported. All adverse events will be reported until 28 days after the last dose of study drug. After this period, the Investigator should report any SAEs that are believed to be related to prior study drug treatment.

For safety analysis of the double-blind treatment period treatment-emergent adverse events (TEAEs) will be defined as:

• AEs that started or worsened on or after first intake of randomized treatment until last positive dose of randomized treatment + 28 days

Adverse events that are reported after informed consent but before the first intake of randomized treatment will be considered as non-treatment-emergent AEs. These might include AEs that occur during the screening period.

Post-treatment AEs are not expected to occur, but will be defined as AEs that are reported more than 28 days after the last dose of randomized treatment for patients who do not enter the 12-month safety follow-up period. Those AEs will be listed.

Pirfenidone — F. Hoffmann-La Roche Ltd

The analysis of AEs within the framework of the primary study analysis will focus on treatment-emergent AEs (TEAE).

An overview of patient safety profile will present the number and proportion of patients in each treatment arm experiencing:

- Any and any related treatment-emergent adverse events (TEAE)
- Any and any related serious treatment-emergent adverse events (serious TEAE)
- Any and any related severe treatment-emergent adverse events (TEAEs ≥ Grade 3)
- Any and any related TEAE of special interest (AESI). Adverse events of special interest for this trial include the following:

Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's law: [ALT or AST >3 x ULN + total bilirubin >2 x ULN]

- Any and any related hepatic side effects: elevations in ALT and AST >3 × ULN at the same timepoint in the study.
- Any and any related gastrointestinal (GI) disorder (MedDRA SOC: GI Disorders)
- Any and any related photosensitivity (MedDRA Preferred terms Nodular rash, Photodermatosis, Photosensitivity reaction, Pruritus, Pruritus generalized). Potential updates in those terms will be needed in case the MedDRA version changes.
- Any and any related rash (MedDRA Preferred terms Rash, Rash erythematous, Rash generalized, Rash macular, Rash maculo-papular, Rash papular, Rash pruritic, Solar dermatitis, Solar urticarial, , Sunburn, Erythema, Dry skin). Potential updates in those terms will be needed in case the MedDRA version changes.
- Angioedema (MedDRA preferred term Angioedema).
- Dizziness (MedDRA preferred term Dizziness).
- Fatigue (MedDRA preferred term Fatigue).
- Weight loss (MedDRA preferred term Weight loss).
- Increase in QT interval: In the event of a QTcF interval of >500 ms or an increase from baseline of >60 ms, a repeat ECG must be obtained within 24 hours.
- Any and any related TEAE leading to death
- Any and any related TEAE leading to treatment discontinuation

Pirfenidone — F. Hoffmann-La Roche Ltd

- Any grade 3-4 laboratory liver test results
  - o ASAT (SGOT) results
  - o ALAT (SGPT) results
  - o alkaline phosphatase results
  - o total bilirubin results

The incidence of TEAEs, related TEAEs, non-serious TEAEs, serious TEAEs, related serious TEAEs, grade 3-5 TEAEs and TEAEs leading to treatment discontinuation, dose modification or death will be summarized by treatment arm, by system organ class (SOC) and preferred term (PT) on the basis of the safety population. Frequencies and percentages of patients experiencing (at least) one event in the respective category will be presented by decreasing frequencies. If patients have more than one AE within a SOC or PT they will be counted only once for the respective SOC or PT. Additionally the total numbers of TEAEs will be provided for each SOC and overall.

Similar summary presentations will be provided for the incidence of TEAEs leading to dose reduction and drug interruption and TEAEs leading to hospitalization.

Non serious Treatment-emergent Adverse Events with >5% frequency will be also presented by SOC and PT. In addition, Serious Treatment-emergent Adverse Events, Fatal serious TEAEs and serious TEAEs related to pirfenidone or placebo will be presented in the same table by SOC and PT.

A summary table presenting the numbers and frequency of patients with TEAEs by most extreme CTCAE Grade (Grade 1, Grade 2, Grade 3, Grade 4 and Grade 5) will be provided for each SOC and PT by treatment arm. In case the most extreme intensity is missing, it will be replaced by the initial intensity. If both most extreme and initial intensity are missing, the AE will be included in the Grade ≥3 category and a category for "missing" will be added.

Further, Kaplan-Meier curves for time to onset of first adverse event of the most relevant related TEAEs will be provided by treatment arm when the number of events are enough to do the analyses. These will include the following PTs or groups of AEs: Nausea, Diarrhoea, Weight decreased, Fatigue, Decreased appetite, and photosensitivity, or rash. In addition, the analysis will be done for the SOC GI.

All adverse event data will be listed by patient number and study day of onset including a flag variable for identifying the period of the event (double-blind treatment period or safety follow-up period). If the AE does not belong to any of the periods, the period flag will be missing.

In addition, for regulatory purpose two additional tables will be provided:

Pirfenidone — F. Hoffmann-La Roche Ltd

# <u>Frequency of adverse drug reactions occurring in patients treated with Esbriet</u> (Pirfenidone) in clinical trials

TEAEs from day 1 of dosing until 168 days for MA39189 will be compared with the data from the phase III studies CAPACITY1 and 2 and ASCEND (restricted to first 168 days after first dose). The frequency of patients with related AEs (ADR) will be presented by System Organ Class and will be classified by their occurrences into

- Very common ((>=10% incidence rate)
- common ((>= 1% to <10% incidence rate)
- uncommon (>= 0.1% to <1% incidence rate)
- rare (>= 0.01% to <0.1% incidence rate)

Patients who withdrew from treatment during first 168 days of dosing will be censored at day of withdrawal for this analysis.

#### Rates of Adverse events per 100 patient years

TEAEs and SAEs from day 1 of dosing until 168 days for MA39189 will be compared with the data from the registrational phase III studies in IPF patients CAPACITY1 and 2 and ASCEND (restricted to first 168 days after first dose). The following parameters will be displayed in this analysis:

- duration of study in patient years (PY), calculated as sum of all patient's observation times).
- number of patients with at least one event,
- number of all events, defined as all AEs from all patients with onset date during observation time period
- rate of events per 100 PYs observation time, calculated as [number of events/duration] \* 100
- 95% CI for this rate with
  - o Lower limit =  $100*[number of events z_{1-\alpha/2}* SQRT(number of events)]/duration$
  - o Upper limit = 100\*[number of events +  $z_{1-\alpha/2}$ \* SQRT(number of events)]/duration

where  $z_{1-\alpha/2}$  is the 1- $\alpha/2$  quantile of the standard normal distribution.

Patients who withdrew from treatment during first 168 days of dosing will be censored at day of withdrawal for this analysis. The analysis will be repeated for all TEAEs/SAEs from first day of dosing until 28 days of last dose, irrespective of the different study durations for MA39189 versus the phase III studies.

# 4.6.3 Deaths

Numbers and frequencies of deaths during double-blind period occurring until 28 days after the last dose of double-blind treatment will be presented by treatment arm. Deaths occurring more than 28 days after last dose for patients who did not enter the safety-follow-up period will also be presented separately.

Pirfenidone — F. Hoffmann-La Roche Ltd

All information associated with deaths collected in eCRF panel on study discontinuation will be listed. A flag variable will be included in the listing specifying the study period when the death occurred.

# 4.6.4 Laboratory Data

All of the laboratory tests will be conducted by the trial site's local laboratory.

All parameters will be graded according to NCI CTCAE (CTEP 2010), version 4.03, if applicable. Laboratory parameters that cannot be graded according to the corresponding NCI CTCAE version 4.03 will be assessed with respect to normal range (low, normal, high).

Laboratory parameters including hematology and the chemistry panel will be presented in shift tables of NCI-CTCAE version 4.03 grade at baseline versus worst grade during randomized double-blind treatment period. The laboratory parameters will be presented according to means, standard deviation, minimum, and maximum. Selected laboratory parameters will be also graphically presented over time.

The following laboratory samples will be collected:

- Hematology: white blood cell (WBC) count, red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, differential count (neutrophils, eosinophils, basophils, monocytes, lymphocytes, other cells).
- Chemistry panel (serum or plasma): sodium, potassium, chloride, bicarbonate, glucose, blood urea nitrogen (BUN) or urea, creatinine, total protein, albumin, phosphorus, calcium, total and direct bilirubin, alkaline phosphatase, ALT, AST, uric acid, lactate dehydrogenase (LDH).

Clinical laboratory values will be presented separately for CTCAE-gradable and non-CTCAE gradable parameters by laboratory panel (hematology, serum chemistry). For laboratory analyses, visits will be assigned to visit windows as described in <a href="Section 4.10">Section 4.10</a>. This will also be valid for possible unscheduled visits. In case that multiple evaluable assessments occur within the same visit, the nearest to midpoints value will be used for analyses.

The following summaries will be prepared:

For each laboratory parameter, descriptive statistics of laboratory values at each scheduled visit (derived as described above), and absolute changes from baseline to post-baseline will be presented by treatment arm.

Shift tables presenting categorical changes in CTCAE grade from baseline to worst grade recorded during the double-blind period, in the indicated direction, will be provided for CTCAE-gradable parameters by treatment arm. If no CTCAE grade is available for a specific laboratory variable, shift tables will present worst changes with respect to normal range category (low, normal, high).

Pirfenidone — F. Hoffmann-La Roche Ltd

Liver abnormalities (total bilirubin, alkaline phosphatase, ALAT (SGPT), ASAT (SGOT)) of Grade 3 and 4 will be presented showing numbers and percentages of patients for each parameter separately. Line graphs of liver parameters will be provided.

## 4.6.5 Vital Signs

Vital signs will include measurements of respiratory rate (breaths/min), pulse rate (beats/min), and systolic and diastolic blood pressures (mmHg) while the patient is in a seated position, temperature (C) and weight (kg). Vital signs will be assigned to visit windows as per <a href="Section 4.10">Section 4.10</a>. Descriptive statistics will be used to summarize vital signs data at baseline and at each scheduled post-baseline visit, and for the absolute change from baseline to each scheduled post-baseline visit by treatment arm during double-blind period.

#### 4.6.6 ECG

Single ECG recordings will be obtained at specified time points, as outlined in the Schedule of Assessments (see <u>Appendix 2</u>), and may be obtained at unscheduled time points as indicated.

The following should be recorded in the appropriate eCRF: heart rate (beats/min), RR interval (msec), QRS interval (msec), PR duration (msec), uncorrected QT interval (msec), and the QTcF based on the machine readings of the individual ECG tracings. Any morphologic waveform changes or other ECG abnormalities must be documented on the eCRF. If considered appropriate by the Sponsor, ECGs may be analyzed retrospectively at a central laboratory.

QTcF values of the safety population will be assigned to the following intervals: < 500 ms, 500–550 ms, and > 550 ms. Numbers and percentages of patients with their maximum QTcF interval category will be summarized by treatment arm over time. Absolute changes from the Baseline to each post-baseline visit in QTcF values will be categorized to < 31 ms, 31–60 ms, and > 60 ms. Numbers and percentages of patients in each category will be presented by treatment arm for each post-baseline visit or treatment discontinuation. Planned visits will be used for presentations.

Descriptive statistics for heart rate, RR interval, QRS interval, PR duration, uncorrected QT interval, and the QTcF will be presented for each visit by treatment arm.

A listing containing ECG data will be presented.

#### 4.7 SAFETY FOLLOW-UP ANALYSES

Data collected during the safety- follow-up period will be analyzed in the following way.

Adverse events during the 12-month safety follow-up period for pirfenidone treatment will be defined as:

 AEs that started or worsened on or after the date of safety follow-up period start until the end of the safety follow-up.

Pirfenidone — F. Hoffmann-La Roche Ltd

The safety follow-up population will be used for these analyses.

Summary tables for the incidence of AEs, related AEs, serious AEs, related serious AEs, severe AEs and severe related AEs will be summarized by system organ class (SOC) and preferred term (PT). Frequencies and percentages of patients experiencing (at least) one event in the respective category will be presented by decreasing frequencies. If patients have more than one AE within a SOC or PT they will be counted only once for the respective SOC or PT. Additionally, the total numbers of AEs will be provided for each SOC and overall. As with the end of the double-blind treatment period, an overview of safety will also be presented.

Pirfenidone exposure during safety-follow-up will be analyzed in a similar fashion as described in Section 4.7.1 with regard to treatment duration and amount of drug intake.

Data of laboratory assessments (AST, ALT, bilirubin, and alkaline phosphatase) and vital signs during safety-follow-up period will be analyzed in a similar fashion as described in Section 4.7.4 and Section 4.7.5.

Data will be presented by randomized treatment labeled as 'Randomized Pirfenidone' and 'Randomized Placebo'.

#### 4.8 MISSING DATA

With exception of the tipping point analysis described in section 4.5.8, missing data will not be imputed. Other exceptions will be made for the data related to adverse events and concomitant medications as described below.

For adverse events, missing start dates will only be imputed for determination of whether the adverse event is considered to be treatment-emergent or not.

Incomplete or missing onset dates will be imputed to the earliest date possible (using any reliable portions of the onset date that are available). The onset day is considered unreliable if the month or year portions of the date are missing.

In case the month portion of the AE start date is missing, the AE start date will be imputed to the earliest day possible by using the following principles:

- If Treatment Start Date is missing, then the AE Start Date will be imputed as 01-01-YYYY or the earliest date regarding signature of informed consent, screening date or randomization date, whichever is the later one
- When the Treatment Start Date is not missing, and the years of AE Start Date and Treatment Start Date coincide, the AE onset date will be set to the Treatment Start Date
- When the Treatment Start Date is not missing, and the years of the AE Start
  Date and the Treatment Start Date do not coincide, then the AE Start Date will be
  imputed as 01-01-YYYY or the earliest date regarding signature of informed
  consent, screening date or randomization date, whichever is the later one

Pirfenidone — F. Hoffmann-La Roche Ltd

In case the day portion of the AE Start Date is missing, the AE Start Date will be imputed to the earliest day possible as follows:

- If the Treatment Start Date is missing, then the AE Start Date will be imputed as 01-MMM-YYYY or the earliest date regarding signature of informed consent, screening date or randomization date, whichever is the later one
- When the treatment date is not missing, and the years and months from the AE Start Date and the Treatment Start Date coincide, the AE onset date will be set to the Treatment Start Date
- When the Treatment Start Date is not missing, and AE Start Date is after the Treatment Start Date according to the given year or month, then the AE Start Date will be imputed as 01-MMM-YYYY

If the AE stop date is missing, then the event will be assumed to be ongoing and a stop date will not be imputed.

In the case the treatment end date is missing and it cannot be judged whether the event occurred during the period of Treatment Start Date to Treatment End Date plus 28 days, the AE will be considered treatment-emergent as long as it is not flagged as prior AE.

For imputation and handling of missing intensity or relationship to study medication, please see Section 4.7.2.

All other missing or incomplete adverse event data will be left as missing.

For concomitant medications, missing start or end dates will only be imputed to determine whether the medication is considered to be prior, on-treatment, post-treatment.

In general if only the day is missing from the start date then the missing day will be imputed as 01-MMM-YYYY unless the month is the same month as the start of study medication in which case the missing date will be imputed as the treatment start date.

If both the day and month are missing from the start date then the start date will be imputed as 01-JAN-YYYY.

If both the day and month are missing from the start date year is the same as treatment start date then the start date will be imputed as 'treatment start date', but if the year is after treatment start date, the start date will be imputed as 01-JAN-YYYY.

If the day, month and year are all missing from the start date then the start date will be imputed as 01-JAN for the year in which the patient was recruited to the study.

If the day, month and year are all missing from the start date then the start date will be imputed as 'treatment start date'.

Pirfenidone — F. Hoffmann-La Roche Ltd

If an incomplete stop date has both the year and month present, the day will be imputed as the last day of the month or date of discontinuation/death.

If the AE is ongoing at time of primary analysis, concomitant medication will be summarized for the double-blind treatment period and safety follow-up.

#### 4.9 VISIT WINDOWS

Visit windows for double-blind treatment period will be applied to vital signs and laboratory data and the derived visits will be used in the by-visit summarizations. If multiple observations fall within the same visit window, the observation with the nearest to midpoint value will be used in the analysis, if not stated otherwise. If subjects discontinue from the double-blind treatment period early the data will be assigned to the early discontinuation visit. The date of early discontinuation will be considered as the target date.

The "Baseline" visit is a derived data point to identify baseline values which are used to calculate the change from baseline values. Baseline is defined in Section 4.2.2.

The End of Treatment [EOT] visit will either be a copy of early discontinuation records for patients who prematurely discontinued double-blind treatment period or Week 24 records for patients who completed the double-blind treatment period.

Table 2 Visit Windows

| Analysis Visit [AVISITN] | Target Day | Analysis Window (scheduled Study Days) |
|---|---|---|
| Baseline [0] | 1 | Last valid assessment prior to first intake of randomized study drug (pirfenidone/placebo). |
| | | Generally, it is assumed that measurements referring to the Day 1 (Week 1) visit have been performed before randomized study drug (pirfenidone/placebo) was given. |
| Week 4 [4] | 28 | One day after first dose of randomized treatment to 42 |
| Week 8 [8] | 56 | 43 to 70 |
| Week 12 [12] | 84 | 71 to 98 |
| Week 16 [16] | 112 | 99 to 126 |
| Week 20 [20] | 140 | 127 to 154 |
| Week 24 [24] | 168 | 155 to a maximum of 195 if the patient did not early discontinued. |

Pirfenidone — F. Hoffmann-La Roche Ltd

| Early discontinuation [25] | Not applicable | As occurred |
|---|---|---|
| End of treatment (EOT) [26] | Not applicable | As occurred |
| Follow-up visit (FUP1) [27] | Not applicable | As occurred |
| Safety follow-up<br>visits(SFUP) [28] | Not applicable | As occurred: Month 1 to 6: Monthly visits Month 7 to 12: Approximately every 3 months |
| Additional Safety follow-up visit [29] | Not applicable | As occurred:<br>up to 12 months plus 28 days |

#### 4.10 INTERIM ANALYSES

An independent Data Monitoring Committee (iDMC) will review safety data and advise on trial conduct at least three times during the trial. A first meeting is planned 6 months after start of recruitment, and subsequently at 12 and 18 months. Additional ad hoc meetings or data reviews can be requested at any time by the iDMC or the Sponsor, if warranted. The iDMC will be an independent body who will recommend to continue, modify or stop the trial at each meeting. The procedures that will be used by the iDMC will be detailed in an iDMC charter.

No formal interim analyses for efficacy are planned.

### 4.11 BIOMARKER ANALYSES

Certain biomarkers may be differentially expressed in patients with unclassifiable ILD and may change as a result of pirfenidone treatment (e.g., possibly cytokines, chemokines, and other cellular and molecular markers of lung injury and fibrosis). The blood biomarker samples that are being obtained for this trial may help identify the serum and plasma proteins or blood ribonucleic acid (RNA) biomarkers related to disease progression and/or may be used to assess their response to pirfenidone therapy.

Transcriptomic and protein markers associated with the molecular pathways and cellular processes of lung injury and fibrosis will be measured. This may include, but is not restricted to, measurement of CCL18, MMP7, CXCL13, and COMP.

Serum, plasma, and whole blood (for RNA analysis) samples will be acquired at baseline, Week 4, Week 12, Week 24, and at the Early Treatment Discontinuation Visit (see the Schedule of Assessments, <u>Appendix 2</u>).

Optional Research Biosample Repository (RBR) whole blood samples for deoxyribonucleic acid (DNA) extraction, described in Section 4.5.8 of the protocol, will also be collected at baseline to examine genetic polymorphisms and their potential role in the pathogenesis and associated clinical outcomes of unclassifiable ILD.

Pirfenidone — F. Hoffmann-La Roche Ltd

Biomarkers associated with fibrosis and ILD will be evaluated in plasma, serum, and whole blood ribonucleic acid (RNA) and deoxyribonucleic acid (DNA) samples.

Analyses on biomarker data will not be in the scope of this SAP, but will be planned and described separately.

Pirfenidone — F. Hoffmann-La Roche Ltd

# **REFERENCES**

Antoniou KM, Margaritopoulos GA, Tomassetti S, Bonella F, Costabel U, Poletti V. Interstitial lung disease. Eur Respir Rev 2014;23:40–54.

Khanna D, Albera C, Fischer A, et al. An open-label, phase II study of the safety and tolerability of pirfenidone in patients with scleroderma-associated interstitial lung disease: the LOTUSS trial. J Rheumatol 2016;epub.

Collard HR, Ryerson CJ, Corte TJ, et al. Acute exacerbation of idiopathic pulmonary fibrosis. An international working group report. Am J Respir Crit Care Med 2016;194:265–75.

Ryerson CJ, Urbania TH, Richeldi L, et al. Prevalence and prognosis of unclassifiable interstitial lung disease. Eur Respir J 2013;42:750–7.

Fischer A, Brown KK, du Bois RM, et al. Mycophenolate mofetil improves lung function in connective tissue disease-associated interstitial lung disease. J Rheumatol 2013;40:640–6.

Eakin EG, Resnikoff PM, Prewitt LM, et al. Validation of a new dyspnea measure: the UCSD Shortness of Breath Questionnaire. University of California, San Diego. Chest. 1998 Mar;113(3):619-24.

Ries AL, Minimally clinically important difference for the UCSD Shortness of Breath Questionnaire, Borg Scale, and Visual Analog Scale. COPD. 2005 Mar;2(1):105-10.

Rubin, DB. Multiple Imputation for Nonresponse in Surveys New York John Wiley and Sons 1987

Jones PW, Quirk FH, Baveystock CM, The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7.

Nishimura K, Tsukino M, Hajiro T, Health-related quality of life in patients with chronic obstructive pulmonary disease. Curr Opin Pulm Med. 1998 Mar;4(2):107-15.

St. George's Respiratory Questionnaire: http://www.healthstatus.sgul.ac.uk/sgrq

S S Birring, B Prudon, A J Carr, S J Singh, M D L Morgan, I D Pavord, Development of a symptom specific health status measure for patients with chronic cough: Leicester Cough Questionnaire (LCQ). Thorax 2003;58:339-343.

Pirfenidone — F. Hoffmann-La Roche Ltd

# Appendix 1 PROTOCOL SYNOPSIS

TITLE: MULTICENTER, INTERNATIONAL, DOUBLE-BLIND, TWO-

ARM, RANDOMIZED, PLACEBO-CONTROLLED PHASE II

TRIAL OF PIRFENIDONE IN PATIENTS WITH

**UNCLASSIFIABLE PROGRESSIVE FIBROSING ILD** 

PROTOCOL MA39189

**NUMBER:** 

**VERSION NUMBER:** 3.0

**EUDRACT NUMBER:** 2016-002744-17

**IND NUMBER:** 67284

**TEST PRODUCT:** Pirfenidone (RO0220912)

PHASE:

**INDICATION:** Fibrotic interstitial lung disease of unknown origin

**SPONSOR:** F. Hoffmann-La Roche Ltd

#### **Objectives and Endpoints**

This trial will evaluate the efficacy and safety of pirfenidone in patients with fibrosing interstitial lung disease (ILD) who cannot be classified with moderate or high confidence into any other category of fibrosing ILD by multidisciplinary team (MDT) review ("unclassifiable" ILD).

#### **Efficacy Objective**

The primary efficacy objective for this trial is to evaluate the effect of pirfenidone vs. placebo on lung function parameters on the basis of the following endpoint:

• Rate of decline in forced vital capacity (FVC) measured in mL by daily handheld spirometer over the 24-week double-blind treatment period.

#### **Safety Objective**

The safety objective for this trial is to evaluate the safety of pirfenidone vs. placebo on the basis of the following endpoints:

- Nature, frequency, severity, and timing of treatment-emergent adverse events
- Dose reductions and treatment interruptions
- Clinical laboratory test results
- 12-lead electrocardiograms (ECGs)
- Withdrawals from trial treatment or trial discontinuations.

Pirfenidone — F. Hoffmann-La Roche Ltd

#### **Exploratory Objective**

One exploratory objective for this trial is to evaluate the role of MMF (mycophenolate mofetil/sodium or mycophenolic acid) treatment in ILD on the basis of the following endpoint:

 Efficacy and safety data from subgroups of patients who did or did not receive MMF treatment.

In addition, exploratory biomarkers associated with fibrosis and ILD will be evaluated in plasma, serum, and whole blood ribonucleic acid (RNA) and deoxyribonucleic acid (DNA) samples.

#### **Trial Design**

#### **Description of Trial**

This is a multicenter, international, double-blind, two-arm, randomized, placebo-controlled Phase II trial in patients with fibrosing ILD who cannot be classified with moderate or high confidence into any other category of fibrosing ILD by MDT review ("unclassifiable ILD"). Patients will be randomized in a 1:1 ratio, on a double-blind basis using a stratified algorithm, to receive either pirfenidone (801 mg three times daily [TID]) or placebo. The randomized patients will be stratified by concomitant MMF treatment (yes/no), the presence/absence of interstitial pneumonia with autoimmune features (IPAF) as defined by the MDT.

Most established MDTs have access to clinical, radiologic, and pathology expertise, and should have a sufficient case load of ILDs per year. Access to rheumatology expertise will be at the discretion of the MDT.

In total, approximately 90 clinical centers (sites) in Australia, Europe, the Middle East, and North America are expected to enroll approximately 250 patients. Patients who are withdrawn from the trial will not be replaced. The trial design is represented in

Appendix 3 PRO Questionnaires

After discussing the risks and benefits of the trial with the investigator and providing informed consent, patients will be required to taper and/or discontinue all prohibited medications (Section 4.4.2 of the CSP) in the 28 days prior to the start of screening during the washout period. If a prohibited medication must be tapered, the process must start early enough so that the patient discontinues the medication in the 28 days prior to the start of screening. After completing the washout period, patients will enter screening, which lasts up to 21 days. During screening, patients will be evaluated for eligibility based on the inclusion and exclusion criteria. Patients not taking a prohibited medication will forgo the washout period and directly enter screening.

At the end of screening, patients will be randomized (Day 1) to receive either pirfenidone or placebo (1:1 ratio).

Following treatment initiation, the daily dosage will be titrated to the full dosage of nine capsules per day over a 14-day period. After the titration period, trial treatment will continue through Week 24 and monitoring will be conducted by trial visits. Patients should remain on a stable maintenance dose for the duration of the treatment period unless the dose is reduced or dosing is interrupted to manage an adverse event. Any patient with an actual or anticipated interruption of trial treatment for a period of ≥28 consecutive days will be reported by telephone to Roche's medical monitor or designee to discuss the circumstances of the case. Once the patient restarts trial treatment, the

Pirfenidone — F. Hoffmann-La Roche Ltd

dose must be re-titrated over 14 days. A Follow-up Visit will occur 28 days after the end of the 24-week double-blind treatment period.

After completion of the double-blind treatment period and the Follow-up Visit at Week 28, the Sponsor will offer the possibility to the patients to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. During the safety follow up period, the patients should be evaluated by the investigator initially at monthly visits during the first 6 months and subsequently at each visit occurring approximately every 3 months thereafter. A final Follow-up Visit will be performed at the end of the safety period, 28 days after the last open-label dose.

Table 1 Titration Schedule

| Treatment Days | Dosage |
|-------------------|---------------------------------------------|
| Days 1 through 7 | One capsule three times daily with meals |
| Days 8 through 14 | Two capsules three times daily with meals |
| Day 15 onwards | Three capsules three times daily with meals |

The Sponsor will provide trial treatment on a double-blind basis. The design that will be utilized in this trial is shown in Appendix 3 PRO Questionnaires below.

Figure 1 Trial Schema



<sup>&</sup>lt;sup>1</sup> Patients will be required to taper and/or discontinue all prohibited medications in the 28 days prior to the start of screening during the washout period. Patients not taking a prohibited medication will forgo the washout period and directly enter screening.

D=Day; ICF=informed consent form

#### Pirfenidone — F. Hoffmann-La Roche Ltd

<sup>&</sup>lt;sup>2</sup> Informed consent must be documented before any trial-specific screening procedure is performed, and may be obtained either at the Washout or Screening Visits.

<sup>&</sup>lt;sup>3</sup> After completion of the double-blind treatment period and the Follow-up Visit at Week 28, the Sponsor will offer the possibility to the patients to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. A final Follow-up Visit will be performed at the end of the safety period, 28 days after the last open-label dose.

The primary objective of this trial is to evaluate the efficacy of pirfenidone vs. placebo on lung function parameters by examining the rate of decline in FVC (measured in mL). A handheld spirometry device will be used by the patient to measure daily FVC at home. Confirmatory site (trial center) based FVC measurements will be conducted every 4 weeks (see Schedule of Assessments, <a href="Appendix 2">Appendix 2</a>). Blood samples will be obtained from patients in order to analyze clinical laboratory values and biomarkers.

#### **Number of Patients**

Approximately 250 patients with unclassifiable fibrosing ILD will be enrolled in this trial.

#### **Target Population**

#### **Inclusion Criteria**

Patients must meet the following criteria for trial entry:

- 1. Signed Informed Consent Form
- 2. Age ≥18–85 years
- 3. Able to comply with the trial protocol, according to the investigator's judgment
- 4. Confirmed fibrosing ILD which, following MDT review, cannot be classified with either high or moderate confidence as a specific idiopathic interstitial pneumonia or other defined ILD (e.g. chronic hypersensitivity or connective tissue disease-ILD [CTD-ILD])
- 5. Progressive disease as considered by the investigator using the following definition:
  - a. Patient deterioration within the last 6 months, which is defined as:
    - i. A rate of decline in FVC >5% OR
    - ii. Significant symptomatic worsening not due to cardiac, pulmonary, vascular, or other causes.
- 6. Extent of fibrosis >10% on high-resolution computed tomography (HRCT; visual scoring) within the last 12 months
- 7. FVC ≥45% of predicted value
- 8. Diffusing capacity of the lung for carbon monoxide (DLco) ≥30% of predicted value
- 9. Forced expiratory volume in 1 second (FEV₁)/FVC ratio ≥0.7
- 10. 6-minute walk distance (6MWD) ≥150 meters
- 11. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of <1% per year during the treatment period and for at least 58 days after the last dose of trial treatment:
  - a. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
  - Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives including those that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices

Pirfenidone — F. Hoffmann-La Roche Ltd

c. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

- a. With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 118 days after the last dose of trial treatment. Men must refrain from donating sperm during this same period
- b. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 118 days after the last dose of trial treatment to avoid exposing the embryo
- c. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

#### **Exclusion Criteria**

Patients who meet any of the following criteria will be excluded from trial entry:

- 1. Diagnosis with moderate or high confidence of nonspecific interstitial pneumonia (NSIP) and any ILD with an identifiable cause such as CTD-ILD, chronic hypersensitivity pneumonitis (cHP), or others
- 2. Diagnosis of idiopathic pulmonary fibrosis (IPF) independent of the confidence level
- History of unstable angina or myocardial infarction during the previous 6 months
- 4. Pregnant or lactating, or intending to become pregnant during the trial
- 5. A positive urine pregnancy test, which was confirmed with a positive serum pregnancy test. Women with a confirmed pregnancy will be excluded from trial participation and must discontinue trial treatment
- 6. Treatment with high dose systemic corticosteroids (i.e., >15 mg/d of prednisolone or equivalent), or any immunosuppressant other than MMF, at any time at least 4 weeks prior to screening. Patients being treated with MMF should be on a stable dose that is expected to remain stable throughout the trial and was started at least 3 months prior to screening
- 7. Patients previously treated with pirfenidone or nintedanib
- 8. Patients treated with N-acetyl-cysteine (NAC) for fibrotic lung disease, at any time within the 4 weeks of the screening period
- 9. Drug treatment for any type of pulmonary hypertension (e.g. sildenafil, endothelin receptor antagonist [ERA], etc.)
- 10. Participation in a trial of an investigational medical product within the last 4 weeks
- 11. Significant co-existent emphysema (extent greater than extent of fibrosis on HRCT within the last 12 months)

Pirfenidone — F. Hoffmann-La Roche Ltd

- 12. Significant other organ co-morbidity including hepatic or renal impairment
- 13. Previous intolerance or allergy to the trial treatment
- 14. Pregnant patients, or women of child-bearing potential, not using a reliable contraceptive method
- 15. Unable to provide informed written consent
- 16. Predicted life expectancy <12 months or on an active transplant waiting list
- 17. Use of any tobacco product in the 12 weeks prior to the start of screening, or any unwillingness to abstain from their use through to the Follow-up Visit
- 18. Illicit drug or alcohol abuse within 12 months prior to screening, according to the investigator's judgment
- 19. Planned major surgery during the trial
- 20. Hypersensitivity to the active substance or to any of the excipients of pirfenidone
- 21. History of angioedema
- 22. Concomitant use of fluvoxamine
- 23. Clinical evidence of any active infection which according to the investigator's judgment may interfere with trial conduct, measurement of pulmonary function, or impact the course of the ILD
- 24. Any history of hepatic impairment, elevation of transaminase enzymes, or the confirmation of any of the following liver function test (LFT) criteria above the specified limits:
  - a. Total bilirubin above the upper limit of normal (ULN)
  - b. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 × ULN
  - c. Alkaline phosphatase >2.0 × ULN.
- 25. Creatinine clearance <30 mL/min, calculated using the Cockcroft-Gault formula
- 26. Any serious medical condition, clinically significant abnormality on an ECG at screening, or laboratory test results (hematology, serum chemistry, and urinalysis) that, in the opinion of the investigator, may pose an additional risk to the patient following the administration of trial treatment
- 27. An ECG with a heart rate corrected QT interval (corrected using Fridericia's formula [QTcF]) ≥500 ms at screening, or a family or personal history of long QT syndrome.

Re-screening may be considered for patients who do not show sufficient disease deterioration in accordance to the protocol at the time of the initial screening. Rescreening is permitted if there is strong evidence of clinical worsening based on the Investigator's judgement and only upon receipt of official approval from the Study Management Team. In such cases, re-screening may be performed after a minimum of 4-weeks lapse from the initial screening date.

#### **End of Trial and Length of Trial**

After completion of the double-blind treatment period and the Follow-up Visit at Week 28, the Sponsor will offer the possibility to the patients to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. The end of the clinical trial is defined as the date when the last patient, last visit (LPLV) occurs or the date at which the last data point which is required for the statistical analysis is received, whichever is the later date. For this trial, LPLV will occur when the

Pirfenidone — F. Hoffmann-La Roche Ltd

last patient has completed the final safety Follow-up Visit, 28 days after the final openlabel dose, or when the last data point is collected in the safety follow-period.

For each patient the total length of the trial is expected to be up to a maximum of 91 weeks. The trial duration includes the washout period of up to 4 weeks, the screening period of up to 3 weeks, the double-blind treatment period of 24 weeks, the follow-up period of 4 weeks, the open-label safety follow-up period up to 12 months (52 weeks) and a final safety Follow-up Visit 4 weeks after the last dose.

# **Investigational Medicinal Products**

#### Pirfenidone and Placebo

Pirfenidone and placebo will be supplied by the Sponsor as 267 mg capsules in a bottle. For information on the formulation and handling of pirfenidone, see the Investigator's Brochure or local prescribing information for pirfenidone.

Placebo will be supplied by the Sponsor in the form of capsules with identical appearance and size as the pirfenidone capsule. The placebo capsules will contain microcrystalline cellulose.

#### **Statistical Methods**

#### **Primary Analysis**

The primary efficacy objective for this trial is to evaluate the efficacy of pirfenidone vs. placebo on lung function parameters on the basis of rate of decline in FVC in mL measured by handheld spirometry over the 24-week double-blind treatment period.

The primary analysis will be based on the intent-to-treat (ITT) population. Patients who discontinue treatment prematurely will be analyzed based on the available data. No imputation method will be applied.

The primary analysis of the primary endpoint will compare the mean FVC decline in each treatment arm using a student's t-test with a two-sided significance level  $\alpha$ =0.05. The mean FVC decline for each treatment arm will be calculated using the estimated FVC decline for each individual patient. The individual FVC decline will be estimated by applying a linear regression model to all data points collected during the 24-week double-blind treatment period.

#### **Determination of Sample Size**

The purpose of this trial is hypothesis generation regarding the efficacy of pirfenidone vs. placebo on lung function parameters on the basis of rate of decline in FVC, as measured by daily handheld spirometry.

A total sample size of approximately 250 patients is planned, and patients will be randomized in a 1:1 ratio. The randomization will be stratified by concomitant MMF treatment (yes/no), the presence/absence of IPAF as defined by the MDT.

Pirfenidone — F. Hoffmann-La Roche Ltd

The planned sample size is based on the statistical hypothesis of the primary endpoint and assumes 80% power and a two-sided significance level of 5% using a student's t-test. It is assumed, after inspection of historical data, that FVC decline in the placebo arm is 85 mL with a common standard deviation of 70 mL, which can be reduced to 60 mL with a common standard deviation of 70 mL in the pirfenidone arm. In this scenario, 125 patients per treatment arm are needed to detect this treatment effect with 80% power.

#### **Interim Analyses**

There are no planned interim efficacy analyses for this trial. Safety interim analyses will be performed at least three times during the trial, at approximately 6, 12, and 18 months after the start of recruitment.

Pirfenidone — F. Hoffmann-La Roche Ltd

# Appendix 2 Schedule of Assessments

| | Washout <sup>a</sup> | Screening | Doubl | Double-blind treatment | | | | | | Early treatment discontinuation <sup>b</sup> | Follow-<br>up <sup>u</sup> | Additional<br>safety<br>follow-up <sup>c</sup> | Additional<br>safety<br>follow-up<br>final visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day<br>Week | –50 to –22 | −21 to −1 | Randomization<br>1 | 28<br>4 | 56<br>8 | 84<br>12 | 112<br>16 | 140<br>20 | 168<br>24 | | 196<br>28 | up to 12<br>months | up to 12<br>months<br>plus 28<br>days |
| Window (days,<br>unless otherwise<br>stated) | | | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 b | ±5 | ±5 | ±5 |
| Treatment Period<br>Visit | | | | | | | | | | | | Month 1 to 6:<br>Monthly visits<br>Month 7 to12:<br>Approximately<br>every<br>3 months | |
| Informed consent d,e | х | х | | | | | | | | | | | |
| Review Eligibility<br>Criteria | | х | | | | | | | | | | | |
| Demographic data <sup>e</sup> | Х | х | | | | | | | | | | | |
| General medical history and baseline conditions <sup>e</sup> | х | х | | | | | | | | | | | |
| Vital signs <sup>f</sup> | | х | Х | х | х | Х | Х | Х | х | х | Х | х | _ |

Pirfenidone — F. Hoffmann-La Roche Ltd

| | Washout <sup>a</sup> | Screening | Doubl | Double-blind treatment | | | | | | Early treatment discontinuation <sup>b</sup> | Follow-<br>up <sup>u</sup> | Additional<br>safety<br>follow-up <sup>c</sup> | Additional<br>safety<br>follow-up<br>final visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day<br>Week | –50 to –22 | −21 to −1 | Randomization<br>1 | 28<br>4 | 56<br>8 | 84<br>12 | 112<br>16 | 140<br>20 | 168<br>24 | | 196<br>28 | up to 12<br>months | up to 12<br>months<br>plus 28<br>days |
| Window (days,<br>unless otherwise<br>stated) | | | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 b | ±5 | ±5 | ±5 |
| Treatment Period<br>Visit | | | | | | | | | | | | Month 1 to 6:<br>Monthly visits<br>Month 7 to12:<br>Approximately<br>every<br>3 months | |
| Weight | | х | | | | | | | х | х | | | |
| Height | | х | | | | | | | | | | | |
| Complete physical examination <sup>g</sup> | | х | x | | | | | | х | х | | | |
| ECG h | | х | х | | | х | | | х | х | Х | | |
| Hematology <sup>i</sup> | | х | Х | | | х | | | х | х | | | |
| Chemistry <sup>j</sup> | | х | Х | х | x <sup>k</sup> | х | x <sup>k</sup> | x <sup>k</sup> | х | х | | <b>X</b> <sup>k</sup> | |
| Pregnancy test <sup> </sup> | | х | Х | х | х | х | х | Х | х | x | | х | |

| | Washout <sup>a</sup> | Screening | Doubl | Double-blind treatment | | | | | | Early treatment discontinuation <sup>b</sup> | Follow-<br>up <sup>u</sup> | Additional<br>safety<br>follow-up <sup>c</sup> | Additional<br>safety<br>follow-up<br>final visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day<br>Week | -50 to -22 | –21 to –1 | Randomization<br>1<br>1 | 28<br>4 | 56<br>8 | 84<br>12 | 112<br>16 | 140<br>20 | 168<br>24 | | 196<br>28 | up to 12<br>months | up to 12<br>months<br>plus 28<br>days |
| Window (days,<br>unless otherwise<br>stated) | | | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 b | ±5 | ±5 | ±5 |
| Treatment Period<br>Visit | | | | | | | | | | | | Month 1 to 6:<br>Monthly visits<br>Month 7 to12:<br>Approximately<br>every<br>3 months | |
| Trial treatment administration | | | х | х | х | х | х | х | | | x <sup>m</sup> | х | |
| Spirometry (FVC, FEV <sub>1</sub> ) | | х | х | х | х | Х | х | х | х | х | | | |
| Daily spirometry (handheld device) n,o | | х | х | х | х | х | х | х | х | х | | | |
| DLco | | х | Х | | | х | | | х | х | | | |
| 6MWD p | | х | Х | | | х | | | х | х | | | |
| Leicester Cough<br>Questionnaire <sup>q</sup> | | | х | | | х | | | х | х | | | |

| | Washout <sup>a</sup> | Screening | Doubl | Double-blind treatment | | | | | | Early treatment discontinuation <sup>b</sup> | Follow-<br>up <sup>u</sup> | Additional<br>safety<br>follow-up <sup>c</sup> | Additional<br>safety<br>follow-up<br>final visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day<br>Week | -50 to -22 | -21 to -1 | Randomization<br>1 | 28<br>4 | 56<br>8 | 84<br>12 | 112<br>16 | 140<br>20 | 168<br>24 | | 196<br>28 | up to 12<br>months | up to 12<br>months<br>plus 28<br>days |
| Window (days,<br>unless otherwise<br>stated) | | | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 b | ±5 | ±5 | ±5 |
| Treatment Period<br>Visit | | | | | | | | | | | | Month 1 to 6:<br>Monthly visits<br>Month 7 to12:<br>Approximately<br>every<br>3 months | |
| UCSD-SOBQ q | | | х | | | х | | | х | х | | | |
| SGRQ q | | | Х | | | х | | | х | х | | | |
| Cough visual analog score q | | | х | | | х | | | х | х | | | |
| Serum for biomarker assessments | | | х | х | | х | | | х | х | | | |
| Plasma for biomarker assessments | | | Х | х | | х | | | х | х | | | |

| | Washout <sup>a</sup> | Screening | Doubl | Double-blind treatment | | | | | | Early treatment discontinuation <sup>b</sup> | Follow-<br>up <sup>u</sup> | Additional<br>safety<br>follow-up <sup>c</sup> | Additional<br>safety<br>follow-up<br>final visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day<br>Week | -50 to -22 | -21 to -1 | Randomization<br>1 | 28<br>4 | 56<br>8 | 84<br>12 | 112<br>16 | 140<br>20 | 168<br>24 | | 196<br>28 | up to 12<br>months | up to 12<br>months<br>plus 28<br>days |
| Window (days,<br>unless otherwise<br>stated) | | | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 b | ±5 | ±5 | ±5 |
| Treatment Period<br>Visit | | | | | | | | | | | | Month 1 to 6:<br>Monthly visits<br>Month 7 to12:<br>Approximately<br>every<br>3 months | |
| Whole blood for <i>PAX</i> gene biomarker assessment | | | х | х | | х | | | х | х | | | |
| Concomitant medications r | х | х | х | х | х | Х | х | х | х | х | х | х | х |
| Adverse events s | | х | Х | Х | х | х | х | Х | х | х | Х | Х | х |
| Whole blood sample for RBR (optional) <sup>t</sup> | | | х | | | | | | | | | | |

6MWD=6-minute walk distance; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; DLco=diffusing capacity of the lung for carbon monoxide; ECG=electrocardiogram; eCRF=electronic case report form; FEV<sub>1</sub>=forced expiratory volume in 1 second; FVC=forced vital capacity; IMP=investigational medicinal product; LDH=lactate dehydrogenase; LFT=liver function test; PRO=patient-reported outcome; RBC=red blood cell; RBR=Research Biosample Repository; SGRQ=St. George's Respiratory Questionnaire; SOBQ=Shortness of Breath Questionnaire; UCSD=University of California, San Diego; WBC=white blood cell

Notes: all assessments should be performed within 7 days of the scheduled visit, unless otherwise specified.

- <sup>a</sup> Patients will be required to taper and/or discontinue all prohibited medications in the 28 days prior to the start of screening during the washout period. Patients not taking a prohibited medication will forgo the washout period and directly enter screening.
- Patients who discontinue trial treatment prematurely will return to the site (clinic) for an Early Treatment Discontinuation Visit 28 (± 5) days after the last dose of the double-blind treatment, thus ending their participation in the trial. For patients who end their participation in the double-blind treatment period due to unblinding, they may be offered to continue into the open-label period according to the investigator's judgment. These patients will attend the Early Treatment Discontinuation Visit (28 (± 5) days after the last dose of the double-blind treatment) and on the same day begin their participation in the 12-month open-label pirfenidone safety follow-up period.
- c After completion of the double-blind treatment period and the Follow-up Visit at Week 28, the Sponsor will offer the possibility to the patients to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. During the 12-month safety follow-up period, initially, patients will be evaluated at monthly visits for the first 6 months. At the end of the first 6 months, patients will be evaluated at each site visit occurring approximately every 3 months until the end of the safety follow-up period. A final Follow-up Visit will be performed at the end of the safety period, 28 (± 5) days after the last open-label dose.
- Informed consent must be documented before any trial-specific screening procedure is performed, and may be obtained either at the Washout or Screening Visits.
- <sup>e</sup> Any procedures that were not completed during washout, must be completed at the Screening Visit.
- function Includes respiratory rate, pulse rate, and systolic and diastolic blood pressures while the patient is in a seated position, and temperature. Abnormalities observed at baseline should be recorded on the General Medical History and Baseline Conditions eCRF. At subsequent visits, new or worsened clinically significant abnormalities should be recorded on the Adverse Event eCRF. All vital sign measurements are to be obtained prior to any blood draws scheduled at the same time.

Pirfenidone — F. Hoffmann-La Roche Ltd

- Includes evaluation of the head, eyes, ears, nose, and throat, and the cardiovascular, dermatological, musculoskeletal, respiratory, gastrointestinal, genitourinary, and neurological systems. Abnormalities observed at baseline should be recorded on the General Medical History and Baseline Conditions eCRF. At subsequent visits, new or worsened clinically significant abnormalities should be recorded on the Adverse Event eCRF.
- h All ECGs are to be obtained prior to other procedures scheduled at the same time.
- Hematology includes WBC count, RBC count, hemoglobin, hematocrit, platelet count, differential count (neutrophils, eosinophils, basophils, monocytes, lymphocytes, other cells).
- <sup>j</sup> Chemistry panel (serum or plasma) includes sodium, potassium, chloride, bicarbonate, glucose, BUN or urea, creatinine, total protein, albumin, phosphorus, calcium, total and direct bilirubin, alkaline phosphatase, ALT, AST, uric acid, LDH.
- <sup>k</sup> Only LFTs (AST, ALT, bilirubin, and alkaline phosphatase) will be conducted at these visits. During the Safety Follow-up period, LFTs will be performed every month during the first 6 months and subsequently at each visit occurring approximately every 3 months thereafter, until the end of this period.
- All women of childbearing potential will have a serum pregnancy test at screening. Urine pregnancy tests will be performed at the specified subsequent visits. If a urine pregnancy test is positive, it must be confirmed by a serum pregnancy test. During the Safety Follow-up period, urine pregnancy tests will be performed every month during the first 6 months at each site visit. Urine pregnancy tests will continue to be performed on a monthly basis during the remainder of the Safety Follow-up period with patients performing the test at home (using kits provided by the site) during months where there is no site visit and at each site visit occurring approximately every 3 months. Patients will be instructed to contact the site immediately in case the result of the home pregnancy test is positive. In such cases, the patient must visit the site for a confirmatory serum pregnancy test.
- <sup>m</sup> Open-label treatment with pirfenidone will be started at this visit, if the patient requests continued treatment with pirfenidone.
- <sup>n</sup> Handheld spirometry will be conducted by the patient every day in a seated position.
- o To provide handling evaluations and quality assurance for the daily spirometer assessments, nursing visits to the patient's home (or at another suitable location) will occur at least three times during the trial, namely between Weeks 1 and 4, between Weeks 8 and 12, and between Weeks 16 and 20. Additional home nursing visits may be conducted according to the investigator's judgment.

- <sup>p</sup> 6-Minute Walk Distance (6MWD) is used to evaluate the functional capacity of patients with lung disease.
- q Questionnaires will be self-administered prior to the patient receiving any information on disease status and prior to the performance of non-PRO assessments.
- Includes any medication (e.g., prescription drugs, over-the-counter drugs, vaccines, herbal or homeopathic remedies, nutritional supplements) used by a patient from the washout period until 28 days after the last dose of trial treatment.
- s After informed consent has been obtained but prior to initiation of trial treatment, only serious adverse events caused by a protocol-mandated intervention should be reported. After initiation of trial treatment, all adverse events will be reported until 28 days after the last dose of trial treatment. After this period, all deaths, regardless of cause, should be reported. In addition, the Sponsor should be notified if the investigator becomes aware of any serious adverse event that is believed to be related to prior trial treatment. The investigator should follow each adverse event until the event has resolved to baseline grade or better, the event is assessed as stable by the investigator, the patient is lost to follow-up, or the patient withdraws consent. Every effort should be made to follow all serious adverse events considered to be related to trial treatment or trial-related procedures until a final outcome can be reported.
- <sup>t</sup> Not applicable for a site that has not been granted approval for RBR sampling.
- <sup>u</sup> If a patient discontinues the trial between weeks 24 and 28, final assessments according to the Follow-up visit for week 28 should be performed.

a.

Pirfenidone — F. Hoffmann-La Roche Ltd

# Appendix 3 PRO Questionnaires

# **Leicester Cough Questionnaire**

| ca | | | sess the impact of y<br>he response that b | | | | |
|---|---|---|---|---|---|---|---|
| 1. | In the last 2 we | eks, have you had | chest or stomach | pains as a result | of your cough? | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the time | None of the time |
| 2. | In the last 2 we | eks, have you bee | n bothered by phle | gm production wh | nen you cough? | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | Every time | Most times | Several times | Sometimes | Occasionally | Rarely | Never |
| 3. | In the last 2 we | eks, have you bee | n tired because of | your cough? | | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the tim |
| 4. | In the last 2 we | eks, have you felt | in control of your co | ough? | | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | None of the time | Hardly any of the<br>time | A little of the time | Some of the time | A lot of the time | Most of the time | All of the time |
| 5. | How often durin | ng the last 2 weeks | have you felt emb | arrassed by your | coughing? | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the time | None of the tim |
| 6. | In the last 2 we | eks, my cough has | s made me feel and | cious | | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the time | None of the time |
| 7. | In the last 2 we | eks, my cough has | s interfered with my | job, or other dail | y tasks | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the tim |
| 8. | In the last 2 we | eks, I felt that my | cough interfered wit | th the overall enjo | syment of my life | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the time |
| 9. | In the last 2 we | eks, exposure to p | aints or fumes has | made me cough | | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the tim |
| 10 | In the last 2 we | eks, has your coud | h disturbed your s | leep? | | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the time | None of the tim |
| 11 | In the last 2 we | eks, how many tim | nes a day have you | had coughing fits | s? | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | All of the time<br>(continuously) | Most times during<br>the day | Several times during<br>the day | Sometimes during the day | Occasionally through<br>the day | Rarely | None |
| 12 | In the last 2 we | eks, my cough has | s made me feel frus | | TOWNWAY CENT | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the | None of the time |

Pirfenidone — F. Hoffmann-La Roche Ltd

| | | | | | time | |
|---|---|---|---|---|---|---|
| 13.In the last 2 wee | ks, my cough has | s made me feel fed | up | | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the time |
| 14.In the last 2 wee | ks, have you suff | ered from a hoarse | voice as a resul | t of your cough? | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the time |
| 15.In the last 2 wee | ks, have you had | a lot of energy? | | | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| None of the time | Hardly any of the time | A little of the time | Some of the time | A lot of the time | Most of the time | All of the time |
| 16.In the last 2 wee | ks, have you wor | ried that your coug | h may indicate a | serious illness? | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the time |
| 17.In the last 2 wee cough? | ks, have you bee | n concerned that o | ther people think | something is wro | ng with you becar | use of your |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the time |
| 18.In the last 2 wee | ks, my cough has | s interrupted conve | rsations or teleph | none calls | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Every time | Most times | A lot of the time | Some of the time | A little of the time | Hardly any of the time | None of the time |
| 19.In the last 2 wee | ks, I feel that my | cough has annoye | d my partner, fan | nily or friends | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Every time I cough | Most times when I cough | Several times when I cough | Sometimes when I cough | Occasionally when<br>I cough | Rarely | Never |
| Thank you for comp | leting this question | onnaire. | | | | |

# Scoring

The Leicester Cough Questionnaire is a patient-reported questionnaire evaluating the impact of cough on quality of life. The questionnaire comprises 19 items and takes 5 to 10 minutes to complete. Each item assesses symptoms, or the impact of symptoms, over the last 2 weeks on a seven-point Likert scale. Scores in three domains (physical, psychological and social) are calculated as a mean for each domain (range 1 to 7). A total score (range 3 to 21) is also calculated by adding the domain scores together. Higher scores indicate better quality of life.

The scores from each of the following questions are added together to provide the mean score for each domain:

1. Physical: 1, 2, 3, 9, 10, 11, 14, 15

2. Psychological: 4, 5, 6, 12, 13, 16, 17

3. Social: 7, 8, 18, 19

Domain scores: total score from items in domain/number of items in domain (range 1–7).

Total scores: addition of domain scores (range 3–21).

Pirfenidone — F. Hoffmann-La Roche Ltd

#### UCSD-SOBQ

The University of California, San Diego-Shortness of Breath Questionnaire (UCSD-SOBQ) is a symptom-specific, 24-item, patient-self-administered questionnaire that assesses shortness of breath while doing a variety of activities of daily living.

### **UCSD MEDICAL CENTER**

#### **PULMONARY REHABILITATION PROGRAM**

#### SHORTNESS-OF-BREATH QUESTIONNAIRE

© 1995 The Regents of the University of California

Please rate the breathlessness you experience when you do, or if you were to do, each of the following tasks. **Do not skip any items.** If you've never performed a task, or no longer perform it, give your best estimate of the breathlessness you would experience while doing that activity. Please review the two sample questions below before turning the page to begin the questionnaire.

Pirfenidone — F. Hoffmann-La Roche Ltd

When I do, or if I were to do, the following tasks, I would rate my breathlessness as:

0 None at all

1

2

3

- 4 Severe
- 5 Maximum or unable to do because of breathlessness

Harry has felt moderately short of breath during the past 7 days while brushing his teeth and so circles a three for this activity.

| | | | | | | - |
|----|------------------|---|---|---|---|-----|
| 2 | Mowing the lawn0 | 1 | 7 | 3 | 4 | (5) |
| 4. | Moving the lawn | - | - | | - | |

Anne has never mowed the lawn before but estimates that she would have been too breathless to do this activity during the past 7 days. She circles a five for this activity.

When I do, or if I were to do, the following tasks, I would rate my breathlessness as:

0 None at all
1
2
3
4 Severe
5 Maximum or unable to do because of breathlessness

| 1. | At rest | 1 | 2 | 3 | 4 | 5 |
|----|----------------------------------------|---|---|---|---|---|
| 2. | Walking on a level at my own pace | 1 | 2 | 3 | 4 | 5 |
| 3. | Walking on a level with others my age0 | 1 | 2 | 3 | 4 | 5 |
| 4. | Walking up a hill 0 | 1 | 2 | 3 | 4 | 5 |
| 5. | Walking up stairs0 | 1 | 2 | 3 | 4 | 5 |
| 6. | While eating0 | 1 | 2 | 3 | 4 | 5 |
| 7. | Standing up from a chair0 | 1 | 2 | 3 | 4 | 5 |
| 8. | Brushing my teeth | 1 | 2 | 3 | 4 | 5 |
| 9. | Shaving and/or brushing my hair | 1 | 2 | 3 | 4 | 5 |

Pirfenidone — F. Hoffmann-La Roche Ltd
| 10. | Showering/bathing 0 | 1 | 2 | 3 | 4 | 5 |
|-----|---------------------|---|---|---|---|---|
|-----|---------------------|---|---|---|---|---|

When I do, or if I were to do, the following tasks, I would rate my breathlessness as:

0 None at all 1

2

3

- 4 Severe
- 5 Maximum or unable to do because of breathlessness

| 11. | Dressing0 | 1 | 2 | 3 | 4 | 5 |
|-----|------------------------------------------|---|---|---|---|---|
| 12. | Picking things up and tidying up a room0 | 1 | 2 | 3 | 4 | 5 |
| 13. | Doing the dishes | 1 | 2 | 3 | 4 | 5 |
| 14. | Sweeping/vacuuming | 1 | 2 | 3 | 4 | 5 |
| 15. | Making the bed | 1 | 2 | 3 | 4 | 5 |
| 16. | Shopping0 | 1 | 2 | 3 | 4 | 5 |
| 17. | Doing laundry | 1 | 2 | 3 | 4 | 5 |
| 18. | Washing the car | 1 | 2 | 3 | 4 | 5 |
| 19. | Mowing the lawn 0 | 1 | 2 | 3 | 4 | 5 |
| 20. | Watering the lawn0 | 1 | 2 | 3 | 4 | 5 |
| 21. | Sexual activities 0 | 1 | 2 | 3 | 4 | 5 |

Pirfenidone — F. Hoffmann-La Roche Ltd

0 None at all 1

2

3 4 Severe

5 Maximum or unable to do because of breathlessness

## How much do the following limit you in your daily life?

| 22. | Shortness of breath 0 | 1 | 2 | 3 | 4 | 5 |
|-----|--------------------------------------------|---|---|---|---|---|
| 23. | Fear of "hurting myself" by overexertion 0 | 1 | 2 | 3 | 4 | 5 |
| 24. | Fear of shortness of breath | 1 | 2 | 3 | 4 | 5 |

## **Scoring**

Twenty one items assess the severity of shortness of breath during specific activities associated with daily living if patients do not routinely perform the activity, they are asked to estimate the degree of shortness of breath anticipated. Three additional items ask about limitations due to: shortness of breath, fear of harm from overexertion and fear of shortness of breath.

Each of the 24 activities are rated on how dyspnea affects the activity on a 6-point scale: 0 = None at all to 5 = Maximal or unable to do because of breathlessness

The scores from all 24 questions are totalled to provide a score in the range 0 - 120.

Pirfenidone — F. Hoffmann-La Roche Ltd

#### **SGRQ**

The St. George's Respiratory Questionnaire (SGRQ) is an index designed to measure and quantify health-related health status in patients with chronic airflow limitations.

## ST. GEORGE'S RESPIRATORY QUESTIONNAIRE ENGLISH FOR THE UNITED STATES

#### ST. GEORGE'S RESPIRATORY QUESTIONNAIRE (SGRQ)

This questionnaire is designed to help us learn much more about how your breathing is troubling you and how it affects your life. We are using it to find out which sopests of your illness cause you the most problems, rather than what the doctors and nurses think your problems are

Please read the instructions carefully and ask if you do not understand anything.

Do not spend too long deciding about your answers.

| Before completing the rest of the questionnaire: | | | | | |
|---|---|---|---|---|---|
| Please check one box to show how you describe<br>your current health: | Verygood | Good | Fair | Poor | Very poor |

Copyright reserved P.W. Jones. PhD FRCP Professor of Respiratory Medicine, St. George's University of London, Jenner Wing, Cranmer Terrace, London SW17 ORE, UK.

USA / English version «Past three months» version Tel. +44 (0) 20 8725 5371 Fax +44 (0) 20 8725 5955

continued...

Pirfenidone — F. Hoffmann-La Roche Ltd

# St. George's Respiratory Questionnaire PART 1

| | | Pla | se chart | (√) one be | x for each qu | section. |
|---|---|---|---|---|---|---|
| | | almost<br>every<br>day | se criecii<br>several<br>days<br>a week | a few<br>days<br>a month | only with<br>respiratory | not<br>at<br>all |
| 1. | Over the past 3 months, I have coughed: | | | | | |
| 2. | Over the past 3 months, I have brought up phiegm (sputum): | | | | | |
| 3. | Over the past 3 months, I have had shortness of breath: | | | | | |
| 4. | Over the past 3 months, I have had wheezing attacks: | | | | | |
| 5. | How many times during the past 3 months have severe or very unpleasant respiratory attacks? | e you suffe | ered from | | | |
| | | | non | 3 time<br>2 time<br>1 time<br>e of the time | es 🗆 | |
| 6. | How long did the worst respiratory attack last?<br>(Go to Question 7 if you did not have a severe | attack) | | | | |
| | | 300 | | Pleas<br>eek or mo | se check (✓) | one: |
| | | | 1000 | r more da | | |
| | | | 30 | 1 or 2 day | _ | |
| | | | les | s than a da | | |
| 7. | Over the past 3 months, in a typical week, how (with few respiratory problems) have you had? | many goo | od days | | | |
| | | | | | se check (✓) | one: |
| | | | | o good day<br>2 good day | | |
| | | | | 4 good day | | |
| | | near | | ay was goo | | |
| | | 1017.00 | | ay was goo | | |
| 8. | If you wheeze, is it worse when you get up in th | e morning | 9? | | | |
| | | | | | se sheck (*) | one: |
| | | | | 36 | lo 📙 | |
| | | | | Ye | 25 | |

Pirfenidone — F. Hoffmann-La Roche Ltd

## St. George's Respiratory Questionnaire PART 2

| Linear reported transportation and the property of the propert | | | |
|---|---|---|---|
| How would you describe your respiratory condition | nr | Please | check (🗸) one |
| The mi | st import | ant problem I have | |
| | | e a lot of problems | П |
| Oduse | | me a few problems | ī |
| | | auses no problems | ī |
| | - | auses no problems | _ |
| If you have ever held a job: | | | |
| | | Please ( | check (✓) one |
| My respiratory problems made | me slop | working altogether | L |
| My respiratory problems interfere with my job | or made | me change my job | |
| My respiratory p | roblems d | lo not affect my job | |
| Section 2 | | | |
| | ake you | feel short of breath | these days. |
| These are questions about what activities usually m | | | these days. |
| These are questions about what activities usually m | och staten<br>/) the bo | nent please check<br>or that applies | these days. |
| These are questions about what activities usually m | och staten<br>/) the bo<br>to you fi | nent please oheck<br>x that applies<br>hose days: | these days. |
| These are questions about what activities usually m<br>For ea<br>(- | och staten<br>/) the bo | nent please check<br>or that applies | these days. |
| These are questions about what activities usually m<br>For ea<br>(-<br>Sitting or lying still | och staten<br>/) the bo<br>to you fi | nent please oheck<br>x that applies<br>hose days: | these days. |
| These are questions about what activities usually m For ea ( Sitting or lying still Washing or dressing yourself | och staten /) the bo to you fi | nent please check<br>x that applies<br>hese days:<br>False | these davs. |
| These are questions about what activities usually m For ea ( Sitting or lying still Washing or dressing yourself Walking around the house | och staten /) the bo to you fi | nent please check<br>x that applies<br>hese days:<br>False | these days. |
| These are questions about what activities usually m For ea (* Sitting or lying still Washing or dressing yourself Walking around the house Walking outside on level ground | och staten /) fine be to you fi | nent please check<br>x that applies<br>hese days:<br>False | these days. |
| Sitting or lying still<br>Washing or dressing yourself<br>Walking around the house | och staten /) the be to you fi | nent please check<br>x that applies<br>hese days:<br>False | these days. |
| These are questions about what activities usually m For ea (* Sitting or lying still Washing or dressing yourself Walking around the house Walking outside on level ground | och staten /) fine be to you fi | nent please oheck<br>x that applies<br>hose days: | these davs. |

## St. George's Respiratory Questionnaire

| FARTZ | | | | |
|---|---|---|---|---|
| Section 3 | | | | |
| These are more questions about your cough and sh | ortness | of breath <u>ti</u> | ese day | 15. |
| Fores | sch state | ment please | check | |
| | | x that appli | | |
| · | to you | hese days | | |
| | True | False | | |
| Coughing hurts | | | | |
| Coughing makes me fired | | | | |
| I am short of breath when I talk | | | | |
| I am short of breath when I bend over | | | | |
| My coughing or breathing disturbs my sleep | | | | |
| I get exhausted easily | | | | |
| Section 4 | | | | |
| These are questions about other effects that your re | 5.0 | . mahla | mare In- | arm one sense the |
| days. | spirator | y problema | шау па | ve on you me |
| | | 12271700 | | |
| | | | | ment, please<br>ne box that |
| | | | | these days: |
| | | 5.0 | True | False |
| My cough or breathing is emb | arrassing | in public | | |
| My respiratory problems are a nuisance to my family, fri | ends or r | eighbors | | |
| I get afraid or panic when I canno | t catch r | ny breath | | |
| I feel that I am not in control of my res | piratory | problems | | |
| I do not expect my respiratory problem | | | | |
| I have become frail or an invalid because of my re- | | 33 | | |
| The state of the s | | fe for me | | |
| Everything seems too | | 14.30 | $\overline{\Box}$ | П |
| Lifetyting seems oc | inaci o | anenon | _ | |
| Section 5 | | | | |
| These are questions about your respiratory treatme section 6. | nt. If yo | u are not re | ceiving | treatment go |
| Fo | r each st | atement, ple | ase | |
| | * (*) the | box that a | pplies | |
| | Total Action | hese days. | | |
| | | False | | |
| | True | | | |
| My treatment does not help me very much | True | | | |
| My treatment does not help me very much | True | | | |

USA/ US English version

4

continued...

Pirfenidone — F. Hoffmann-La Roche Ltd

## St. George's Respiratory Questionnaire PART 2

| Section 6 | | | | |
|---|---|---|---|---|
| These are questions about how your activities might l | be affec | ted by your i | espirato | ry problems |
| | | each stateme<br>the box tha | t apples | to you |
| | Deca | ause or your i | True | False |
| (4.6 1 6 4 4 4 | e e per | | | raise |
| I take a long time to get | | | H | H |
| I cannot take a bath or shower, or I take walk slower than other people my a | | | H | H |
| Jobs such as household chores take a long time, or I | | | $\overline{\Box}$ | |
| If I walk up one flight of stairs, I have<br>If I hurry or walk fast. I have to | - | | | |
| My breathing makes it difficult to do things such as walk up stairs, light gardening such | as weed | 100000000000000000000000000000000000000 | | |
| My breathing makes it difficult to do things such as<br>dig in the garden or shovel snow, jog or walk briskly | / (5 mile | and the second s | | |
| My breathing makes it difficult to do things<br>manual work, ride a b<br>or play | oike. run | | | |
| Section 7 | | | | |
| We would like to know how your respiratory problems | usuall | <u>y</u> affect your | daily life | 38 |
| the box that | t applies | t, please chec<br>to you becau<br>ory problems: | se of | |
| | True | False | | |
| I cannot play sports or do other physical activities | | | | |
| I cannot go out for entertainment or recreation | | H | | |
| cannot go out of the house to do the shopping | | | | |
| I cannot do household chores | | | | |
| cannot move far from my bed or chair | | | | |

Pirfenidone — F. Hoffmann-La Roche Ltd

## St. George's Respiratory Questionnaire

| Here is a list of other activities that your respiratory problems may prevent you fro<br>do not have to check these, they are just to remind you of ways your shortness of<br>affect you): | |
|---|---|
| Going for walks or walking the dog | |
| Doing activities or chores at home or in the garden | |
| Sexual intercourse | |
| Going to a place of worship, or a place of entertainment | |
| Going out in bad weather or into smoky rooms | |
| Visiting family or friends or playing with children | |
| Please write in any other important activities that your respiratory problems may sto | p you from |
| doing: | |
| Now please check the box (one only) that you think best describes how your respira affect you: | atory problems |
| It does not stop me from doing anything I would like to do | |
| It stops me from doing one or two things I would like to do | |
| It stops me from doing most of the things I would like to do | |
| it stops me from doing everything I would like to do | |
| Thank you for completing this questionnaire. Before you finish would you please make a<br>answered all the questions. | ure that you have |

#### STRUCTURE OF SGRQ

The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction.

**Part 1 (Questions 1-8)** addresses the frequency of respiratory symptoms. It is not designed to be a precise epidemiological tool, but to assess the patient's perception of their recent respiratory problems.

Part 2 (Sections 9-16) addresses the patient's current state (i.e. how they are these days).

The Activity score measures disturbances to daily physical activity. The Impacts score covers a range of disturbances of psycho-social function. Validation studies for the original SGRQ showed that this component relates in part to respiratory symptoms, but it also correlates quite

Pirfenidone — F. Hoffmann-La Roche Ltd

strongly with exercise performance (6-minute walk test), breathlessness in daily life (MRC breathlessness score) and disturbances of mood (anxiety and depression). The Impacts score is, therefore, the broadest component of the questionnaires, covering the whole range of disturbances that respiratory patients experience in their lives.

Three component scores are calculated for the SGRQ

**Symptoms** – concerned with the effect of respiratory symptoms their frequency and severity

**Activity** concerned with activities that cause or are limited by breathlessness

**Impacts** covers a range of aspects concerned with social functioning and psychological disturbances resulting from airway disease.

**Total score** summaries the impact of disease on overall health status. Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status.

#### SGRQ SCORES IN HEALTHY SUBJECTS

Means (95% confidence intervals) for SGRQ scores in normal subjects with no history of respiratory disease

| N | Age-years | FEV1 as<br>%<br>predicted | Symptoms score | Activity score | Impacts<br>Score | Total<br>Score |
|---|---|---|---|---|---|---|
| 72 | 46 (17 - 80) | 95 (91-<br>99) | 12 (9-15) | 9 (7-12) | 2 (1-3) | 6 (5-7) |

Pirfenidone — F. Hoffmann-La Roche Ltd

## **Scoring**

Questions 1-7 The eCRF screens should be set up so that where a patient has ticked a box, a value of 1 is entered for the appropriate question. By default, the empty boxes are entered as 0. Where a patient has missed a question the cells on the spreadsheet are left blank. Example: Response = 1c, 'Over the last year I have coughed a few days a month'. A value of 1 is entered for 1c and a value of 0 is entered for 1a, 1b, 1d and 1e. If no tick was present for question 1 then 1a to 1e would be left blank.

Question 8 Where a patient has ticked 'Yes' to having a worse wheeze in the morning, a value of 1 is entered for the appropriate question. All other responses are entered as 0. Example: Do you have a wheeze? = 'Yes' and Worse in the morning = 'Yes'. then response to question 8 = 1. Do you have a wheeze? = 'Yes' and Worse in the morning = 'No'. Or, Do you have a wheeze? = 'No'. then response to question 8=0.

Questions 9, 10 & 17 Where a patient has ticked a box, a value of 1 is entered for the appropriate question. The empty boxes are entered as 0. Where a patient has missed the question the cells on the spreadsheet are left blank. Example: Response = 10a, 'My chest trouble made me stop work'. A value of 1 is entered for 10a and a value of 0 is entered for 10b and 10c. If no tick was present for question 10, then 10a to 10c would be left blank.

Questions 11 – 16 Where a patient has ticked 'True' a value of 1 is entered for the appropriate question and where a patient has ticked 'False' a value of 0 is entered. Where a patient has missed a question the cell on the spreadsheet is left blank.

Example: 15a = 'True' then 15a = 1.

14c = 'False' then <math>14c = 0.

13h = missing then 13h is left blank

In response to question 14, if a patient is not receiving medication, enter the responses as zero, otherwise the calculator will read the values as missing.

Missing Questions

There should not be any missing items in the questionnaire, but the SGRQ can have up to 24% of missing items in the questionnaire. If more than 24% of items are missing the scores will be missing.

Pirfenidone — F. Hoffmann-La Roche Ltd

#### **ITEM WEIGHTS**

Once the questions have been answered the following weights are applied to the individual responses

#### PART 1

Over the past 3 months, I have coughed:

| Most<br>days/week | Several days/<br>week | A few days a month | Only with chest infections | Not at all |
|---|---|---|---|---|
| 80.6 | 63.2 | 29.3 | 28.1 | 0.0 |

Over the past 3 months, I have brought up phlegm (sputum):

| Most<br>days/week | Several days/<br>week | A few days a month | Only with chest infections | Not at all |
|---|---|---|---|---|
| 76.8 | 60.0 | 34.0 | 30.2 | 0.0 |

3) Over the past 3 months, I have had shortness of breath:

| Most<br>days/week | Several days/<br>week | A few days a month | Only with chest infections | Not at all |
|---|---|---|---|---|
| 87.2 | 71.4 | 43.7 | 35.7 | 0.0 |

4) Over the past 3 months, I have had attacks of wheezing:

| Most<br>days/week | Several days/<br>week | A few days a month | Only with chest infections | Not at all |
|---|---|---|---|---|
| 86.2 | 71.40 | 45.6 | 36.4 | 0.0 |

5) During the past 3 months, how many severe or very bad unpleasant attacks of chest trouble have you had?

Pirfenidone — F. Hoffmann-La Roche Ltd

| More than three | 3 attacks | 2 attacks | 1 attack | None |
|-----------------|-----------|-----------|----------|------|
| 86.7 | 73.5 | 60.3 | 44.2 | 0.0 |

## 6) How long did the worst attack of chest trouble last?

| a week or more | 3 or more days | 1 or 2 days | Less than a day | None |
|----------------|----------------|-------------|-----------------|------|
| 89.7 | 73.5 | 58.8 | 41.9 | 0.0 |

Pirfenidone — F. Hoffmann-La Roche Ltd

# 7) Over the past 3 months, in an average week, how many good days (with little chest trouble) have you had?

| No good days | 1 or 2 good<br>days | 3 or 4 good<br>days | Nearly every day | Every day |
|---|---|---|---|---|
| 93.3 | 76.6 | 61.5 | 15.4 | 0.0 |

## 8) If you have a wheeze, is it worse in the morning?

| No | Yes |
|-----|------|
| 0.0 | 62.0 |

#### PART 2

The weights in Part 2 are also applied to the individual responses to each question. The worse the impact the higher the weight. This means that weights are not applied sequentially in the order that the response is given.

## 9) How would you describe your chest condition?

| The most important problem I have | 83 .2 |
|-----------------------------------|-------|
| Causes me quite a lot of problems | 82.5 |
| Causes me a few problems | 34.6 |
| Causes no problem | 0.0 |

#### 10) If you have ever had paid employment?

My chest trouble made me stop work 88.9

Pirfenidone — F. Hoffmann-La Roche Ltd

| My chest trouble interferes with my work or made me change my work | 77.6 |
|-----------------------------------------------------------------------|------|
| My chest trouble does not affect my work | 0.0 |
| 11) Questions about what activities usually make you feel breathless. | |
| Sitting or lying still | 90.6 |
| Getting washed or dressed | 82.8 |
| Walking around the home | 80.2 |
| Walking outside on the level | 81.4 |
| Walking up a flight of stairs | 76.1 |
| Walking up hills | 75.1 |
| Playing sports or games | 72.1 |

| 12) | More o | uestions | about | vour | cough | and | breathles | sness. |
|-----|--------|----------|-------|------|-------|-----|-----------|--------|

| My cough hurts | 81.1 |
|-----------------------------------------------------------------------|------|
| My cough makes me tired | 79.1 |
| I get breathless when I talk | 84.5 |
| I get breathless when I bend over | 76.8 |
| My cough or breathing disturbs my sleep | 87.9 |
| I get exhausted easily | 84.0 |
| 13) Questions about other effects your chest trouble may have on you. | |
| My cough or breathing is embarrassing in public | 74.1 |
| My chest trouble is a nuisance to my family, friends or neighbours | 79.1 |
| I get afraid or panic when I cannot get my breath | 87.7 |
| I feel that I am not in control of my chest problem | 90.1 |
| I do not expect my chest to get any better | 82.3 |
| I have become frail or an invalid because of my chest | 89.9 |
| Exercise is not safe for me | 75.7 |
| Everything seems too much of an effort | 84.5 |
| 14) Questions about your medication. | |
| My medication does not help me very much | 88.2 |
| Pirfenidone — F. Hoffmann-La Roche Ltd | |
| Statistical Analysis Plan MA39189, Version 3.0, 17-July-2020 | |

| | I get embarrassed using my medication in public | 53.9 |
|---|---|---|
| | I have unpleasant side effects from my medication | 81.1 |
| | My medication interferes with my life a lot | 70.3 |
| 15) | Questions about how activities may be affected by your breathing. | |
| | I take a long time to get washed or dressed | 74.2 |
| | I cannot take a bath or shower, or I take a long time | 81.0 |
| | I walk more slowly than other people, or I stop for rests | 71.7 |
| | Jobs such as housework take a long time, or I have to stop for rests | 70.6 |
| | If I walk up one flight of stairs, I have to go slowly or stop | 71.6 |
| | If I hurry or walk fast, I have to stop or slow down | 72.3 |
| | My breathing makes it difficult to do things such as walk up hills, carry things up stairs, light gardening such as weeding, dance, play bowls or play golf | 74.5 |
| | My breathing makes it difficult to do things such as carry heavy loads, dig the garden or shovel snow, jog or walk at 5 miles per hour, play tennis or swim | 71.4 |
| | My breathing makes it difficult to do things such as very heavy manual work, run, cycle, swim fast or play competitive sports | 63.5 |

Pirfenidone — F. Hoffmann-La Roche Ltd

16) We would like to know how your chest trouble usually affects your daily life.

| I cannot play sports or games | 64.8 |
|-------------------------------------------------|------|
| I cannot go out for entertainment or recreation | 79.8 |
| I cannot go out of the house to do the shopping | 81.0 |
| I cannot do housework | 79.1 |
| I cannot move far from my bed or chair | 94.0 |

17) Tick the statement which you think best describes how your chest affects you.

| It does not stop me doing anything I would like to do | 0.0 |
|---------------------------------------------------------|------|
| It stops me doing one or two things I would like to do | 42.0 |
| It stops me doing most of the things I would like to do | 84.2 |
| It stops me doing everything I would like to do | 96.7 |

#### SCORING ALGORITHM

Three component scores are calculated: Symptoms; Activity; Impacts

One **Total** score is also calculated.

#### PRINCIPLE OF CALCULATION

Each questionnaire response has a unique empirically derived 'weight'. The lowest possible weight is zero and the highest is 100.

Pirfenidone — F. Hoffmann-La Roche Ltd

Each component of the questionnaire is scored separately in three steps:

i. The weights for all items with a positive response are summed.

ii The weights for missed items are deducted from the maximum possible weight for each component. The weights for all missed items are deducted from the maximum

possible weight for the Total score.

iii. The score is calculated by dividing the summed weights by the adjusted maximum

possible weight for that component and expressing the result as a percentage :

Score = 100 x Summed weights from positive items in that component

Sum of weights for all items in that component

The Total score is calculated in similar way:

Score =  $100 \times \text{Summed}$  weights from positive items in the questionnaire

Sum of weights for all items in the questionnaire

Sum of maximum possible weights for each component and Total:

Symptoms 662.5

Activity 1209.1

Impacts 2117.8

Total 3989.4

(Note: these are the maximum possible weights that could be obtained for the worst possible state of the patient).

Pirfenidone — F. Hoffmann-La Roche Ltd

It will be noted that the questionnaire requests a single response to questions 1-7, 9-10 and 17. If multiple responses are given to one of these questions then averaging the weights for the positive responses for that question are acceptable

#### SYMPTOMS COMPONENT

This is calculated from the summed weights for the positive responses to questions 1-8.

#### **ACTIVITY COMPONENT**

This is calculated from the summed weights for the positive responses to guestions 11 and 15.

#### **IMPACTS COMPONENT**

This is calculated from the summed weights for the positive responses to questions 9-10, 12-14 and 16-17.

#### **TOTAL SCORE**

The Total score is calculated by summing all positive responses in the questionnaire and expressing the result as a percentage of the total weight for the questionnaire

## **HANDLING MISSED ITEMS**

There should not be any missed items but if there are missing items the scores should be calculated using the following rules:

following should be used: The following method is recommended for missing items:

#### **Symptoms**

Pirfenidone — F. Hoffmann-La Roche Ltd

| The Symptoms component will tolerate a maximum of 2 missed items. The weight for the missed item is subtracted from the total possible weight for the Symptoms component (662.5) and from the Total weight (3989.4). |
|---|
| Pirfenidone — F. Hoffmann-La Roche Ltd |
| Statistical Analysis Plan MA39189, Version 3.0, 17-July-2020 |

## **Activity**

The Activity component will tolerate a maximum of 4 missed items. The weight for the

missed item is subtracted from the total possible weight for the Activity component (1209.1) and from the Total weight (3989.4).

#### **Impacts**

The Impacts component will tolerate a maximum of 6 missed items. The weight for the missed item is subtracted from the total possible weight for the Impacts component (2117.8) and from the Total weight (3989.4).

This visual analogue scale is designed to help us learn about the severity of your cough. This scale is 100mm (10cm) in length.

During the last week, how do you rate the severity of your cough; 0 mm representing no cough and 100 mm representing the worst cough ever? Please indicate the severity of your cough by placing an  $\mathbf{X}$  on the line.

Pirfenidone — F. Hoffmann-La Roche Ltd

## **Cough Visual Analogue Scale (VAS)**

During the last week, how do you rate the severity of your cough; 0 mm representing no cough and 100 mm representing the worst cough ever? Please indicate the severity of your cough by placing an  $\mathbf{X}$  on the line.

## Worst Cough ever (100mm)



Pirfenidone — F. Hoffmann-La Roche Ltd

#### STATISTICAL ANALYSIS PLAN

TITLE: MULTICENTER, INTERNATIONAL, DOUBLE-

BLIND, TWO-ARM, RANDOMIZED, PLACEBO-CONTROLLED PHASE II TRIAL OF PIRFENIDONE

IN PATIENTS WITH UNCLASSIFIABLE

PROGRESSIVE FIBROSING ILD

PROTOCOL NUMBER: MA39189

STUDY DRUG: Pirfenidone (RO0220912)

**VERSION NUMBER:** Version 2.0 Final 29-Oct-2018

IND NUMBER: 67284

**Eudract Number:** 2016-002744-17

SPONSOR: F. Hoffmann-La Roche Ltd

PLAN PREPARED BY:

(F. Hoffmann-La Roche Ltd)

**DATE FINAL:** 29 October 2018

## SIGNATURE PAGE

| Roche Biostatistician | |
|-----------------------|---------------------|
| | 30-0ct 2018 Date |
| Study Biostatistician | |
| | 31-007-2018<br>Date |
| | 30-Oct-2018 |

Pirfenidone — F. Hoffmann-La Roche Ltd

Statistical Analysis Plan MA39189, Version 2.0, 29-Oct-2018

# STATISTICAL ANALYSIS PLAN AMENDMENT RATIONALE

The following changes were made compared to the first version of the SAP:

| Version | Date | Change number | Change description |
|---|---|---|---|
| 2 | 08-Oct-2018 | 1 | Clarification related to the aim and timeline of the primary analysis and final analysis of the study are included under section Outcome Measures. |
| 2 | 08-Oct-2018 | 2 | Week 28 is included in all descriptive efficacy tables. |
| 2 | 08-Oct-2018 | 3 | The safety follow-up period definition is changed as stated in section <u>On-treatment Assessments (12-Month Safety Follow-up Period)</u> . |
| 2 | 08-Oct-2018 | 4 | Disposition is updated in section <u>Patient Disposition</u> . |
| 2 | 08-Oct-2018 | 5 | Details were added in order to analyze valid daily spirometry data in section <a href="Demographic and Baseline Characteristics">Demographic and Baseline Characteristics</a> . |
| 2 | 08-Oct-2018 | 6 | Additional analyses needed in the safety follow-up period based on safety follow-up population are presented under section <u>Safety Follow-up analyses</u> . |
| 2 | 08-Oct-2018 | 7 | Safety follow-up visits were included under section <u>Visit Windows</u> . |
| 2 | 08-Oct-2018 | 8 | Listings of stratification factors, separated types of adverse events and pregnancy data were removed from the corresponding sections. |
| 2 | 29-Oct-2018 | 9 | Post-medications during safety follow-up period are adapted as per new period definition in section <a href="Previous and Concomitant Medication">Previous and Concomitant Medication</a> . |

## **TABLE OF CONTENTS**

| SIC | SNATURE PA | \GE | 2 |
|-----|-------------|---------------------------------------------------|----|
| ST | ATISTICAL A | NALYSIS PLAN AMENDMENT RATIONALE | 3 |
| 1. | BACKGRO | UND | 11 |
| 2. | STUDY DE | SIGN | 11 |
| | 2.1 | Protocol Synopsis | 12 |
| | 2.2 | Outcome Measures | 12 |
| | 2.2.1 | Primary Efficacy Outcome Measures | 13 |
| | 2.2.2 | Secondary Efficacy Outcome Measures | 13 |
| | 2.2.3 | Exploratory Efficacy Outcome Measures | 14 |
| | 2.2.4 | Safety Outcome Measures | 14 |
| | 2.3 | Determination of Sample Size | 14 |
| | 2.4 | Interim Analysis | 15 |
| 3. | STUDY CO | NDUCT | 15 |
| | 3.1 | Randomization, BLINDING AND UNBLINDING PROCEDURES | 15 |
| | 3.2 | Independent Review Facility | 15 |
| | 3.3 | Data Monitoring | |
| 4. | STATISTIC | AL METHODS | 16 |
| | 4.1 | Analysis Populations | 16 |
| | 4.1.1 | Intent-to-treat Population | 16 |
| | 4.1.2 | Per Protocol Population | 16 |
| | 4.1.3 | Safety Population | 16 |
| | 4.1.4 | Safety Follow-up Population | 16 |
| | 4.2 | Trial Periods, Observation and analysis times | 17 |
| | 4.2.1 | Study Days | 17 |
| | 4.2.2 | Baseline and Screening Observations | 17 |

Pirfenidone — F. Hoffmann-La Roche Ltd

| | 4.2.3<br>(Double-bli | On-treatment Assessments for Efficacy Analyses ind Treatment Period) | . 18 |
|---|---|---|---|
| | 4.2.4<br>(Double-bli | On-treatment Assessments for Safety Analyses ind Treatment Period) | . 18 |
| | 4.2.5<br>Follow-up l | On-treatment Assessments (12-Month Safety<br>Period) | . 18 |
| | 4.2.6 | Cut-off points | . 18 |
| | 4.3 | Analysis of Treatment arm Comparability | . 19 |
| | 4.4 | Analysis of Study Conduct | . 19 |
| | 4.4.1 | Patient Disposition | . 19 |
| | 4.4.2 | Major Protocol Deviations | . 21 |
| | 4.4.3 | Demographic and Baseline Characteristics | . 21 |
| | 4.4.4 | Previous and Concomitant Medication | . 24 |
| | 4.4.5 | Compliance | . 25 |
| | 4.5 | Efficacy Analysis | . 25 |
| | 4.5.1 | Primary Efficacy Endpoints | . 26 |
| | 4.5.2 | Secondary Efficacy Endpoints | . 27 |
| | 4.5.3 | Exploratory Efficacy Endpoints | . 29 |
| | 4.5.4 | Analyses of Patient-Reported Outcomes | . 30 |
| | 4.5.5 | Sensitivity Analyses | . 32 |
| | 4.5.6 | Subgroup Analyses | . 32 |
| | 4.6 | Pharmacokinetic and Pharmacodynamic Analyses | . 33 |
| | 4.7 | Safety Analyses | . 33 |
| | 4.7.1 | Exposure of Study Medication | . 34 |
| | 4.7.1.1 | Treatment duration | . 34 |
| | 4.7.1.2 | Doses and Dose modifications or interruptions | . 34 |
| | 4.7.2 | Adverse Events | . 35 |
| | 4.7.3 | Deaths | . 38 |
| | 4.7.4 | Laboratory Data | . 38 |
| | 4.7.5 | Vital Signs | . 39 |
| ·fο | nidone — F Ho | offmann-La Rocha Ltd | |

| | 4.7.6 | ECG | . 39 |
|----|----------|---------------------------|------|
| | 4.8 | Safety Follow-up analyses | |
| | 4.9 | Missing Data | |
| | 4.10 | Visit Windows | |
| | 4.11 | Interim Analyses | . 43 |
| | 4.12 | Biomarker Analyses | . 43 |
| RF | FERENCES | | 15 |

Pirfenidone — F. Hoffmann-La Roche Ltd

## LIST OF TABLES

| Table 1 | Definition of Baseline and Screening Observations | 17 |
|------------|---------------------------------------------------|----|
| Table 2 | Visit Windows | 42 |
| | LIST OF APPENDICES | |
| APPENDIX 1 | PROTOCOL SYNOPSIS | 46 |
| APPENDIX 2 | SCHEDULE OF ASSESSMENTS | 54 |
| | PATIENT REPORTED OUTCOME<br>ONNAIRE | 62 |

Pirfenidone — F. Hoffmann-La Roche Ltd

## **LIST OF ABBREVIATIONS**

| Abbreviation | Definition |
|--------------|----------------------------------------------------------|
| 6MWD | 6-minute walk distance |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| AST | aspartate aminotransferase |
| BID | two times daily |
| BTPS | body temperature and pressure saturated with water vapor |
| BP | blood pressure |
| BUN | blood urea nitrogen |
| CAPACITY | Clinical Studies Assessing Pirfenidone in idiopathic |
| | pulmonary fibrosis: Research of Efficacy and Safety |
| | Outcomes |
| cHP | chronic hypersensitivity pneumonitis |
| CI | confidence interval |
| CRO | contract research organization |
| CSP | clinical study protocol |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTD | connective tissue disease |
| CYP | cytochrome P450 |
| DLco | diffusing capacity of the lung for carbon monoxide |
| DNA | deoxyribonucleic acid |
| DSMB | Data and Safety Monitoring Board |
| EC | Ethics Committee |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| EEA | European Economic Area |
| ERA | endothelin receptor antagonist |
| FDA | Food and Drug Administration |
| FEV1 | forced expiratory volume in 1 second |
| FVC | forced vital capacity |
| GCP | Good Clinical Practice |
| GERD | gastroesophageal reflux disease |
| HIPAA | Health Insurance Portability and Accountability Act |
| HRCT | high-resolution computed tomography |
| ICH | International Conference on Harmonisation |
| iDMC | independent Data Monitoring Committee |

Pirfenidone — F. Hoffmann-La Roche Ltd

| T | |
|--------|---------------------------------------------------------------|
| IL | interleukin |
| ILD | interstitial lung disease |
| IMP | investigational medicinal product |
| IND | investigational New Drug |
| IPAF | interstitial pneumonia with autoimmune features |
| IPF | idiopathic pulmonary fibrosis |
| IRB | Institutional Review Board |
| ITT | intent-to-treat |
| IxRS | interactive voice or web-based response system |
| LDH | lactate dehydrogenase |
| LFT | liver function test |
| LOTUSS | An open-Label, randOmized, Phase 2 sTUdy of the safety |
| | and tolerability of pirfenidone when administered to patients |
| | with Systemic Sclerosis-related interstitial lung disease |
| LPLV | last patient, last visit |
| MDT | multidisciplinary team |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMF | mycophenolate mofetil/sodium or mycophenolate acid |
| NAC | N-acetyl-cysteine |
| NCI | National Cancer Institute |
| NGS | next-generation sequencing |
| NSIP | nonspecific interstitial pneumonia |
| PDGF | platelet-derived growth factor |
| PDMS | protocol deviation management system |
| PFS | progression-free survival |
| PFTs | pulmonary function tests |
| PRO | patient-reported outcome |
| QTcF | QT interval corrected using Fridericia's formula |
| RBC | red blood cells |
| RBR | Research Biosample Repository |
| RNA | ribonucleic acid |
| RoW | Rest of the World |
| SAP | Statistical Analysis Plan |
| SBP | systolic blood pressure |
| SGRQ | St. George's Respiratory Questionnaire |
| SOBQ | Shortness of Breath Questionnaire |
| SOC | System Organ Class |
| SOP | standard operating procedure |
| SpO2 | oxyhemoglobin saturation at rest |

## Pirfenidone — F. Hoffmann-La Roche Ltd

| SSc | systemic sclerosis |
|------|-------------------------------------|
| TGF | transforming growth factor |
| TID | three times daily |
| UCSD | University of California, San Diego |
| UIP | usual interstitial pneumonia |
| ULN | upper limit of normal |
| US | United States |
| VAS | Visual Analogue Scale |
| VC | vital capacity |
| WBC | white blood cells |
| WGS | whole genome sequencing |

Pirfenidone — F. Hoffmann-La Roche Ltd

#### 1. BACKGROUND

As described in the Clinical Study Protocol (CSP) Section 1.3, no approved treatments are available for the 15% of patients with interstitial lung disease (ILD) who have unclassifiable disease. Therapeutic management is based on the most probable diagnosis after multidisciplinary discussions and consideration of the expected disease behavior (Antoniou et al. 2014). The data for pirfenidone in idiopathic pulmonary fibrosis (IPF) are sufficiently encouraging to hypothesize that a beneficial clinical effect would also be observed with this agent in patients with unclassifiable fibrosing ILD.

There are several key areas for uncertainty in the assessment of the benefit-risk profile for pirfenidone (Esbriet®) in the unclassifiable ILD patient population. Fibrosing ILD might have a different natural history compared with IPF and the efficacy of pirfenidone treatment may be different in patients with unclassifiable ILD compared with patients with IPF.

Mycophenolate mofetil/sodium or mycophenolic acid (MMF) may have an effect on the disease course of patients with unclassifiable ILD, in particular patients with interstitial pneumonia with autoimmune features (IPAF). Patients may be receiving treatment with MMF as a concomitant therapy at the start of the trial and therefore the patient population in this trial will be stratified according to use of MMF. Patients receiving MMF concomitant therapy at the start of the trial are allowed to continue with this treatment throughout the study including the 24-week double-blind and 12-month safety follow-up periods. A similar approach had been used previously in a study of the safety and tolerability of pirfenidone in patients with systemic sclerosis-related ILD (SSc-ILD; an open-Label, randOmized. Phase 2 sTUdy of the safety and tolerability of pirfenidone when administered to patients with Systemic Sclerosis-related interstitial lung disease [LOTUSS]) (Khanna et al. 2016). The results of this trial also include data concerning the use of MMF as concomitant treatment with pirfenidone. The conclusion from this trial was that MMF, which was taken concomitantly with pirfenidone by 63.5% of patients, did not appear to affect the tolerability of pirfenidone and no particular safety concerns were noted following the combined use of MMF and pirfenidone.

## 2. STUDY DESIGN

This is a multicenter, international, double-blind, two-arm, randomized, placebo-controlled Phase II trial in patients with fibrosing ILD who cannot be classified with moderate or high confidence into any other category of fibrosing ILD by multidisciplinary team (MDT) review ("unclassifiable ILD"). Patients will be randomized in a 1:1 ratio, on a double-blind basis using a stratified algorithm, to receive either pirfenidone (801 mg TID) or placebo. The randomized patients will be stratified by concomitant MMF treatment (yes/no), the presence/absence of IPAF as defined by the MDT.

In total, approximately 90 clinical centers (sites) in Australia, Europe, the Middle East, and North America are expected to enroll approximately 250 patients. Patients who are withdrawn from the trial will not be replaced.

Pirfenidone — F. Hoffmann-La Roche Ltd

After discussing the risks and benefits of the trial with the investigator and providing informed consent, patients will be required to taper and/or discontinue all prohibited medications (Section 4.4.2 in the CSP) in the 28 days prior to the start of screening during the washout period. If a prohibited medication must be tapered, the process must start early enough so that the patient discontinues the medication in the 28 days prior to the start of screening. After completing the washout patients will enter screening, which lasts up to 21 days. During screening, patients will be evaluated for eligibility based on the inclusion and exclusion criteria. Patients not taking a prohibited medication will forgo the washout period and directly enter screening.

At the end of screening, patients will be randomized (Day 1) to receive either pirfenidone or placebo (1:1 ratio).

Following treatment initiation, the daily dosage will be titrated to the full dosage of nine capsules per day over a 14-day period. After the titration period, trial treatment will continue through Week 24 and monitoring will be conducted by site visits. Patients should remain on a stable maintenance dose for the duration of the treatment period unless the dose is reduced or dosing is interrupted to manage an adverse event (see CSP Section 5.1.1). Any patient with an actual or anticipated interruption of trial treatment for a period of ≥28 consecutive days will be reported by telephone to Roche's medical monitor or designee to discuss the circumstances of the case. A Follow-up Visit will occur 28 days after the end of the 24-week double-blind treatment period.

After completion of the double-blind treatment period and the Follow-up visit at Week 28, patients will be given the opportunity to receive open-label pirfenidone within a safety follow-up period of up to 12 months of the trial protocol. A final Follow-up visit will be performed at the end of the safety period, 28 days after the last open-label dose. During the safety follow-up period, the patients should be evaluated by the investigator initially at monthly visits during the first 6 months and subsequently at each visit occurring approximately every 3 months thereafter.

### 2.1 PROTOCOL SYNOPSIS

The Protocol Synopsis is in <u>Appendix 1</u> and the Schedule of Assessments in <u>Appendix 2</u> For additional details, please see the CSP Version 3, 28 June 2018 (and its Appendices).

#### 2.2 OUTCOME MEASURES

This trial will evaluate the efficacy and safety of pirfenidone in patients with fibrosing interstitial lung disease (ILD) who cannot be classified with moderate or high confidence into any other category of fibrosing ILD by multidisciplinary team (MDT) review ("unclassifiable" ILD).

The primary analysis of the primary and secondary efficacy outcome measures of this study is planned to be performed when the last patient reached the date of the last follow-up visit after end of the double-blind treatment period.

Pirfenidone — F. Hoffmann-La Roche Ltd

## 2.2.1 Primary Efficacy Outcome Measures

The primary efficacy objective for this trial is to evaluate the effect of pirfenidone vs. placebo on lung function parameters on the basis of Forced Vital Capacity (FVC) measurements. FVC will be measured daily by the patients by use of a handheld spirometer.

The primary efficacy endpoint is defined as:

 rate of decline in FVC in mL measured by daily handheld spirometry over the 24week double-blind treatment period.

## 2.2.2 <u>Secondary Efficacy Outcome Measures</u>

The secondary efficacy objective for this trial is to evaluate the efficacy of pirfenidone compared with placebo from baseline until Week 24 on other functional parameters, outcomes, and patient reported outcomes (PROs).

The following endpoints will be analyzed:

- Change in percent predicted FVC and in mL measured by spirometry during clinic visits
- Categorical change in FVC of >5% (absolute change in percent predicted and relative change in mL), measured both by daily spirometry as well as by spirometry during clinic visits
- Categorical change in FVC of >10% (absolute change in percent predicted and relative change in mL), measured both by daily spirometry as well as by spirometry during clinic visits
- Change in percent predicted diffusing capacity of the lung for carbon monoxide (DLco)
- Change in (6-minute walk distance) 6MWD in meters
- Change in University of California, San Diego Shortness of Breath Questionnaire (UCSD-SOBQ) score
- Change in score in Leicester Cough Questionnaire
- Change in cough visual analog scale
- Change in total and sub-scores of the St. George's Respiratory Questionnaire (SGRQ)
- Non-elective hospitalization, both respiratory and all cause
- Incidence of, and time to first, investigator-reported acute exacerbations
- Progression free survival (PFS), defined as the time to the first occurrence of a >10% absolute decline in percent predicted FVC (measured during a clinic visit), a >50 m decline of 6MWD, or death
- PFS, alternatively defined as the time to the first occurrence of a >10% relative decline in FVC (measured during a clinic visit), non-elective respiratory hospitalization, or death

Pirfenidone — F. Hoffmann-La Roche Ltd

- Time to death from any cause
- Time to death from respiratory diseases

## 2.2.3 Exploratory Efficacy Outcome Measures

One exploratory objective for this trial is to evaluate the role of mycophenolate mofetil/sodium or mycophenolic acid (MMF) treatment in ILD and to evaluate potential biomarkers associated with fibrosis and ILD.

The exploratory endpoints associated are:

- Efficacy and safety data from subgroups of patients who did or did not receive MMF treatment
- Biomarker data from plasma, serum, and whole blood ribonucleic acid (RNA) and deoxyribonucleic acid (DNA) samples

#### 2.2.4 <u>Safety Outcome Measures</u>

The safety objective for this trial is to evaluate the safety of pirfenidone vs. placebo by investigating the following endpoints:

- Nature, frequency, severity, and timing of treatment-emergent adverse events
- Dose reductions and treatment interruptions
- Clinical laboratory test results
- 12-lead ECGs
- Withdrawals from trial treatment or trial discontinuations

All analyses with regard to the safety outcome measures will be performed from the date of first randomized treatment intake until 28 days after the last positive dose during the double-blind randomized treatment period.

#### 2.3 DETERMINATION OF SAMPLE SIZE

The purpose of this trial is hypothesis generation regarding the efficacy of pirfenidone vs. placebo on lung function parameters on the basis of rate of decline in FVC, as measured by daily handheld spirometry.

A total sample size of approximately 250 patients is planned, and patients will be randomized in a 1:1 ratio. The randomization will be stratified by concomitant MMF treatment (yes/no), the presence/absence of IPAF as defined by the MDT.

The planned sample size is based on the statistical hypothesis of the primary endpoint and assumes 80% power and a two-sided significance level of 5% using a student's ttest. It is assumed, after inspection of historical data, that FVC decline in the placebo arm is 85 mL with a common standard deviation of 70 mL, which can be reduced to 60 mL with a common standard deviation of 70 mL in the pirfenidone arm. In this

Pirfenidone — F. Hoffmann-La Roche Ltd
scenario, 125 patients per treatment arm are needed to detect this treatment effect with 80% power.

These assumptions are based upon the following considerations: in IPF, the annual rate of decline of FVC is approximately 200 mL. Owing to the fact that patients with unclassifiable ILD have rates of disease progression in the range of patients with IPF, albeit with a lower mortality rate (Ryerson et al. 2013), a similar decline rate of 200 mL/year, equivalent to a 100 mL decline over a treatment period of 24 weeks, can be expected. However, a yet unknown proportion of patients in this trial will be treated concomitantly with MMF. In a previous study of CTD-ILD (Fischer et al. 2013), MMF was found to have beneficial effects on lung functions in these patients. While CTD-ILD is a distinct entity from the current trial population, both conditions may share some autoimmune features. Therefore assuming a smaller FVC decline of 85 mL in the placebo arm compared with 60 mL in the pirfenidone arm over the 24-week double-blind treatment period appears justified. In addition, the potential confounding effect of concomitant MMF therapy in these patients justifies stratification to ensure equal distribution of patients who receive and do not receive treatment with MMF.

#### 2.4 INTERIM ANALYSIS

There are no planned interim efficacy analyses for this trial.

#### 3. <u>STUDY CONDUCT</u>

The study conduct is described in <u>Section 2</u>.

#### 3.1 RANDOMIZATION, BLINDING AND UNBLINDING PROCEDURES

Patients will be randomized 1:1 to receive either pirfenidone or placebo. The randomization process will be conducted using a validated interactive voice or webbased response system (IxRS). To guard against systematic selection bias and ensure comparability of treatment arm, the randomization will be stratified by concomitant MMF treatment (yes/no), the presence/absence of IPAF as defined by the MDT.

To maintain the double-blind nature of the trial, the pirfenidone and placebo treatments will be identical in appearance (see CSP Section 4.3.1.1).

The investigational site personnel and the patients will be blinded to treatment assignment following randomization. The iDMC and any personnel performing any interim analysis (as applicable) will be unblinded to the treatment throughout the trial.

#### 3.2 INDEPENDENT REVIEW FACILITY

Not applicable.

#### 3.3 DATA MONITORING

An independent Data Monitoring Committee (iDMC) will review safety data and advice on study conduct at least three times during the study. Efficacy data will only be provided if requested by the iDMC. A first meeting is planned 6 months after start of recruitment,

Pirfenidone — F. Hoffmann-La Roche Ltd

and subsequently at 12 and 18 months. Details on procedures and safety review by the iDMC are described within an iDMC charter.

#### 4. STATISTICAL METHODS

Categorical data will be summarized using frequencies and percentages (including a category for missing, if appropriate). Percentages will be based on the number of patients in each treatment arm for the analysis population, if not otherwise specified.

Continuous endpoints will be summarized using descriptive statistics (mean, standard deviation, minimum, 25th and 75th quartiles, median, and maximum).

Where data will be summarized over time, the following timepoints will be presented as applicable: Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28 (if applicable) and early discontinuation visit.

Data analysis of data collected during the 12-month safety follow-up period will be described in section 4.8.

Where applicable other analysis methods will be specified below.

#### 4.1 ANALYSIS POPULATIONS

#### 4.1.1 Intent-to-treat Population

The intent-to-treat (ITT) population is defined as all randomized patients. Patients in the ITT population will be assigned to treatment arm as randomized (planned treatment). The ITT population is the primary analysis population for all efficacy analyses. The time period for all efficacy analyses is defined from date of randomization until the treatment completion date of the double-blind treatment period or the date of early discontinuation collected on the early treatment discontinuation eCRF page in case a patient does not complete the planned 24 weeks of double-blind treatment.

#### 4.1.2 Per Protocol Population

Not applicable.

### 4.1.3 <u>Safety Population</u>

The safety population is defined as all patients with at least one intake of pirfenidone or placebo, i.e. at least one record in the drug-log of the double-blind period with a non-zero dose. Patients in the safety population will be assigned to treatment arm according to the actual treatment they received.

## 4.1.4 <u>Safety Follow-up Population</u>

For the 12-month safety follow-up period, the safety follow-up population will be defined as all patients who have received at least one dose of pirfenidone after the randomized treatment end plus 28 days.

Pirfenidone — F. Hoffmann-La Roche Ltd

Safety analyses for the 12-month follow-up period will be performed from the date of the first pirfenidone drug intake during safety follow-up period up to the study completion/discontinuation visit.

## 4.2 TRIAL PERIODS, OBSERVATION AND ANALYSIS TIMES

Where durations are to be calculated (e.g. treatment duration), these will be derived based on the interval in days (end date – start date + 1) and converted to months and years if needed, using 30.4375 and 365.25, respectively, as denominator if not otherwise specified.

For the investigational medicinal product (IMP) exposure, treatments administered from the date of first randomized pirfenidone/placebo treatment up to the date of completion of double-blind treatment or date of early treatment discontinuation, will be regarded.

For drug safety, analyses will be restricted to AEs or assessments that occurred from the first day of randomized treatment until the date of last positive dose of randomized treatment plus 28 days.

Safety analyses for the 12-month follow-up period will be performed using the time window from the safety follow-up period start up to the study completion/discontinuation visit.

#### 4.2.1 Study Days

Study days will be defined as the number of days since randomization, and is calculated as:

- Study day = Assessment date randomization date + 1, for assessments on or after the randomization date.
- Study day = Assessment date randomization date, for assessments before the randomization date.

The day of randomization will be study day 1.

# 4.2.2 <u>Baseline and Screening Observations</u>

## Table 1 Definition of Baseline and Screening Observations

| | Definition |
|---|---|
| Baseline data | Baseline is defined as the last valid assessment prior to first intake of randomized study drug (pirfenidone/placebo). |
| | This may not be the same as the Day 1 (Week 1) visit as per eCRF. In case that Day 1 (Week 1) visit data is missing and the randomized |

Pirfenidone — F. Hoffmann-La Roche Ltd

| | treatment is given, data from the screening period will be used as baseline. In addition, if randomized treatment is not given then baseline will be defined as the last valid assessment collected either screening or day 1. |
|---|---|
| | Generally, it is assumed that measurements referring to the Day 1 (Week 1) visit have been performed before randomized study drug (pirfenidone/placebo) was given. |
| | Adverse events occurring on the date of first randomized pirfenidone/placebo treatment will not be considered baseline, but treatment-emergent. |
| Screening data | Screening measurements are all the measurements performed before the randomization date. |

# 4.2.3 <u>On-treatment Assessments for Efficacy Analyses (Double-blind Treatment Period)</u>

For efficacy analyses, on-treatment assessments will be the assessments performed on or after the randomization date until the double-blind treatment completion or discontinuation date.

# 4.2.4 <u>On-treatment Assessments for Safety Analyses (Double-blind Treatment Period)</u>

For safety analyses, on-treatment assessments will be the assessments performed on or after the first dose of randomized pirfenidone/placebo date until the last positive dose of randomized treatment plus 28 days.

#### 4.2.5 On-treatment Assessments (12-Month Safety Follow-up Period)

Details of all data recorded during the 12-month safety follow-up period will be presented. This period starts on the day of the first positive dose of pirfenidone on or after the 28 days follow-up visit for patients who completed the double-blind treatment period without being discontinued the study. The safety follow-up period ends with the study completion/discontinuation visit, with a maximum duration of 12 months plus 28 days. Safety follow-up analyses will be presented separately from double-blind treatment phase ones.

#### 4.2.6 Cut-off points

The clinical cut-off for the primary analysis will occur when the last patient has completed the final safety Follow-up Visit, 28 days after the double-blind treatment period.

There will be a second cut-off for the final analysis when all patients have completed the 12-month safety follow-up period.

Pirfenidone — F. Hoffmann-La Roche Ltd

For each patient the total length of the trial is expected to be up to a maximum of 91 weeks. The trial duration includes the washout period of up to 4 weeks, the screening period of up to 3 weeks, the double-blind treatment period of 24 weeks, the follow-up period of 4 weeks, the open-label safety follow-up period up to 12 months (52 weeks) plus 28 days and a final safety Follow-up Visit 4 weeks after the last dose.

### 4.3 ANALYSIS OF TREATMENT ARM COMPARABILITY

To ensure the comparability of the treatment arm, the randomization will be stratified by the availability of a previous MMF treatment (yes/no) and the presence/absence of IPAF as defined by MDT to ensure an equal distribution of patients.

These stratification factors will be included in the analysis of the primary endpoint as a sensitivity analysis. Please refer to the corresponding section <u>4.4.5</u> for further details.

Outputs for concordance between the stratification factors by eCRF and by IxRS will also be presented.

## 4.4 ANALYSIS OF STUDY CONDUCT

Unless otherwise specified, all analyses described in this section will be performed on the ITT population, presenting data by treatment arm.

#### 4.4.1 Patient Disposition

An overview on patient disposition, showing number and percentages of patients enrolled, screened, failed screening, randomized, treated, completed or early discontinued the double-blind treatment period, patients entering the 12-month safety follow-up period and their current status (ongoing, completion, discontinued) in that period will be provided. For patients who have early discontinued the double-blind treatment period or the study, frequencies of reasons for early discontinuation will be provided. A listing with all the patient disposition data will be also presented.

The following definitions will be used:

- Patients randomized: All patients who have been randomized to receive either pirfenidone or placebo, i.e. have a randomization date.
- Patients randomized and not treated: all randomized patients who have not received at least one dose of the randomized treatment.
- Patients randomized and treated: all randomized patients who have received at least one dose of the randomized treatment.
- Patients randomized and treated with sufficient post-baseline efficacy data: all randomized patients who have received at least one dose of the randomized treatment and have at least one post-baseline assessment of FVC (mL).

Pirfenidone — F. Hoffmann-La Roche Ltd

- Completion of double-blind treatment period: eCRF question "Did the patient complete course of double-blind treatment?" is ticked "Yes" (eCRF form "Double-blind treatment Completion/Early Discontinuation").
- Early discontinuation (non-completion) of double-blind treatment period: eCRF question "Did the patient complete course of double-blind treatment?" is ticked "No" (eCRF form "Double-blind treatment Completion/Early Discontinuation").
- Early discontinuation (non-completion) of study: eCRF question "Did the subject early discountinue from the study?" is ticked "Yes" (eCRF form "Study Completion/Early Discontinuation") for patients who discontinued double-blind treatment period.
- Early discontinuation (non-completion) of study: eCRF question "Did the subject early discountinue from the study?" is ticked "Yes" (eCRF form "Study Completion/Early Discontinuation") for patients who completed double-blind treatment period and did not enter 12-month safety follow-up period.
- Status during the 12-month safety follow-up (entered, ongoing, completed).
   Completers are defined as those patients that have filled the study completion/discontinuation form. Otherwise, the patient is considered ongoing in the safety follow-up phase.
- Completion of study: eCRF question "Did the subject complete the study?" is ticked "Yes" (eCRF form "Study Completion/Early Discontinuation")
- Early discontinuation (non-completion) of study: eCRF question "Did the subject early discountinue from the study?" is ticked "Yes" (eCRF form "Study Completion/Early Discontinuation")

An overview on patients' enrolment will be provided based on the randomized subjects by country and center separately for the pirfenidone and placebo arm.

Kaplan-Meier (KM) plots for time to treatment discontinuation will be provided for all randomized patients and by randomized arm, based on the date subject completed or early discontinued from double-blind treatment period, as per eCRF. If the patient completed the treatment without treatment discontinuation, then it will be censored to the date of treatment completion.

In addition, KM plots for time to study discontinuation will be presented for all randomized patients by arm, based on the study discontinuation date. If the patient completed the study as planned per protocol, then the patient will be censored to the study completion date.

In addition, a consort diagram with some of the categories above will be presented.

Pirfenidone — F. Hoffmann-La Roche Ltd

## 4.4.2 Major Protocol Deviations

Major protocol deviations and eligibility violations will be summarized by frequency tables and all patients with protocol deviations will be listed. Protocol deviations will be collected in the protocol deviation management system (PDMS), reviewed by the medical monitors, and will be provided in a SAS dataset via the Biometrics Computing Environment (BCE). All deviations provided in that dataset will be considered as major protocol deviations.

### 4.4.3 Demographic and Baseline Characteristics

Baseline and disease characteristics such as demographics, medical history and tobacco use history will be summarized by descriptive statistics or frequency tables for each treatment arm.

# **Demographics**

The following demographic characteristics will be summarized by treatment arm:

- Age (years): as entered in the eCRF at the screening visit.
- Age categories: <65, and ≥ 65.</li>
- Age categories: <45, ≥45 to <65 years, ≥65 to <85 years, and ≥ 85 years.
- Gender: Male/Female.
- Race: White, American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, Unknown. In case that more than one race will be ticked, a concatenated variable, containing all races will be presented (e.g. Asian/White).
- Ethnicity: Hispanic or Latino, Not Hispanic or Latino, Not reported, Unknown.
- · Weight (kg) at baseline
- Height (cm) at baseline
- BMI (kg/m2) at baseline. BMI will be calculated as: weight(kg) / (height(m))2
- Female reproductive status: childbearing potential without contraceptive protection, Childbearing potential with contraceptive protection, surgically sterilized, Postmenopausal, Pre-menarchal, Non childbearing potential.

Data on female reproductive status will be presented descriptively.

Demographic data will be also listed.

#### **Medical History**

Pirfenidone — F. Hoffmann-La Roche Ltd

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), version 20.1 or higher and will be summarized presenting numbers and frequencies by primary System Organ Class (SOC) and Preferred Term (PT) by treatment arm. If patients have more than one disease within a SOC or PT they will be counted only once for the respective SOC or PT.

A listing with past and ongoing medical history data from the washout period will be presented.

## Tobacco use history

The history of tobacco use will be summarized by treatment arm with the following characteristics:

- Tobacco use history (never, current, previous)
- Nicotine exposure (pack-years), smokers only

Numbers and percentages of patients will be provided for tobacco use history. Nicotine exposure will be summarized descriptively.

## Diagnosis and time from uILD Diagnosis

Frequencies and percentages will be presented for the uILD category collected into the eCRF page MDT/Diagnosis (Eligibility).

The time in months since the original uILD diagnosis will be calculated as

Date of randomization – Date of ILD diagnosis and will be summarized descriptively by randomized treatment arm. The number and percentage of patients with a historical high-resolution computed tomography and with a historical surgical lung biopsy will also be presented.

Descriptive statistics of the time from most recent historical high-resolution computed tomography (months) and historical surgical lung biopsy will be presented. As above, the date of randomization will be used as reference date for calculation of duration.

#### Stratification Factors

The number and percentage of patients that fall into each of the four groups based on the two stratification factors: Concomitant MMF treatment (yes/no), and the presence/absence of IPAF as defined by the MDT will be presented by treatment arm.

#### **Baseline Spirometry Test**

The values recorded for the baseline assessments of the spirometry tests were the following:

Pirfenidone — F. Hoffmann-La Roche Ltd

- Forced vital capacity (FVC) (L and % predicted)
- Forced expiratory volume in 1 second (FEV1) (L and % predicted)
- FEV1 (L) / FVC (L) ratio (1)
- Carbon monoxide diffusing capacity (DLco) (% predicted)

Descriptive statistics will be provided for these parameters separately for treatment arm.

## **Historical Spirometry Test**

The number and percentage of patients who performed spirometry test (FVC, DLco, FEV1, and FEV1/FVC ratio) in the past will be provided. The most recent assessment before the Screening visit will be collected:

- Hemoglobin corrected DLco (mmol/min/kPa and %)
- DLco/Va (KCO) (mL/min/mmHg/L and % predicted)
- FVC (L and % predicted)
- FEV1 (L and % predicted)
- FEV1(L)/FVC(L) ratio (1)

These historical spirometry test parameters will be summarized using descriptive statistics by treatment arm. Both, absolute and percent predicted values will be presented. Frequencies and percentages will be presented for the high-resolution computed tomography and the surgical lung biopsy.

#### Baseline Daily Spirometry (Handheld Device) and Site Spirometry

A handheld spirometry device will be used by the patient to measure daily FVC at home. Confirmatory site (trial center) based FVC measurements will be conducted every 4 weeks. The following blow categories will be collected:

| Not acceptable maneuvers | Acceptable maneuvers |
|--------------------------|----------------------|
| Rejected | Accepted |
| Borderline Accepted | |

Only acceptable maneuvers will be considered for the analysis. If one patient has more than one accepted measurement per day, all of them will be used for the analysis.

Pirfenidone — F. Hoffmann-La Roche Ltd

FVC (mL) will be measured daily with a handheld device.

Descriptive statistics of the baseline site measurements will be provided for these parameters separately by treatment arm together with the efficacy results.

#### **Baseline 6-minute walk distance (6MWD)**

The 6MWD is used to evaluate the functional capacity of patients with lung disease. The 6MWD measures the distance a patient is able to walk quickly on a flat, hard surface in a period of 6 minutes.

The number and percentage of patients that

- Performed the 6-minute walking test (yes/no),
- Rested for at least 10 minutes (yes/no),
- Stopped the test before 6 minutes (yes/no),
- Required O2 (yes/no)

at the baseline visit will be summarized by randomized treatment group.

The values of the parameters recorded for the 6MWD test are:

- Vital signs (Heart rate (beats/min), systolic blood pressure (mmHg), diastolic pressure (mmHg)) (before the test, at the end of the test)
- Distance walked (m),
- Oxyhemoglobin saturation (SPO2) (before the test (at rest), at the end of the test),
- Oxygen (O2) requirements (L) (at the end of the test)

will be summarized descriptively by treatment arm.

#### 4.4.4 Previous and Concomitant Medication

Previous and concomitant medications will be presented based on the safety population. Post medications administrated during the safety follow-up period will be presented based on the safety follow-up population.

Previous and concomitant medications are non-study medications. Concomitant therapy includes any medication used by a patient from the washout period until 28 days after the last dose of trial treatment. The previous and concomitant medication will be coded using the Genentech (GNE) drug dictionary. This is a proprietary Roche Dictionary which is used to code concomitant medications in the Trial Management System (TMS) coding tool. The Standardized Medication Name (CMDECOD), which is the medication generic

Pirfenidone — F. Hoffmann-La Roche Ltd

or combination generic as defined by the Drug Thesaurus (proprietary Genentech/Roche dictionary), and the Medication Class (CMCLAS), which is the primary medication class as defined by the Drug Thersaurus, will be used for the analyses.

Therapies will be classified as previous or concomitant as follows:

Previous: If the medication start date is prior to start of double-blind treatment,

Concomitant: If medication is taken at anytime between the start of double-blind treatment and 28 days after last positive dose of randomized treatment.

Post (safety follow-up): if the medication is taken during the safety follow-up period, i.e., on or after the first dose of open-label pirfenidone.

The number and frequency of previous and concomitant medications taken by patients in the two treatment arms will be presented by Medication Class and Standardized Medication Name. If patients receive more than one drug within a Medication Class or Standardized Medication Name they will be counted only once for the respective Medication Class or Standardized Medication Name.

A separated table will be presented for post medications during the safety follow-up period.

All medications will be listed identifying the previous/concomitant and post medications.

The missing imputation rules for the medication dates are described under section 4.8.

#### 4.4.5 Compliance

With respect to the home-based daily measurements compliance of patients will be investigated. It will be analyzed if gaps of measurements occur over time. A gap is thereby defined as 7 or more than 7 consecutive days of missing measurements or non-accepted (borderline accepted or rejected) quality blows. A summary table displaying number of patients with gaps in daily measurements, number of gaps and duration of gaps will be provided by treatment arm for data from handheld spirometer.

#### 4.5 EFFICACY ANALYSIS

The primary and secondary efficacy analyses will include all patients in ITT population, with patients grouped according to their assigned treatment.

The primary analysis of the primary efficacy endpoint of this study is planned to be performed when the last patient reached the date of the last follow-up visit after end of the double-blind treatment period (clinical cut-off date).

Pirfenidone — F. Hoffmann-La Roche Ltd

## 4.5.1 **Primary Efficacy Endpoints**

The primary efficacy objective for this trial is to evaluate the efficacy of pirfenidone vs. placebo on lung function parameters on the basis of rate of decline in FVC in mL measured by handheld spirometer over the 24-week double-blind treatment period.

The primary null hypothesis (H0) is that the mean FVC decline for both treatments is equal:

$$H0: \mu 1 = \mu 2$$

where  $\mu 1$  denotes the mean FVC decline for patients receiving Pirfenidone, and  $\mu 2$  denotes the mean FVC decline for patients receiving Placebo.

The primary alternative hypothesis (H1) is that the mean FVC decline for both treatments is not equal:

$$H1: \mu1 \neq \mu2$$

The primary analysis will be based on the ITT population. Patients who discontinue treatment prematurely will be analyzed based on the available data. No imputation method will be applied for the primary endpoint.

The primary analysis of the primary endpoint will compare the mean FVC decline in each treatment arm using a student's t-test with a two-sided significance level  $\alpha$ =0.05.

The mean FVC decline for each treatment arm will be calculated using the estimated FVC decline for each individual patient. The estimated FVC decline for individual patients will be obtained by applying a linear regression model to all data points collected during the 24-week double-blind treatment period:

$$X_{iz} = \alpha_i + \beta_i D_{iz} + u_{iz}$$

where

 $X_{it}$  = the FVC measurements (mL) of patient i on day t, with i=1,...,N and t=1,...,T, being N the total number of patients randomized and T the total number of days with assessment.

 $D_{it}$  = study day t of patient i

 $\alpha_i, \beta_i$  = intercept and slope of the individual linear regression of patient i

The time-adjusted decline for patient i is then obtained by estimating the patients' individual difference in predicted values between baseline and week 24 from the linear regression.

Pirfenidone — F. Hoffmann-La Roche Ltd

In a further step, the time-adjusted mean FVC decline is estimated by calculating the mean over all individual time-adjusted declines of all patients by treatment arm.

A summary table displaying the mean FVC decline together with two-sided 95% confidence intervals based on percentiles of the t-distribution will be provided by treatment arm. The mean FVC decline in each treatment arm will be compared using a student's t-test with a two-sided significance level  $\alpha$ =0.05

As a sensitivity analysis to the primary analysis, the time-adjusted mean FVC decline will be estimated by a repeated measures mixed model with patient effects fitted as random and day of measurement and treatment fitted as fixed effects. Please refer to <a href="Section-4.5.5">Section 4.5.5</a> for further details.

A detailed description of SAS code to be used for the repeated measures mixed model is provided together with the respective table shell.

#### 4.5.2 <u>Secondary Efficacy Endpoints</u>

For secondary endpoints, all data from baseline until Week 24 will be taken into account for the statistical analysis. In a similar manner to the primary endpoint data, patients who discontinue early will be analyzed based on the data collected until withdrawal.

The secondary efficacy objective for this trial is to evaluate the efficacy of pirfenidone compared with placebo on the basis of the following endpoints:

- Descriptive statistics for values and changes from baseline over time of all spirometry test parameters will be presented.
- The decline of FVC in mL measured by spirometry during site (clinic) visits will be compared between the treatment arms in the same fashion as described for the primary endpoint
- The absolute change in percent predicted FVC measured by spirometry during site visits at week 24 will be compared between the treatment arms using a rank analysis of covariance (ANCOVA). Change from baseline will be used as an outcome variable and standardized rank baseline value will be used as a covariate
- Categorical changes in FVC of >5% and >10% will be compared between the treatment arms using a Cochran-Mantel-Haenszel test stratified by concomitant MMF medication use (Yes/No), and the presence/absence of IPAF as defined by the MDT
- Absolute change from baseline to week 24 in percent predicted DLco will be compared between the treatment arms using a rank ANCOVA. Change from baseline to week 24 will be used as an outcome variable and standardized rank baseline value will be used as a covariate

Pirfenidone — F. Hoffmann-La Roche Ltd

- A summary table presenting the values of DLco (%) and its change from baseline will be presented over time and by treatment arm.
- The absolute change in 6MWD will be analyzed using a rank ANCOVA model.
   The 6MWD recorded at 24 weeks will be used as an outcome variable and standardized rank baseline 6MWD will be used as a covariate
  - A summary table presenting the 6MWD parameters and their change from baseline will be presented over time and by treatment arm.
- The absolute change in UCSD-SOBQ total score will be analyzed using a rank ANCOVA model. The UCSD-SOBQ total score recorded at 24 weeks will be used as an outcome variable and standardized rank baseline UCSD-SOBQ score will be used as a covariate Please see section 4.5.4 for further details.
- The absolute change in Leicester Cough Questionnaire total score will be analyzed using a rank ANCOVA model. The Leicester Cough Questionnaire total score recorded at 24 weeks will be used as the outcome variable and standardized rank baseline Leicester Cough Questionnaire total score will be used as a covariate. Please see section 4.5.4 for further details.
- The change in cough visual analog scale will be analyzed using a rank ANCOVA model. The result recorded at 24 weeks will be used as the outcome variable and the standardized rank baseline result will be used as a covariate. Please see section 4.5.4 for further details.
- The change in total of the SGRQ will be analyzed using a rank ANCOVA model.
  The scores recorded at 24 weeks will be used as outcome variables and the
  standardized rank baseline scores will be used as covariates. Please see section
  4.5.4 for further details.
- The time from randomization to the first occurrence of all-cause non-elective hospitalization and respiratory non-elective hospitalization will be analyzed using Kaplan-Meier (KM) techniques:
  - KM plots of time to first occurrence of the different events will be provided by treatment arm. Frequencies and percentages of patients with events and patients censored will be provided. Descriptive statistics of KM estimates of the time to first occurrence (weeks) will be presented.
  - Log-rank tests based on the time to the first event will be used to compare the two treatment arms.
  - Hazard ratios and corresponding 95% CI will be calculated by applying Cox-proportional hazard models in which the four groups from the two randomization stratification factors are included in the model.
- The incidence of investigator reported acute exacerbations in the two treatment arms will be compared with Fisher's exact test.
- o Incidence of, and time to first, investigator-reported acute exacerbations Pirfenidone F. Hoffmann-La Roche Ltd

- Progression free survival (PFS), defined as the time to the first occurrence of a >10% absolute decline in percent predicted FVC, a >50 m decline of 6MWD, or death from any cause, will be analyzed using Kaplan-Meier techniques:
  - KM plots of time to first occurrence of the combined primary efficacy endpoint will be provided by treatment arm.
  - Frequencies and percentages of patients with events and patients censored will be provided. Descriptive statistics of KM estimates of PFS (weeks) will be presented.
  - The PFS of two randomized treatment arms will be compared with a logrank test.
  - Hazard ratios and corresponding 95% CI will be calculated by applying Cox-proportional hazard models.
- An alternative definition of PFS (also in weeks), namely the time to the first
  occurrence of a >10% relative decline in FVC, non-elective respiratory
  hospitalization, or death, will be analyzed using Kaplan-Meier techniques as
  defined for the point above; and the two treatment arms will be compared with a
  log-rank test. In addition, hazard ratios and corresponding 95% CI will be
  calculated by applying Cox-proportional hazard models
- Time to death from any cause and time to death from respiratory diseases
  assessed by the SOC "Respiratory, thoracic and mediastinal disorders" (in weeks)
  will be analyzed using Kaplan-Meier techniques as defined above; and the two
  treatment arms will be compared with a log-rank test. In addition, hazard ratios
  and corresponding 95% CI will be calculated by applying Cox-proportional
  hazard models.

For all secondary endpoints p-values will be reported in a descriptive fashion. No multiplicity adjustments for statistical testing will be done.

#### 4.5.3 Exploratory Efficacy Endpoints

The exploratory objectives for this trial are to evaluate the role of MMF treatment in ILD and to investigate potential biomarkers associated with fibrosis and ILD.

For the MMF objective, primary and selected secondary endpoints will be investigated by means of a subgroup analyses that stratifies patients according to whether they received MMF treatment. In addition, the overall safety summary will be presented by this subgroup. The selected secondary endpoints are:

- Deaths from any cause and respiratory disease-related
- Hospitalizations from any cause and respiratory disease-related

Pirfenidone — F. Hoffmann-La Roche Ltd

The analysis of these exploratory efficacy endpoints by subgroup are defined under section Section 4.5.6.

The mean FVC decline in each treatment arm will be calculated as in the primary analysis for the subgroups of patients that received MMF treatment and compared using a student's t-test with a two-sided significance level  $\alpha$ =0.05. Exploratory efficacy endpoints are discussed in the sensitivity and subgroup sections (see Section 4.5.5 and Section 4.5.6, respectively).

Moreover, additional categorical analyses for the percent predicted DLco and 6MWD will be presented as exploratory:

- Categorical change of >15% absolute decline from baseline to week 24 in percent predicted DLco will be compared between the treatment arms using a logistic regression.
- Categorical change of >50% absolute decline from baseline to week 24 in 6MWD
   (m) will be compared between the treatment arms using a logistic regression.

For the biomarker objective, assessments of the exploratory biomarkers and their relationship with drug responses will be described in a separate analysis plan.

## 4.5.4 Analyses of Patient-Reported Outcomes

Several PRO assessments will be conducted in this trial, including the UCSD-SOBQ, the Leicester Cough Questionnaire, the cough visual analog scale, and the SGRQ.

PRO data will be collected via questionnaires to document the treatment effect and to evaluate the benefit of pirfenidone. The questionnaires, translated into the local language as required, will be completed in their entirety at specified time points during the trial. To ensure instrument validity and that data standards meet health authority requirements, questionnaires will be self-administered before the patient receives any information on disease status and prior to the performance of non-PRO assessments, unless otherwise specified.

#### St. George's Respiratory Questionnaire (SGRQ)

The St. George's Respiratory Questionnaire (SGRQ) is an index designed to measure and quantifies health-related health status in patients with chronic airflow limitations. The SGRQ is a 50-item questionnaire, addressing the frequency of respiratory symptoms (items 1-8), the patient's current state (sections 9-16). From the 50 items a total score, as well as three component scores (Symptoms, Activities, Impacts) will be derived. The total score ranges from 0, presenting the best possible health status to 100, presenting the worst possible health status.

The change in SGRQ total score will be of primary interest when assessing health-related quality of life (HRQoL).

Pirfenidone — F. Hoffmann-La Roche Ltd

The analysis of PROs assessed by SGRQ total score and by SGRQ component scores for symptoms, activity, and impacts will be analyzed as follows:

- The absolute score values and changes from baseline for the total and each subscore will be presented descriptively over time by treatment arm.
- Changes from baseline to week 24 or early discontinuation visit will be compared between the treatment arms using a rank ANCOVA with change from baseline as outcome variable and standardized rank baseline value as covariate. This analysis will be done only for the total score.

The SGRQ and the details for calculating the score can be found in Appendix 3.

# The University of California, San Diego-Shortness of Breath Questionnaire (UCSD-SOBQ)

The University of California, San Diego-Shortness of Breath Questionnaire (UCSD-SOBQ) is a symptom-specific, 24-item, patient-self-administered questionnaire that assesses shortness of breath while doing a variety of activities of daily living. Each of the 24 activities are rated on how dyspnea affects the activity on a 6-point scale: 0 = None at all to 5 = Maximal or unable to do because of breathlessness. The scores will be summarized to a total score, ranging from 0 - 120.

The total score of the UCSD SOBQ will be summarized as follows:

- The absolute total scores and changes from baseline will be presented descriptively over time by treatment arm.
- Changes from baseline to week 24 or early discontinuation visit will be compared between the treatment arms using a rank ANCOVA with change from baseline as outcome variable and standardized rank baseline value as covariate.

Additional details on the UCSD SOBQ can be found in Appendix 3

## The Leicester Cough Questionnaire

The Leicester Cough Questionnaire is a patient-reported questionnaire evaluating the impact of cough on quality of life. The questionnaire comprises 19 items and takes 5 to 10 minutes to complete. Each item assesses symptoms, or the impact of symptoms, over the last 2 weeks on a seven-point Likert scale. Scores in three domains (physical, psychological and social) are calculated as a mean for each domain (range 1 to 7). A total score (range 3 to 21) is also calculated by adding the domain scores together. Higher scores indicate better quality of life.

The total score and the physical, psychological and social domain scores of the Leicester Cough Questionnaire will be analyzed as follows:

Pirfenidone — F. Hoffmann-La Roche Ltd

- The scores and changes from baseline will be presented descriptively over time by treatment arm.
- Changes from baseline to week 24 or early discontinuation visit will be compared between the treatment arms using a rank ANCOVA with change from baseline as outcome variable and standardized rank baseline value as covariate. This analysis will be done only for the total score.

Details on calculating the domain scores can be found in Appendix 3

### The Cough VAS

This visual analogue scale is designed to help us learn about the severity of your cough. This scale is 100mm (10cm) in length.

The cough VAS score will be summarized descriptively by visit and treatment arm. The change in cough VAS will be analyzed using a rank ANCOVA model. The change in VAS score for cough recorded at 24 weeks will be used as the outcome variable and the standardized rank baseline result will be used as a covariate. Please refer to <a href="Appendix 3">Appendix 3</a> for further details.

## 4.5.5 <u>Sensitivity Analyses</u>

As a sensitivity analysis to the primary analysis, the time-adjusted mean FVC decline will be estimated by a repeated measures mixed model with patient effects fitted as random and day of measurement and treatment fitted as fixed effects. Corresponding model estimates will be tabulated.

A second model adding the stratification factors as covariates will be also presented.

Additional covariates such as gender, age and height that are used to determine FVC % predicted will be examined as well.

Additionally, the impact of different assumptions with respect to the variance-covariance matrix underlying the repeated measures mixed model will be investigated.

#### 4.5.6 Subgroup Analyses

Subgroup analyses will be conducted for the exploratory endpoint, as described in Section 4.5.3. The following subgroups will be based on:

- The four groups resulting from combinations of the two stratification factors:
  - Concomitant MMF treatment (yes/no)
  - Presence/absence of IPAF as defined by the MDT
- Gender: Male, Female

Pirfenidone — F. Hoffmann-La Roche Ltd

- Age (years): <65 years, ≥ 65 years</li>
- Percent predicted FVC at Baseline: <65%, ≥65% to < 80%, ≥80%</li>
- Percent predicted DLco at Baseline: <35%, ≥35%</li>
- Body weight: <60 kg, ≥60 kg</li>

#### 4.6 PHARMACOKINETIC AND PHARMACODYNAMIC ANALYSES

No pharmacokinetic or pharmacodynamic analyses are planned for this study.

#### 4.7 SAFETY ANALYSES

All safety analyses of data from the double-blind treatment period will be based on the safety population, i.e., the safety population will include all randomized patients who received at least one dose of trial treatment, with patients grouped according to treatment received. Safety data from the follow-up period will be summarized based on the safety follow-up population.

The safety objective for this trial is to evaluate the safety of pirfenidone vs. placebo.

No formal statistical testing will be performed for safety parameters.

Data collected during the 12-month safety follow-up will be analyzed separately (see section 4.8).

The safety analysis will involve investigating the nature, frequency, severity, and timing of treatment-emergent adverse events. The specific parameters that will be investigated include all adverse events, adverse events Grade ≥3 according to the NCI CTCAE version 4.03, adverse events of special interest, and serious adverse events. The primary interest in this trial will be adverse events Grade ≥3 related to pirfenidone or placebo.

Prior to the first administration, only serious adverse events caused by a protocol-mandated intervention will be recorded. These adverse events will be listed.

The incidence, type, and severity of adverse events will be summarized according to the primary System Organ Class (SOC) and within each SOC, by the Medical Dictionary for Regulatory Activities (MedDRA) version 20.1 or higher preferred term.

Adverse events Grade ≥3, adverse events of special interest, and serious adverse events will be analyzed in a similar way to all adverse events.

Descriptive statistics will be presented for dose modifications and treatment interruptions. Adverse events leading to treatment interruption or dose modification will also be summarized.

Pirfenidone — F. Hoffmann-La Roche Ltd

Laboratory parameters including hematology and the chemistry panel will be presented in shift tables of NCI-CTCAE version 4.03 grade at baseline vs. worst grade during treatment period. The laboratory parameters will be presented according to means, standard deviation, minimum, and maximum. Selected laboratory parameters will be also graphically presented over time. Liver abnormalities for the parameters total bilirubin, alkaline phosphatase, ALAT (SGPT) and ASAT (SGOT)) will be also presented.

The results from the 12-lead ECGs will be summarized and presented.

## 4.7.1 <u>Exposure of Study Medication</u>

All analyses described in this section refer to the data collected in the drug-log for the double-blind randomized treatment period. Unknown doses will be excluded from the exposure analyses.

#### 4.7.1.1 Treatment duration

Summaries of dosing, treatment duration, dose interruptions or reductions during the randomized double-blind treatment period will be provided for each treatment arm separately.

The overall treatment duration (weeks), including and excluding dose interruptions, will be summarized descriptively by treatment arm. The overall treatment duration including dose interruptions will be defined as follows:

[Date of last positive dose of randomized treatment received (pirfenidone/placebo) – date of first intake of randomized treatment) + 1)] / 7.

The overall treatment duration excluding dose interruptions will be derived from the treatment administration panels using the time windows described above, considering only days on treatment. i.e. positive dose.

Details on treatment administration, reductions or interruptions will be listed.

#### 4.7.1.2 Doses and Dose modifications or interruptions

The total dose (mg), the average daily dose (mg/d) and the last dose administered (mg/d) will be presented descriptively for each of the study treatments.

The average daily dose will be calculated by summing up the number of capsules taken, divided by the overall treatment duration including dose interruptions as defined above.

Numbers and proportions of patients with at least one dose modification, or drug interruption, will be presented for each treatment arm separately. Numbers and proportions of patients with 1, 2, 3 or more dose modifications, or treatment interruptions, will be given.

Pirfenidone — F. Hoffmann-La Roche Ltd

The total number of dose modifications, reductions or treatment interruptions, will be presented together with numbers and frequencies of reasons for dose modification, reduction or treatment interruption.

Dose modifications, reductions or treatment interruptions will be presented as given in the drug logs dose strength and number of capsules taken.

In addition, dose intensity will be analyzed descriptively by treatment arm over time. For calculation of dose intensities, the time from first administration of randomized treatment to the end date of randomized treatment will be considered. The following formula will be used for calculation:

Dose intensity (DI) = (total dose received / total dose planned)\*100.

## 4.7.2 <u>Adverse Events</u>

Verbatim descriptions of adverse events (AEs) will be mapped to a preferred term (PT) and system organ class (SOC) using the Medical Dictionary for Regulatory Agencies (MedDRA®). MedDRA version 20.1 or above and related SMQ lists will be used for coding.

AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03. For AEs of varying severity, the most severe grade as documented on the eCRF will be used in the summaries. An AE will be considered severe if the most extreme grade will be larger or equal to 3.

After informed consent has been obtained but prior to initiation of trial treatment, only serious adverse events caused by a protocol-mandated intervention (e.g. invasive procedures such as biopsies, discontinuation of medications) should be reported. All adverse events will be reported until 28 days after the last dose of study drug. After this period, the Investigator should report any SAEs that are believed to be related to prior study drug treatment.

For safety analysis of the double-blind treatment period treatment-emergent adverse events (TEAEs) will be defined as:

 AEs that started or worsened on or after first intake of randomized treatment until last positive dose of randomized treatment + 28 days

Adverse events that are reported after informed consent but before the first intake of randomized treatment will be considered as non-treatment-emergent AEs. These might include AEs that occur during the screening period.

Post-treatment AEs are not expected to occur, but will be defined as AEs that are reported more than 28 days after the last dose of randomized treatment for patients who do not enter the 12-month safety follow-up period. Those AEs will be listed.

Pirfenidone — F. Hoffmann-La Roche Ltd

The analysis of AEs within the framework of the primary study analysis will focus on treatment-emergent AEs (TEAE).

An overview of patient safety profile will present the number and proportion of patients in each treatment arm experiencing:

- Any and any related treatment-emergent adverse events (TEAE)
- Any and any related serious treatment-emergent adverse events (serious TEAE)
- Any and any related severe treatment-emergent adverse events (TEAEs ≥ Grade 3)
- Any and any related TEAE of special interest (AESI). Adverse events of special interest for this trial include the following:

Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's law: [ALT or AST >3 x ULN + total bilirubin >2 x ULN]

- Any and any related hepatic side effects: elevations in ALT and AST >3 x ULN at the same timepoint in the study.
- Any and any related gastrointestinal (GI) disorder (MedDRA SOC: GI Disorders)
- Any and any related photosensitivity (MedDRA Preferred terms Photodermatosis, Photosensitivity reaction, Pruritus, Pruritus allergic, Pruritus generalized). Potential updates in those terms will be needed in case the MedDRA version changes.
- Any and any related rash (MedDRA Preferred terms Nodular rash, Rash, Rash erythematous, Rash generalized, Rash macular, Rash maculo-papular, Rash papular, Rash pruritic, Rash follicular, Exfoliative Rash, Solar dermatitis, Solar urticarial, Sunburn, Erythema, Dry skin). Potential updates in those terms will be needed in case the MedDRA version changes.
- Angioedema (MedDRA preferred term Angioedema).
- Dizziness (MedDRA preferred term Dizziness).
- Fatigue (MedDRA preferred term Fatigue).
- Weight loss (MedDRA preferred term Weight loss).
- Increase in QT interval: In the event of a QTcF interval of >500 ms or an increase from baseline of >60 ms, a repeat ECG must be obtained within 24 hours.
- Any and any related TEAE leading to death

Pirfenidone — F. Hoffmann-La Roche Ltd

- Any and any related TEAE leading to treatment discontinuation
- Any grade 3-4 laboratory liver test results
  - o ASAT (SGOT) results
  - o ALAT (SGPT) results
  - o alkaline phosphatase results
  - o total bilirubin results

The incidence of TEAEs, related TEAEs, non-serious TEAEs, serious TEAEs, related serious TEAEs, grade 3-5 TEAEs and TEAEs leading to treatment discontinuation, dose modification or death will be summarized by treatment arm, by system organ class (SOC) and preferred term (PT) on the basis of the safety population. Frequencies and percentages of patients experiencing (at least) one event in the respective category will be presented by decreasing frequencies. If patients have more than one AE within a SOC or PT they will be counted only once for the respective SOC or PT. Additionally the total numbers of TEAEs will be provided for each SOC and overall.

Similar summary presentations will be provided for the incidence of TEAEs leading to dose reduction and drug interruption and TEAEs leading to hospitalization.

Non serious Treatment-emergent Adverse Events with >5% frequency will be also presented by SOC and PT. In addition, Serious Treatment-emergent Adverse Events, Fatal serious TEAEs and serious TEAEs related to pirfenidone or placebo will be presented in the same table by SOC and PT.

A summary table presenting the numbers and frequency of patients with TEAEs by most extreme CTCAE Grade (Grade 1, Grade 2, Grade 3, Grade 4 and Grade 5) will be provided for each SOC and PT by treatment arm. In case the most extreme intensity is missing, it will be replaced by the initial intensity. If both most extreme and initial intensity are missing, the AE will be included in the Grade ≥3 category and a category for "missing" will be added.

Further, Kaplan-Meier curves for time to onset of first adverse event of the most relevant related TEAEs will be provided by treatment arm when the number of events are enough to do the analyses. These will include the following PTs or groups of AEs: Nausea, Diarrhoea, Weight decreased, Fatigue, Decreased appetite, and photosensitivity, or rash. In addition, the analysis will be done for the SOC GI.

All adverse event data will be listed by patient number and study day of onset including a flag variable for identifying the period of the event (double-blind treatment period or safety follow-up period). If the AE does not belong to any of the periods, the period flag will be missing.

Pirfenidone — F. Hoffmann-La Roche Ltd

## **4.7.3** Deaths

Numbers and frequencies of deaths and of deaths occurring within 28 days after the last dose of double-blind treatment will be presented by treatment arm.

All information associated with deaths collected in eCRF panel on study discontinuation will be listed. A flag variable will be included in the listing specifying the study period when the death occurred.

### 4.7.4 Laboratory Data

All of the laboratory tests will be conducted by the trial site's local laboratory.

All parameters will be graded according to NCI CTCAE (CTEP 2010), version 4.03, if applicable. Laboratory parameters that cannot be graded according to the corresponding NCI CTCAE version 4.03 will be assessed with respect to normal range (low, normal, high).

Laboratory parameters including hematology and the chemistry panel will be presented in shift tables of NCI-CTCAE version 4.03 grade at baseline versus worst grade during randomized double-blind treatment period. The laboratory parameters will be presented according to means, standard deviation, minimum, and maximum. Selected laboratory parameters will be also graphically presented over time.

The following laboratory samples will be collected:

- Hematology: white blood cell (WBC) count, red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, differential count (neutrophils, eosinophils, basophils, monocytes, lymphocytes, other cells).
- Chemistry panel (serum or plasma): sodium, potassium, chloride, bicarbonate, glucose, blood urea nitrogen (BUN) or urea, creatinine, total protein, albumin, phosphorus, calcium, total and direct bilirubin, alkaline phosphatase, ALT, AST, uric acid, lactate dehydrogenase (LDH).

Clinical laboratory values will be presented separately for CTCAE-gradable and non-CTCAE gradable parameters by laboratory panel (hematology, serum chemistry). For laboratory analyses, visits will be assigned to visit windows as described in <u>Section 4.9</u>. This will also be valid for possible unscheduled visits. In case that multiple evaluable assessments occur within the same visit, the nearest to midpoints value will be used for analyses.

The following summaries will be prepared:

For each laboratory parameter, descriptive statistics of laboratory values at each scheduled visit (derived as described above), and absolute changes from baseline to post-baseline will be presented by treatment arm.

Pirfenidone — F. Hoffmann-La Roche Ltd

Shift tables presenting categorical changes in CTCAE grade from baseline to worst grade recorded during the double blind period, in the indicated direction, will be provided for CTCAE-gradable parameters by treatment arm. If no CTCAE grade is available for a specific laboratory variable, shift tables will present worst changes with respect to normal range category (low, normal, high).

Liver abnormalities (total bilirubin, alkaline phosphatase, ALAT (SGPT), ASAT (SGOT)) of Grade 3 and 4 will be presented showing numbers and percentages of patients for each parameter separately. Line graphs of liver parameters will be provided.

### 4.7.5 Vital Signs

Vital signs will include measurements of respiratory rate (breaths/min), pulse rate (beats/min), and systolic and diastolic blood pressures (mmHg) while the patient is in a seated position, temperature (C) and weight (kg). Vital signs will be assigned to visit windows as per <a href="Section 4.9">Section 4.9</a>. Descriptive statistics will be used to summarize vital signs data at baseline and at each scheduled post-baseline visit, and for the absolute change from baseline to each scheduled post-baseline visit by treatment arm during double-blind period.

#### 4.7.6 ECG

Single ECG recordings will be obtained at specified time points, as outlined in the Schedule of Assessments (see <a href="Appendix 2">Appendix 2</a>), and may be obtained at unscheduled time points as indicated.

The following should be recorded in the appropriate eCRF: heart rate (beats/min), RR interval (msec), QRS interval (msec), PR duration (msec), uncorrected QT interval (msec), and the QTcF based on the machine readings of the individual ECG tracings. Any morphologic waveform changes or other ECG abnormalities must be documented on the eCRF. If considered appropriate by the Sponsor, ECGs may be analyzed retrospectively at a central laboratory.

QTcF values of the safety population will be assigned to the following intervals: < 500 ms, 500–550 ms, and > 550 ms. Numbers and percentages of patients with their maximum QTcF interval category will be summarized by treatment arm over time. Absolute changes from the Baseline to each post-baseline visit in QTcF values will be categorized to < 31 ms, 31–60 ms, and > 60 ms. Numbers and percentages of patients in each category will be presented by treatment arm for each post-baseline visit or treatment discontinuation. Planned visits will be used for presentations.

Descriptive statistics for heart rate, RR interval, QRS interval, PR duration, uncorrected QT interval, and the QTcF will be presented for each visit by treatment arm.

A listing containing ECG data will be presented.

#### 4.8 SAFETY FOLLOW-UP ANALYSES

Data collected during the safety-follow-up period will be analyzed in the following way.

Pirfenidone — F. Hoffmann-La Roche Ltd

Adverse events during the 12-month safety follow-up period for pirfenidone treatment will be defined as:

 AEs that started or worsened on or after the date of safety follow-up period start until the end of the safety follow-up.

The safety follow-up population will be used for these analyses.

Summary tables for the incidence of AEs, related AEs, serious AEs, related serious AEs, severe AEs and severe related AEs will be summarized by system organ class (SOC) and preferred term (PT). Frequencies and percentages of patients experiencing (at least) one event in the respective category will be presented by decreasing frequencies. If patients have more than one AE within a SOC or PT they will be counted only once for the respective SOC or PT. Additionally, the total numbers of AEs will be provided for each SOC and overall. As with the end of the double-blind treatment period, an overview of safety will also be presented.

Pirfenidone exposure during safety-follow-up will be analyzed in a similar fashion as described in section 4.7.1 with regard to treatment duration and amount of drug intake.

Data of laboratory assessments (AST, ALT, bilirubin, and alkaline phosphatase) and vital signs during safety-follow-up period will be analyzed in a similar fashion as described in section 4.7.4 and 4.7.5.

Data will be presented by randomized treatment labeled as 'Randomized Pirfenidone' and 'Randomized Placebo'.

#### 4.9 MISSING DATA

In general, missing data will not be imputed. Exceptions will be made for the data related to adverse events and concomitant medications as described below.

For adverse events, missing start dates will only be imputed for determination of whether the adverse event is considered to be treatment-emergent or not.

Incomplete or missing onset dates will be imputed to the earliest date possible (using any reliable portions of the onset date that are available). The onset day is considered unreliable if the month or year portions of the date are missing.

In case the month portion of the AE start date is missing, the AE start date will be imputed to the earliest day possible by using the following principles:

- If Treatment Start Date is missing, then the AE Start Date will be imputed as 01-01-YYYY or the earliest date regarding signature of informed consent, screening date or randomization date, whichever is the later one
- When the Treatment Start Date is not missing, and the years of AE Start Date and Treatment Start Date coincide, the AE onset date will be set to the Treatment Start Date

Pirfenidone — F. Hoffmann-La Roche Ltd

When the Treatment Start Date is not missing, and the years of the AE Start
Date and the Treatment Start Date do not coincide, then the AE Start Date will be
imputed as 01-01-YYYY or the earliest date regarding signature of informed
consent, screening date or randomization date, whichever is the later one

In case the day portion of the AE Start Date is missing, the AE Start Date will be imputed to the earliest day possible as follows:

- If the Treatment Start Date is missing, then the AE Start Date will be imputed as 01-MMM-YYYY or the earliest date regarding signature of informed consent, screening date or randomization date, whichever is the later one
- When the treatment date is not missing, and the years and months from the AE Start Date and the Treatment Start Date coincide, the AE onset date will be set to the Treatment Start Date
- When the Treatment Start Date is not missing, and AE Start Date is after the Treatment Start Date according to the given year or month, then the AE Start Date will be imputed as 01-MMM-YYYY

If the AE stop date is missing, then the event will be assumed to be ongoing and a stop date will not be imputed.

In the case the treatment end date is missing and it cannot be judged whether the event occurred during the period of Treatment Start Date to Treatment End Date plus 28 days, the AE will be considered treatment-emergent as long as it is not flagged as prior AE.

For imputation and handling of missing intensity or relationship to study medication, please see Section 4.7.2.

All other missing or incomplete adverse event data will be left as missing.

For concomitant medications, missing start or end dates will only be imputed to determine whether the medication is considered to be prior, on-treatment, post-treatment.

In general if only the day is missing from the start date then the missing day will be imputed as 01-MMM-YYYY unless the month is the same month as the start of study medication in which case the missing date will be imputed as the treatment start date.

If both the day and month are missing from the start date then the start date will be imputed as 01-JAN-YYYY.

If both the day and month are missing from the start date year is the same as treatment start date then the start date will be imputed as 'treatment start date', but if the year is after treatment start date, the start date will be imputed as 01-JAN-YYYY.

If the day, month and year are all missing from the start date then the start date will be imputed as 01-JAN for the year in which the patient was recruited to the study.

Pirfenidone — F. Hoffmann-La Roche Ltd

If the day, month and year are all missing from the start date then the start date will be imputed as 'treatment start date'.

If an incomplete stop date has both the year and month present, the day will be imputed as the last day of the month or date of discontinuation/death.

If the AE is ongoing at time of primary analysis, concomitant medication will be summarized for the double-blind treatment period and safety follow-up.

#### 4.10 VISIT WINDOWS

Visit windows for double-blind treatment period will be applied to vital signs and laboratory data and the derived visits will be used in the by-visit summarizations. If multiple observations fall within the same visit window, the observation with the nearest to midpoint value will be used in the analysis, if not stated otherwise. If subjects discontinue from the double-blind treatment period early the data will be assigned to the early discontinuation visit. The date of early discontinuation will be considered as the target date.

The "Baseline" visit is a derived data point to identify baseline values which are used to calculate the change from baseline values. Baseline is defined in section 4.2.2

The End of Treatment [EOT] visit will either be a copy of early discontinuation records for patients who prematurely discontinued double-blind treatment period or Week 24 records for patients who completed the double-blind treatment period.

Table 2 Visit Windows

| Analysis Visit [AVISITN] | Target Day | Analysis Window (scheduled Study Days) |
|---|---|---|
| Baseline [0] | 1 | Last valid assessment prior to first intake of randomized study drug (pirfenidone/placebo). |
| | | Generally, it is assumed that measurements referring to the Day 1 (Week 1) visit have been performed before randomized study drug (pirfenidone/placebo) was given. |
| Week 4 [4] | 28 | One day after first dose of randomized treatment to 42 |
| Week 8 [8] | 56 | 43 to 70 |
| Week 12 [12] | 84 | 71 to 98 |
| Week 16 [16] | 112 | 99 to 126 |
| Week 20 [20] | 140 | 127 to 154 |

Pirfenidone — F. Hoffmann-La Roche Ltd

| Week 24 [24] | 168 | 155 to a maximum of 195 if the patient did not early discontinued. |
|---|---|---|
| Early discontinuation [25] | Not applicable | As occurred |
| End of treatment (EOT) [26] | Not applicable | As occurred |
| Follow-up visit (FUP1) [27] | Not applicable | As occurred |
| Safety follow-up visits(SFUP) [28] | Not applicable | As occurred: Month 1 to 6: Monthly visits Month 7 to 12: Approximately every 3 months |
| Additional Safety follow-up visit [29] | Not applicable | As occurred:<br>up to 12 months plus 28 days |

#### 4.11 INTERIM ANALYSES

An independent Data Monitoring Committee (iDMC) will review safety data and advise on trial conduct at least three times during the trial. A first meeting is planned 6 months after start of recruitment, and subsequently at 12 and 18 months. Additional ad hoc meetings or data reviews can be requested at any time by the iDMC or the Sponsor, if warranted. The iDMC will be an independent body who will recommend to continue, modify or stop the trial at each meeting. The procedures that will be used by the iDMC will be detailed in an iDMC charter.

No formal interim analyses for efficacy are planned.

#### 4.12 BIOMARKER ANALYSES

Certain biomarkers may be differentially expressed in patients with unclassifiable ILD and may change as a result of pirfenidone treatment (e.g., possibly cytokines, chemokines, and other cellular and molecular markers of lung injury and fibrosis). The blood biomarker samples that are being obtained for this trial may help identify the serum and plasma proteins or blood ribonucleic acid (RNA) biomarkers related to disease progression and/or may be used to assess their response to pirfenidone therapy.

Transcriptomic and protein markers associated with the molecular pathways and cellular processes of lung injury and fibrosis will be measured. This may include, but is not restricted to, measurement of CCL18, MMP7, CXCL13, and COMP.

Serum, plasma, and whole blood (for RNA analysis) samples will be acquired at baseline, Week 4, Week 12, Week 24, and at the Early Treatment Discontinuation Visit (see the Schedule of Assessments, Appendix 2).

Optional Research Biosample Repository (RBR) whole blood samples for deoxyribonucleic acid (DNA) extraction, described in Section 4.5.8 of the protocol, will

Pirfenidone — F. Hoffmann-La Roche Ltd

also be collected at baseline to examine genetic polymorphisms and their potential role in the pathogenesis and associated clinical outcomes of unclassifiable ILD.

Biomarkers associated with fibrosis and ILD will be evaluated in plasma, serum, and whole blood ribonucleic acid (RNA) and deoxyribonucleic acid (DNA) samples.

Analyses on biomarker data will not be in the scope of this SAP, but will be planned and described separately.

Pirfenidone — F. Hoffmann-La Roche Ltd

#### **REFERENCES**

Antoniou KM, Margaritopoulos GA, Tomassetti S, Bonella F, Costabel U, Poletti V. Interstitial lung disease. Eur Respir Rev 2014;23:40–54.

Khanna D, Albera C, Fischer A, et al. An open-label, phase II study of the safety and tolerability of pirfenidone in patients with scleroderma-associated interstitial lung disease: the LOTUSS trial. J Rheumatol 2016;epub.

Collard HR, Ryerson CJ, Corte TJ, et al. Acute exacerbation of idiopathic pulmonary fibrosis. An international working group report. Am J Respir Crit Care Med 2016;194:265–75.

Ryerson CJ, Urbania TH, Richeldi L, et al. Prevalence and prognosis of unclassifiable interstitial lung disease. Eur Respir J 2013;42:750–7.

Fischer A, Brown KK, du Bois RM, et al. Mycophenolate mofetil improves lung function in connective tissue disease-associated interstitial lung disease. J Rheumatol 2013;40:640–6.

Eakin EG, Resnikoff PM, Prewitt LM, et al. Validation of a new dyspnea measure: the UCSD Shortness of Breath Questionnaire. University of California, San Diego. Chest. 1998 Mar;113(3):619-24.

Ries AL, Minimally clinically important difference for the UCSD Shortness of Breath Questionnaire, Borg Scale, and Visual Analog Scale. COPD. 2005 Mar;2(1):105-10.

Jones PW, Quirk FH, Baveystock CM, The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7.

Nishimura K, Tsukino M, Hajiro T, Health-related quality of life in patients with chronic obstructive pulmonary disease. Curr Opin Pulm Med. 1998 Mar;4(2):107-15.

St. George's Respiratory Questionnaire: <a href="http://www.healthstatus.sgul.ac.uk/sgrq">http://www.healthstatus.sgul.ac.uk/sgrq</a>

S S Birring, B Prudon, A J Carr, S J Singh, M D L Morgan, I D Pavord, Development of a symptom specific health status measure for patients with chronic cough: Leicester Cough Questionnaire (LCQ). Thorax 2003;58:339-343.

Pirfenidone — F. Hoffmann-La Roche Ltd

# Appendix 1 PROTOCOL SYNOPSIS

TITLE: MULTICENTER, INTERNATIONAL, DOUBLE-BLIND, TWO-

ARM, RANDOMIZED, PLACEBO-CONTROLLED PHASE II

TRIAL OF PIRFENIDONE IN PATIENTS WITH

**UNCLASSIFIABLE PROGRESSIVE FIBROSING ILD** 

PROTOCOL MA39189

**NUMBER:** 

**VERSION NUMBER:** 3.0

**EUDRACT NUMBER:** 2016-002744-17

**IND NUMBER:** 67284

**TEST PRODUCT:** Pirfenidone (RO0220912)

PHASE:

**INDICATION:** Fibrotic interstitial lung disease of unknown origin

**SPONSOR:** F. Hoffmann-La Roche Ltd

#### **Objectives and Endpoints**

This trial will evaluate the efficacy and safety of pirfenidone in patients with fibrosing interstitial lung disease (ILD) who cannot be classified with moderate or high confidence into any other category of fibrosing ILD by multidisciplinary team (MDT) review ("unclassifiable" ILD).

#### **Efficacy Objective**

The primary efficacy objective for this trial is to evaluate the effect of pirfenidone vs. placebo on lung function parameters on the basis of the following endpoint:

• Rate of decline in forced vital capacity (FVC) measured in mL by daily handheld spirometer over the 24-week double-blind treatment period.

#### **Safety Objective**

The safety objective for this trial is to evaluate the safety of pirfenidone vs. placebo on the basis of the following endpoints:

- Nature, frequency, severity, and timing of treatment-emergent adverse events
- Dose reductions and treatment interruptions
- Clinical laboratory test results
- 12-lead electrocardiograms (ECGs)
- Withdrawals from trial treatment or trial discontinuations.

Pirfenidone — F. Hoffmann-La Roche Ltd

## **Exploratory Objective**

One exploratory objective for this trial is to evaluate the role of MMF (mycophenolate mofetil/sodium or mycophenolic acid) treatment in ILD on the basis of the following endpoint:

 Efficacy and safety data from subgroups of patients who did or did not receive MMF treatment.

In addition, exploratory biomarkers associated with fibrosis and ILD will be evaluated in plasma, serum, and whole blood ribonucleic acid (RNA) and deoxyribonucleic acid (DNA) samples.

#### **Trial Design**

#### **Description of Trial**

This is a multicenter, international, double-blind, two-arm, randomized, placebo-controlled Phase II trial in patients with fibrosing ILD who cannot be classified with moderate or high confidence into any other category of fibrosing ILD by MDT review ("unclassifiable ILD"). Patients will be randomized in a 1:1 ratio, on a double-blind basis using a stratified algorithm, to receive either pirfenidone (801 mg three times daily [TID]) or placebo. The randomized patients will be stratified by concomitant MMF treatment (yes/no), the presence/absence of interstitial pneumonia with autoimmune features (IPAF) as defined by the MDT.

Most established MDTs have access to clinical, radiologic, and pathology expertise, and should have a sufficient case load of ILDs per year. Access to rheumatology expertise will be at the discretion of the MDT.

In total, approximately 90 clinical centers (sites) in Australia, Europe, the Middle East, and North America are expected to enroll approximately 250 patients. Patients who are withdrawn from the trial will not be replaced. The trial design is represented in Appendix 3

Patient Reported Outcome Questionnaire

After discussing the risks and benefits of the trial with the investigator and providing informed consent, patients will be required to taper and/or discontinue all prohibited medications (Section 4.4.2 of the CSP) in the 28 days prior to the start of screening during the washout period. If a prohibited medication must be tapered, the process must start early enough so that the patient discontinues the medication in the 28 days prior to the start of screening. After completing the washout period, patients will enter screening, which lasts up to 21 days. During screening, patients will be evaluated for eligibility based on the inclusion and exclusion criteria. Patients not taking a prohibited medication will forgo the washout period and directly enter screening.

At the end of screening, patients will be randomized (Day 1) to receive either pirfenidone or placebo (1:1 ratio).

Following treatment initiation, the daily dosage will be titrated to the full dosage of nine capsules per day over a 14-day period. After the titration period, trial treatment will continue through Week 24 and monitoring will be conducted by trial visits. Patients should remain on a stable maintenance dose for the duration of the treatment period unless the dose is reduced or dosing is interrupted to manage an adverse event. Any patient with an actual or anticipated interruption of trial treatment for a period of ≥28 consecutive days will be reported by telephone to Roche's medical monitor or designee to discuss the circumstances of the case. Once the patient restarts trial treatment, the

Pirfenidone — F. Hoffmann-La Roche Ltd

dose must be re-titrated over 14 days. A Follow-up Visit will occur 28 days after the end of the 24-week double-blind treatment period.

After completion of the double-blind treatment period and the Follow-up Visit at Week 28, the Sponsor will offer the possibility to the patients to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. During the safety follow up period, the patients should be evaluated by the investigator initially at monthly visits during the first 6 months and subsequently at each visit occurring approximately every 3 months thereafter. A final Follow-up Visit will be performed at the end of the safety period, 28 days after the last open-label dose.

Table 1 Titration Schedule

| Treatment Days | Dosage |
|-------------------|---------------------------------------------|
| Days 1 through 7 | One capsule three times daily with meals |
| Days 8 through 14 | Two capsules three times daily with meals |
| Day 15 onwards | Three capsules three times daily with meals |

The Sponsor will provide trial treatment on a double-blind basis. The design that will be utilized in this trial is shown in Appendix 3 Patient Reported Outcome Questionnaire below.

Figure 1 Trial Schema



<sup>&</sup>lt;sup>1</sup> Patients will be required to taper and/or discontinue all prohibited medications in the 28 days prior to the start of screening during the washout period. Patients not taking a prohibited medication will forgo the washout period and directly enter screening.

D=Day; ICF=informed consent form

Pirfenidone — F. Hoffmann-La Roche Ltd

<sup>&</sup>lt;sup>2</sup> Informed consent must be documented before any trial-specific screening procedure is performed, and may be obtained either at the Washout or Screening Visits.

<sup>&</sup>lt;sup>3</sup> After completion of the double-blind treatment period and the Follow-up Visit at Week 28, the Sponsor will offer the possibility to the patients to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. A final Follow-up Visit will be performed at the end of the safety period, 28 days after the last open-label dose.

The primary objective of this trial is to evaluate the efficacy of pirfenidone vs. placebo on lung function parameters by examining the rate of decline in FVC (measured in mL). A handheld spirometry device will be used by the patient to measure daily FVC at home. Confirmatory site (trial center) based FVC measurements will be conducted every 4 weeks (see Schedule of Assessments, <a href="Appendix 2">Appendix 2</a>). Blood samples will be obtained from patients in order to analyze clinical laboratory values and biomarkers.

#### **Number of Patients**

Approximately 250 patients with unclassifiable fibrosing ILD will be enrolled in this trial.

## **Target Population**

#### Inclusion Criteria

Patients must meet the following criteria for trial entry:

- 1. Signed Informed Consent Form
- 2. Age ≥18-85 years
- 3. Able to comply with the trial protocol, according to the investigator's judgment
- 4. Confirmed fibrosing ILD which, following MDT review, cannot be classified with either high or moderate confidence as a specific idiopathic interstitial pneumonia or other defined ILD (e.g. chronic hypersensitivity or connective tissue disease-ILD [CTD-ILD])
- Progressive disease as considered by the investigator using the following definition:
  - a. Patient deterioration within the last 6 months, which is defined as:
    - i. A rate of decline in FVC >5% OR
    - ii. Significant symptomatic worsening not due to cardiac, pulmonary, vascular, or other causes.
- 6. Extent of fibrosis >10% on high-resolution computed tomography (HRCT; visual scoring) within the last 12 months
- 7. FVC ≥45% of predicted value
- 8. Diffusing capacity of the lung for carbon monoxide (DLco) ≥30% of predicted value
- 9. Forced expiratory volume in 1 second (FEV<sub>1</sub>)/FVC ratio ≥0.7
- 10. 6-minute walk distance (6MWD) ≥150 meters
- 11. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of <1% per year during the treatment period and for at least 58 days after the last dose of trial treatment:
  - a. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
  - b. Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives including those that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices

Pirfenidone — F. Hoffmann-La Roche Ltd

c. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

- a. With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 118 days after the last dose of trial treatment. Men must refrain from donating sperm during this same period
- b. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 118 days after the last dose of trial treatment to avoid exposing the embryo
- c. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

#### **Exclusion Criteria**

Patients who meet any of the following criteria will be excluded from trial entry:

- 1. Diagnosis with moderate or high confidence of nonspecific interstitial pneumonia (NSIP) and any ILD with an identifiable cause such as CTD-ILD, chronic hypersensitivity pneumonitis (cHP), or others
- 2. Diagnosis of idiopathic pulmonary fibrosis (IPF) independent of the confidence level
- History of unstable angina or myocardial infarction during the previous 6 months
- 4. Pregnant or lactating, or intending to become pregnant during the trial
- 5. A positive urine pregnancy test, which was confirmed with a positive serum pregnancy test. Women with a confirmed pregnancy will be excluded from trial participation and must discontinue trial treatment
- 6. Treatment with high dose systemic corticosteroids (i.e., >15 mg/d of prednisolone or equivalent), or any immunosuppressant other than MMF, at any time at least 4 weeks prior to screening. Patients being treated with MMF should be on a stable dose that is expected to remain stable throughout the trial and was started at least 3 months prior to screening
- 7. Patients previously treated with pirfenidone or nintedanib
- 8. Patients treated with N-acetyl-cysteine (NAC) for fibrotic lung disease, at any time within the 4 weeks of the screening period
- 9. Drug treatment for any type of pulmonary hypertension (e.g. sildenafil, endothelin receptor antagonist [ERA], etc.)
- Participation in a trial of an investigational medical product within the last 4 weeks
- 11. Significant co-existent emphysema (extent greater than extent of fibrosis on HRCT within the last 12 months)

Pirfenidone — F. Hoffmann-La Roche Ltd
- 12. Significant other organ co-morbidity including hepatic or renal impairment
- 13. Previous intolerance or allergy to the trial treatment
- 14. Pregnant patients, or women of child-bearing potential, not using a reliable contraceptive method
- 15. Unable to provide informed written consent
- 16. Predicted life expectancy <12 months or on an active transplant waiting list
- 17. Use of any tobacco product in the 12 weeks prior to the start of screening, or any unwillingness to abstain from their use through to the Follow-up Visit
- 18. Illicit drug or alcohol abuse within 12 months prior to screening, according to the investigator's judgment
- 19. Planned major surgery during the trial
- 20. Hypersensitivity to the active substance or to any of the excipients of pirfenidone
- 21. History of angioedema
- 22. Concomitant use of fluvoxamine
- 23. Clinical evidence of any active infection which according to the investigator's judgment may interfere with trial conduct, measurement of pulmonary function, or impact the course of the ILD
- 24. Any history of hepatic impairment, elevation of transaminase enzymes, or the confirmation of any of the following liver function test (LFT) criteria above the specified limits:
  - a. Total bilirubin above the upper limit of normal (ULN)
  - b. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)  $> 1.5 \times ULN$
  - c. Alkaline phosphatase >2.0 × ULN.
- 25. Creatinine clearance <30 mL/min, calculated using the Cockcroft-Gault formula
- 26. Any serious medical condition, clinically significant abnormality on an ECG at screening, or laboratory test results (hematology, serum chemistry, and urinalysis) that, in the opinion of the investigator, may pose an additional risk to the patient following the administration of trial treatment
- 27. An ECG with a heart rate corrected QT interval (corrected using Fridericia's formula [QTcF]) ≥500 ms at screening, or a family or personal history of long QT syndrome.

Re-screening may be considered for patients who do not show sufficient disease deterioration in accordance to the protocol at the time of the initial screening. Rescreening is permitted if there is strong evidence of clinical worsening based on the Investigator's judgement and only upon receipt of official approval from the Study Management Team. In such cases, re-screening may be performed after a minimum of 4-weeks lapse from the initial screening date.

#### **End of Trial and Length of Trial**

After completion of the double-blind treatment period and the Follow-up Visit at Week 28, the Sponsor will offer the possibility to the patients to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. The end of the clinical trial is defined as the date when the last patient, last visit (LPLV) occurs or the date at which the last data point which is required for the statistical analysis is received, whichever is the later date. For this trial, LPLV will occur when the

Pirfenidone — F. Hoffmann-La Roche Ltd

last patient has completed the final safety Follow-up Visit, 28 days after the final open-label dose, or when the last data point is collected in the safety follow-period.

For each patient the total length of the trial is expected to be up to a maximum of 91 weeks. The trial duration includes the washout period of up to 4 weeks, the screening period of up to 3 weeks, the double-blind treatment period of 24 weeks, the follow-up period of 4 weeks, the open-label safety follow-up period up to 12 months (52 weeks) and a final safety Follow-up Visit 4 weeks after the last dose.

#### **Investigational Medicinal Products**

#### Pirfenidone and Placebo

Pirfenidone and placebo will be supplied by the Sponsor as 267 mg capsules in a bottle. For information on the formulation and handling of pirfenidone, see the Investigator's Brochure or local prescribing information for pirfenidone.

Placebo will be supplied by the Sponsor in the form of capsules with identical appearance and size as the pirfenidone capsule. The placebo capsules will contain microcrystalline cellulose.

#### **Statistical Methods**

#### **Primary Analysis**

The primary efficacy objective for this trial is to evaluate the efficacy of pirfenidone vs. placebo on lung function parameters on the basis of rate of decline in FVC in mL measured by handheld spirometry over the 24-week double-blind treatment period.

The primary analysis will be based on the intent-to-treat (ITT) population. Patients who discontinue treatment prematurely will be analyzed based on the available data. No imputation method will be applied.

The primary analysis of the primary endpoint will compare the mean FVC decline in each treatment arm using a student's t-test with a two-sided significance level  $\alpha$ =0.05. The mean FVC decline for each treatment arm will be calculated using the estimated FVC decline for each individual patient. The individual FVC decline will be estimated by applying a linear regression model to all data points collected during the 24-week double-blind treatment period.

#### **Determination of Sample Size**

The purpose of this trial is hypothesis generation regarding the efficacy of pirfenidone vs. placebo on lung function parameters on the basis of rate of decline in FVC, as measured by daily handheld spirometry.

A total sample size of approximately 250 patients is planned, and patients will be randomized in a 1:1 ratio. The randomization will be stratified by concomitant MMF treatment (yes/no), the presence/absence of IPAF as defined by the MDT.

Pirfenidone — F. Hoffmann-La Roche Ltd

The planned sample size is based on the statistical hypothesis of the primary endpoint and assumes 80% power and a two-sided significance level of 5% using a student's ttest. It is assumed, after inspection of historical data, that FVC decline in the placebo arm is 85 mL with a common standard deviation of 70 mL, which can be reduced to 60 mL with a common standard deviation of 70 mL in the pirfenidone arm. In this scenario, 125 patients per treatment arm are needed to detect this treatment effect with 80% power.

#### **Interim Analyses**

There are no planned interim efficacy analyses for this trial. Safety interim analyses will be performed at least three times during the trial, at approximately 6, 12, and 18 months after the start of recruitment.

Pirfenidone — F. Hoffmann-La Roche Ltd

# Appendix 2 Schedule of Assessments

| | Washout <sup>a</sup> | Screening | Double-blind treatment | | | | | | | Early treatment discontinuation <sup>b</sup> | Follow-<br>up <sup>u</sup> | Additional<br>safety<br>follow-up <sup>c</sup> | Additional<br>safety<br>follow-up<br>final visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day<br>Week | –50 to –22 | -21 to -1 | Randomization<br>1 | | 56<br>8 | 84<br>12 | 112<br>16 | 140<br>20 | 168<br>24 | | 196<br>28 | up to 12<br>months | up to 12<br>months<br>plus 28<br>days |
| Window (days,<br>unless otherwise<br>stated) | | | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 b | ±5 | ±5 | ±5 |
| Treatment Period<br>Visit | | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | | | Month 1 to 6:<br>Monthly visits<br>Month 7 to12:<br>Approximately<br>every<br>3 months | |
| Informed consent d,e | Х | х | | | | | | | | | | | |
| Review Eligibility<br>Criteria | | х | | | | | | | | | | | |
| Demographic data <sup>e</sup> | х | х | | | | | | | | | | | |
| General medical history and baseline conditions <sup>e</sup> | х | х | | | | | | | | | | | |

Pirfenidone — F. Hoffmann-La Roche Ltd

| | Washout <sup>a</sup> | Screening | Double-blind treatment | | | | | | | Early treatment discontinuation <sup>b</sup> | Follow-<br>up <sup>u</sup> | Additional<br>safety<br>follow-up <sup>c</sup> | Additional<br>safety<br>follow-up<br>final visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day<br>Week | –50 to –22 | -21 to -1 | Randomization<br>1 | 28<br>4 | 56<br>8 | 84<br>12 | 112<br>16 | 140<br>20 | 168<br>24 | | 196<br>28 | up to 12<br>months | up to 12<br>months<br>plus 28<br>days |
| Window (days,<br>unless otherwise<br>stated) | | | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 b | ±5 | ±5 | ±5 |
| Treatment Period<br>Visit | | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | | | Month 1 to 6:<br>Monthly visits<br>Month 7 to12:<br>Approximately<br>every<br>3 months | |
| Vital signs <sup>f</sup> | | х | х | Х | Х | Х | Х | Х | Х | х | Х | Х | |
| Weight | | х | | | | | | | Х | х | | | |
| Height | | х | | | | | | | | | | | |
| Complete physical examination <sup>9</sup> | | х | x | | | | | | х | х | | | |
| ECG h | | х | Х | | | Х | | | Х | х | Х | | |
| Hematology <sup>i</sup> | | х | Х | | | х | | | Х | х | | | |
| Chemistry <sup>j</sup> | | Х | Х | Х | x <sup>k</sup> | Х | x <sup>k</sup> | x <sup>k</sup> | Х | х | | x <sup>k</sup> | _ |
| Pregnancy test | | х | Х | Х | Х | х | Х | х | Х | х | | Х | |

Pirfenidone — F. Hoffmann-La Roche Ltd

| | Washout <sup>a</sup> | Screening | Double-blind treatment | | | | | | | Early treatment discontinuation <sup>b</sup> | Follow-<br>up <sup>u</sup> | Additional<br>safety<br>follow-up <sup>c</sup> | Additional<br>safety<br>follow-up<br>final visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day<br>Week | –50 to –22 | -21 to -1 | Randomization<br>1 | 28<br>4 | 56<br>8 | 84<br>12 | 112<br>16 | 140<br>20 | 168<br>24 | | 196<br>28 | up to 12<br>months | up to 12<br>months<br>plus 28<br>days |
| Window (days,<br>unless otherwise<br>stated) | | | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 b | ±5 | ±5 | ±5 |
| Treatment Period<br>Visit | | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | | | Month 1 to 6:<br>Monthly visits<br>Month 7 to12:<br>Approximately<br>every<br>3 months | |
| Trial treatment administration | | | х | х | Х | х | Х | х | | | x <sup>m</sup> | х | |
| Spirometry (FVC, FEV <sub>1</sub> ) | | х | х | х | Х | х | Х | х | х | х | | | |
| Daily spirometry (handheld device) <sup>n,o</sup> | | х | х | х | х | х | х | х | х | х | | | |
| DLco | | Х | х | | | х | | | Х | х | | | |
| 6MWD <sup>p</sup> | | х | Х | | | х | | | х | х | | | |
| Leicester Cough<br>Questionnaire <sup>q</sup> | | | х | | | х | | | х | х | | | |

Pirfenidone — F. Hoffmann-La Roche Ltd

| | Washout <sup>a</sup> | Screening | Double-blind treatment | | | | | | Early treatment discontinuation b | Follow-<br>up <sup>u</sup> | Additional<br>safety<br>follow-up <sup>c</sup> | Additional<br>safety<br>follow-up<br>final visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day<br>Week | -50 to -22 | -21 to -1 | Randomization<br>1 | 28<br>4 | 56<br>8 | 84<br>12 | 112<br>16 | 140<br>20 | 168<br>24 | | 196<br>28 | up to 12<br>months | up to 12<br>months<br>plus 28<br>days |
| Window (days,<br>unless otherwise<br>stated) | | | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 b | ±5 | ±5 | ±5 |
| Treatment Period<br>Visit | | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | | | Month 1 to 6:<br>Monthly visits<br>Month 7 to12:<br>Approximately<br>every<br>3 months | |
| UCSD-SOBQ q | | | х | | | х | | | Х | х | | | |
| SGRQ <sup>q</sup> | | | х | | | Х | | | Х | х | | | |
| Cough visual analog score <sup>q</sup> | | | х | | | х | | | x | Х | | | |
| Serum for biomarker assessments | | | х | х | | х | | | х | х | | | |
| Plasma for biomarker assessments | | | х | х | | х | | | х | х | | | |

Pirfenidone — F. Hoffmann-La Roche Ltd

| | Washout <sup>a</sup> | Screening | | | | | | | Early treatment discontinuation <sup>b</sup> | Follow-<br>up <sup>u</sup> | Additional<br>safety<br>follow-up <sup>c</sup> | Additional<br>safety<br>follow-up<br>final visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day<br>Week | –50 to –22 | -21 to -1 | Randomization<br>1 | 28<br>4 | 56<br>8 | 84<br>12 | 112<br>16 | 140<br>20 | 168<br>24 | | 196<br>28 | up to 12<br>months | up to 12<br>months<br>plus 28<br>days |
| Window (days,<br>unless otherwise<br>stated) | | | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 b | ±5 | ±5 | ±5 |
| Treatment Period<br>Visit | | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | | | Month 1 to 6:<br>Monthly visits<br>Month 7 to12:<br>Approximately<br>every<br>3 months | |
| Whole blood for PAX gene biomarker assessment | | | х | х | | х | | | х | х | | | |
| Concomitant medications <sup>r</sup> | х | х | х | х | х | х | х | х | х | х | х | Х | х |
| Adverse events s | | х | Х | х | Х | х | х | х | х | х | х | Х | Х |
| Whole blood sample for RBR (optional) <sup>t</sup> | | | х | | | | | | | | | | |

Pirfenidone — F. Hoffmann-La Roche Ltd

6MWD=6-minute walk distance; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; DLco=diffusing capacity of the lung for carbon monoxide; ECG=electrocardiogram; eCRF=electronic case report form; FEV<sub>1</sub>=forced expiratory volume in 1 second; FVC=forced vital capacity; IMP=investigational medicinal product; LDH=lactate dehydrogenase; LFT=liver function test; PRO=patient-reported outcome; RBC=red blood cell; RBR=Research Biosample Repository; SGRQ=St. George's Respiratory Questionnaire; SOBQ=Shortness of Breath Questionnaire; UCSD=University of California, San Diego; WBC=white blood cell

Notes: all assessments should be performed within 7 days of the scheduled visit, unless otherwise specified.

- <sup>a</sup> Patients will be required to taper and/or discontinue all prohibited medications in the 28 days prior to the start of screening during the washout period. Patients not taking a prohibited medication will forgo the washout period and directly enter screening.
- Patients who discontinue trial treatment prematurely will return to the site (clinic) for an Early Treatment Discontinuation Visit 28 (± 5) days after the last dose of the double-blind treatment, thus ending their participation in the trial. For patients who end their participation in the double-blind treatment period due to unblinding, they may be offered to continue into the open-label period according to the investigator's judgment. These patients will attend the Early Treatment Discontinuation Visit (28 (± 5) days after the last dose of the double-blind treatment) and on the same day begin their participation in the 12-month open-label pirfenidone safety follow-up period.
- <sup>c</sup> After completion of the double-blind treatment period and the Follow-up Visit at Week 28, the Sponsor will offer the possibility to the patients to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. During the 12-month safety follow-up period, initially, patients will be evaluated at monthly visits for the first 6 months. At the end of the first 6 months, patients will be evaluated at each site visit occurring approximately every 3 months until the end of the safety follow-up period.. A final Follow-up Visit will be performed at the end of the safety period, 28 (± 5) days after the last open-label dose.
- <sup>d</sup> Informed consent must be documented before any trial-specific screening procedure is performed, and may be obtained either at the Washout or Screening Visits.
- <sup>e</sup> Any procedures that were not completed during washout, must be completed at the Screening Visit.
- Includes respiratory rate, pulse rate, and systolic and diastolic blood pressures while the patient is in a seated position, and temperature.

  Abnormalities observed at baseline should be recorded on the General Medical History and Baseline Conditions eCRF. At subsequent visits, new or worsened clinically significant abnormalities should be recorded on the Adverse Event eCRF. All vital sign measurements are to be obtained prior to any blood draws scheduled at the same time.

Pirfenidone — F. Hoffmann-La Roche Ltd

- Includes evaluation of the head, eyes, ears, nose, and throat, and the cardiovascular, dermatological, musculoskeletal, respiratory, gastrointestinal, genitourinary, and neurological systems. Abnormalities observed at baseline should be recorded on the General Medical History and Baseline Conditions eCRF. At subsequent visits, new or worsened clinically significant abnormalities should be recorded on the Adverse Event eCRF.
- <sup>h</sup> All ECGs are to be obtained prior to other procedures scheduled at the same time.
- <sup>i</sup> Hematology includes WBC count, RBC count, hemoglobin, hematocrit, platelet count, differential count (neutrophils, eosinophils, basophils, monocytes, lymphocytes, other cells).
- <sup>1</sup> Chemistry panel (serum or plasma) includes sodium, potassium, chloride, bicarbonate, glucose, BUN or urea, creatinine, total protein, albumin, phosphorus, calcium, total and direct bilirubin, alkaline phosphatase, ALT, AST, uric acid, LDH.
- <sup>k</sup> Only LFTs (AST, ALT, bilirubin, and alkaline phosphatase) will be conducted at these visits. During the Safety Follow-up period, LFTs will be performed every month during the first 6 months and subsequently at each visit occurring approximately every 3 months thereafter, until the end of this period.
- All women of childbearing potential will have a serum pregnancy test at screening. Urine pregnancy tests will be performed at the specified subsequent visits. If a urine pregnancy test is positive, it must be confirmed by a serum pregnancy test. During the Safety Follow-up period, urine pregnancy tests will be performed every month during the first 6 months at each site visit. Urine pregnancy tests will continue to be performed on a monthly basis during the remainder of the Safety Follow-up period with patients performing the test at home (using kits provided by the site) during months where there is no site visit and at each site visit occurring approximately every 3 months. Patients will be instructed to contact the site immediately in case the result of the home pregnancy test is positive. In such cases, the patient must visit the site for a confirmatory serum pregnancy test.
- <sup>m</sup> Open-label treatment with pirfenidone will be started at this visit, if the patient requests continued treatment with pirfenidone.
- <sup>n</sup> Handheld spirometry will be conducted by the patient every day in a seated position.
- <sup>o</sup> To provide handling evaluations and quality assurance for the daily spirometer assessments, nursing visits to the patient's home (or at another suitable location) will occur at least three times during the trial, namely between Weeks 1 and 4, between Weeks 8 and 12, and between Weeks 16 and 20. Additional home nursing visits may be conducted according to the investigator's judgment.

Pirfenidone — F. Hoffmann-La Roche Ltd

- <sup>p</sup> 6-Minute Walk Distance (6MWD) is used to evaluate the functional capacity of patients with lung disease.
- <sup>q</sup> Questionnaires will be self-administered prior to the patient receiving any information on disease status and prior to the performance of non-PRO assessments.
- Includes any medication (e.g., prescription drugs, over-the-counter drugs, vaccines, herbal or homeopathic remedies, nutritional supplements) used by a patient from the washout period until 28 days after the last dose of trial treatment.
- After informed consent has been obtained but prior to initiation of trial treatment, only serious adverse events caused by a protocol-mandated intervention should be reported. After initiation of trial treatment, all adverse events will be reported until 28 days after the last dose of trial treatment. After this period, all deaths, regardless of cause, should be reported. In addition, the Sponsor should be notified if the investigator becomes aware of any serious adverse event that is believed to be related to prior trial treatment. The investigator should follow each adverse event until the event has resolved to baseline grade or better, the event is assessed as stable by the investigator, the patient is lost to follow-up, or the patient withdraws consent. Every effort should be made to follow all serious adverse events considered to be related to trial treatment or trial-related procedures until a final outcome can be reported.
- <sup>t</sup> Not applicable for a site that has not been granted approval for RBR sampling.
- <sup>u</sup> If a patient discontinues the trial between weeks 24 and 28, final assessments according to the Follow-up visit for week 28 should be performed.

a.

Pirfenidone — F. Hoffmann-La Roche Ltd

# Appendix 3 Patient Reported Outcome Questionnaire

### **Leicester Cough Questionnaire**

| time 2. In the last 2 weeks, have you been bothered by phlegm production when you cough? 1 | stion<br>stly as |
|---|---|
| 1 All of the time Most of the time A lot of the time Some of the time A little of the time time 2. In the last 2 weeks, have you been bothered by phlegm production when you cough? 1 2 3 4 5 6 7 Every time Most times Several times Sometimes Oocasionally Rarely Never 3. In the last 2 weeks, have you been timed because of your cough? 1 1 2 3 4 6 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Most of the time A lot of the time Some of the time A lot of the time Most of the time A lot of the time Some of the time A little of the time Most of the time A lot of the time Some of the time A little of the time Most of the time A lot of the time Some of the time A little of the time Most of the time A lot of the time A lot of the time A lot of the time A lot of the time Some of the time A little of the time Most of the time A lot of the time Some of the time A little of the time | |
| 2. In the last 2 weeks, have you been bothered by phlegm production when you cough? 1 2 3 4 5 6 7 Every time Most times Several times Sometimes Occasionally Rarely Never 3. In the last 2 weeks, have you been tired because of your cough? 1 2 3 4 5 6 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time time between time December of the time A lot of the time A lot of the time A lot of the time between time December of time A lot of the time A lot of the time A lot of the time between time December of the time December of the time A lot of the time A little of the time A little of the time A lot of the time A lot of the time A lot of the time A little of the time A little of the time A lot of the time A lot of the time A lot of the time A little of the time A little of the time A lot | |
| 2. In the last 2 weeks, have you been bothered by phlegm production when you cough? 1 | of the tim |
| Every time Most times Several times Sometimes Occasionally Rarely Never In the last 2 weeks, have you been tired because of your cough? All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time All of the time Most of the time A lot of the time Some of the time A lot of the time All of the tim | |
| Every time Most times Several times Sometimes Occasionally Rarely Never 1. In the last 2 weeks, have you been tired because of your cough? 1. All of the time Most of the time A lot of the time Some of the time A little of the time Imme 4. In the last 2 weeks, have you felt in control of your cough? 1. All of the time Hardly any of the A little of the time Some of the time A lot of the time Imme 5. How often during the last 2 weeks have you felt embarrassed by your coughing? 1. All of the time Most of the time A lot of the time Some of the time A little of the time Imme 6. In the last 2 weeks, my cough has made me feel anxious 1. 2. 3. 4. Some of the time A little of the time Imme 7. In the last 2 weeks, my cough has interfered with my job, or other daily tasks 1. 2. 3. 4. Some of the time A little of the time Imme 8. In the last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 1. 2. 3. 4. Some of the time A little of the time Imme 8. In the last 2 weeks, exposure to paints or fumes has made me cough 1. 2. 3. 4. Some of the time A little of the time Imme 9. In the last 2 weeks, exposure to paints or fumes has made me cough 1. 2. 3. 4. Some of the time A little of the time Imme 1. 4. Some of the time A little of the time Imme 1. 5. Some of the time A little of the time Imme 1. 6. The last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 2. 3. 4. Some of the time A little of the time Imme 8. In the last 2 weeks, exposure to paints or fumes has made me cough 1. 2. 3. 4. Some of the time A little of the time Imme 1. 4. Some of the time A little of the time Imme 1. 5. Some of the time A little of the time Imme 1. 6. The day any of the Imme 1. 7. All of the time Most of the time A lot of the time Some of the time A little of the time Imme 1. 8. In the last 2 weeks, exposure to paints or fumes has made me cough 1. 2. 3. 4. Some of the time A little of the time Imme 1. 6. The day any of the Imme 1. 7. All of the time Most of the ti | |
| 3. In the last 2 weeks, have you been tired because of your cough? 1 | |
| All of the time Most of the time A lot of the time A lot of the time A lot of the time A little of the time Hardly any of the time Most of the time A little of the time Hardly any of the time A little of the time A little of the time Most of the time A little of the time A little of the time A little of the time A little of the time Most of the time A little of the time A lot of the time A little of the time A little of the time A lot of the time A lot of the time A little of the time A lot of the time A lot of the time A little of the time A lot of the time A lot of the time A little of the time A little of the time A lot of the time A lot of the time A little of the time A little of the time A lot of the time A lot of the time A lot of the time A lot of the time A lot of the time A little of the time A little of the time A lot of the time A lot of the time A lot of the time A lot of the time A little of th | ٢ |
| All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 4. In the last 2 weeks, have you felt in control of your cough? 1 2 3 4 5 6 7 None of the time Wost of the time A little of the time Some of the time A lot of the time Hardly any of the time Hardly any of the time A lot of the time A lot of the time A lot of the time Hardly any of the time A lot of the time A | |
| 4. In the last 2 weeks, have you felt in control of your cough? 1 2 3 4 5 6 7 None of the time Hardly any of the time All of the time Most of the time All of the time Al | |
| None of the time Hardly any of the hardly any of the time Hardly any | of the tim |
| None of the time Hardly any of the A little of the time Some of the time A lot of the time Most of the time All of time 5. How often during the last 2 weeks have you felt embarrassed by your coughing? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time time 5. In the last 2 weeks, my cough has made me feel anxious 1 2 3 4 5 6 7 Hardly any of the time None time 6. In the last 2 weeks, my cough has interfered with my job, or other daily tasks 1 2 3 4 5 6 7 Hardly any of the time None time 7. In the last 2 weeks, my cough has interfered with my job, or other daily tasks 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time time 8. In the last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 1 2 3 4 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time time 9. In the last 2 weeks, exposure to paints or fumes has made me cough 1 2 3 4 6 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 6 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 6 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Sometimes during Sometimes during the day | |
| time 5. How often during the last 2 weeks have you felt embarrassed by your coughing? 1 | |
| All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 5. In the last 2 weeks, my cough has made me feel anxious 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 7. In the last 2 weeks, my cough has interfered with my job, or other daily tasks 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 3. In the last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 3. In the last 2 weeks, exposure to paints or fumes has made me cough 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 3. In the last 2 weeks, exposure to paints or fumes has made me cough 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Several times during Sometimes during the day 12. In the last 2 weeks, my cough has made me feel frustrated | the time |
| All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 5. In the last 2 weeks, my cough has made me feel anxious 1 | |
| time 5. In the last 2 weeks, my cough has made me feel anxious 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time time 7. In the last 2 weeks, my cough has interfered with my job, or other daily tasks 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time time 3. In the last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 3. In the last 2 weeks, exposure to paints or fumes has made me cough 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 3. In the last 2 weeks, exposure to paints or fumes has made me cough 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Sometimes during Occasionally through Rarely the day the day the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | |
| All of the time Most of the time A lot of the time Some of the time A little of the time time 7. In the last 2 weeks, my cough has interfered with my job, or other daily tasks 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 8. In the last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 4 1 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 7 8 8 7 8 8 7 8 9 8 9 9 9 9 9 9 9 9 9 9 9 9 9 9 9 9 | of the tin |
| All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time To the last 2 weeks, my cough has interfered with my job, or other daily tasks 1 | |
| time 7. In the last 2 weeks, my cough has interfered with my job, or other daily tasks 1 | |
| All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 3. In the last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 3. In the last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 3. In the last 2 weeks, exposure to paints or fumes has made me cough 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Several times during Sometimes during Occasionally through Rarely the day the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | of the tim |
| All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 3. In the last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 9. In the last 2 weeks, exposure to paints or fumes has made me cough 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Several times during Sometimes during Occasionally through Rarely the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | |
| In the last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 9. In the last 2 weeks, exposure to paints or fumes has made me cough 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Several times during Sometimes during Occasionally through Rarely the day the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | |
| All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 1 | of the tin |
| All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 9. In the last 2 weeks, exposure to paints or fumes has made me cough 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Several times during Sometimes during the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | |
| itime In the last 2 weeks, exposure to paints or fumes has made me cough I 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time IO.In the last 2 weeks, has your cough disturbed your sleep? I 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time II.In the last 2 weeks, how many times a day have you had coughing fits? I 2 3 4 5 6 7 All of the time Most times a day have you had coughing fits? I 2 3 4 5 6 7 All of the time Most times during Several times during Sometimes during the day the day the day II. In the last 2 weeks, my cough has made me feel frustrated | |
| 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Sometimes during Gondinuously) 1 2 3 4 5 6 7 All of the time Most times during Several times during Sometimes during the day the day 1 2 10 Cocasionally through Rarely the day 1 None (continuously) | of the tim |
| All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Sometimes during Sometimes during Occasionally through Rarely (continuously) the day the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | |
| time 10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Sometimes during Sometimes during Occasionally through Rarely (continuously) the day the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | |
| 1 All of the time Most of the time A lot of the time Some of the time A little of the time Hardly any of the time 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Sometimes during Sometimes during Occasionally through Rarely (continuously) the day the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | of the tin |
| time 1 I.In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time Most times during Several times during Sometimes during Occasionally through Rarely (continuously) the day the day the day I.In the last 2 weeks, my cough has made me feel frustrated | |
| time 1 11. In the last 2 weeks, how many times a day have you had coughing fits? 1 2 3 4 5 6 7 All of the time (continuously) the day the day the day the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | |
| 1 2 3 4 5 6 7 All of the time (continuously) the day the day the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | of the tin |
| 1 2 3 4 5 6 7 All of the time (continuously) the day the day the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | |
| (continuously) the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | |
| (continuously) the day the day the day 12. In the last 2 weeks, my cough has made me feel frustrated | |
| | of the tin |

Pirfenidone — F. Hoffmann-La Roche Ltd

| | | | | | time | |
|---|---|---|---|---|---|---|
| 3.In the last 2 wee | ks, my cough has | s made me feel fed | up | | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the time |
| 14.In the last 2 wee | ks, have you suff | ered from a hoarse | e voice as a resul | t of your cough? | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the time |
| 5.In the last 2 wee | ks, have you had | a lot of energy? | | | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| None of the time | Hardly any of the<br>time | A little of the time | Some of the time | A lot of the time | Most of the time | All of the time |
| 16. In the last 2 wee | ks, have you wor | ried that your coug | h may indicate a | serious illness? | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the time |
| 17.In the last 2 wee<br>cough? | eks, have you bee | n concerned that o | ther people think | something is wro | ng with you becar | use of your |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| All of the time | Most of the time | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the time |
| 18.In the last 2 wee | ks, my cough has | s interrupted conve | ersations or teleph | hone calls | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Every time | Most times | A lot of the time | Some of the time | A little of the time | Hardly any of the<br>time | None of the time |
| 19.In the last 2 wee | ks. I feel that my | cough has annoye | d my partner, fan | nily or friends | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | Most times when | Several times when | | | Rarely | Never |
| Every time I cough | I cough | I cough | I cough | I cough | | |

#### **Scoring**

The Leicester Cough Questionnaire is a patient-reported questionnaire evaluating the impact of cough on quality of life. The questionnaire comprises 19 items and takes 5 to 10 minutes to complete. Each item assesses symptoms, or the impact of symptoms, over the last 2 weeks on a seven-point Likert scale. Scores in three domains (physical, psychological and social) are calculated as a mean for each domain (range 1 to 7). A total score (range 3 to 21) is also calculated by adding the domain scores together. Higher scores indicate better quality of life.

The scores from each of the following questions are added together to provide the mean score for each domain:

1. Physical: 1, 2, 3, 9, 10, 11, 14, 15

2. Psychological: 4, 5, 6, 12, 13, 16, 17

3. Social: 7, 8, 18, 19

Domain scores: total score from items in domain/number of items in domain (range 1–7).

Total scores: addition of domain scores (range 3–21).

Pirfenidone — F. Hoffmann-La Roche Ltd

#### UCSD-SOBQ

The University of California, San Diego-Shortness of Breath Questionnaire (UCSD-SOBQ) is a symptom-specific, 24-item, patient-self-administered questionnaire that assesses shortness of breath while doing a variety of activities of daily living.

# UCSD MEDICAL CENTER PULMONARY REHABILITATION PROGRAM

#### SHORTNESS-OF-BREATH QUESTIONNAIRE

© 1995 The Regents of the University of California

Please rate the breathlessness you experience when you do, or if you were to do, each of the following tasks. **Do not skip any items.** If you've never performed a task, or no longer perform it, give your best estimate of the breathlessness you would experience while doing that activity. Please review the two sample questions below before turning the page to begin the questionnaire.

Pirfenidone — F. Hoffmann-La Roche Ltd

When I do, or if I were to do, the following tasks, I would rate my breathlessness as:

- None at all
  None at all
  Severe
  Maximum or unable to do because of breathlessness

Harry has felt moderately short of breath during the past 7 days while brushing his teeth and so circles a three for this activity.

| 2. | Mowing the lawn | .0 | 1 | 2 | 3 | 4 | (5) | ) |
|----|-----------------|----|---|---|---|---|-----|---|
|----|-----------------|----|---|---|---|---|-----|---|

Anne has never mowed the lawn before but estimates that she would have been too breathless to do this activity during the past 7 days. She circles a five for this activity.

# When I do, or if I were to do, the following tasks, I would rate my breathlessness as:

0 None at all

2

3

- 4 Severe
- 5 Maximum or unable to do because of breathlessness

| 1. | At rest0 | 1 | 2 | 3 | 4 | 5 |
|----|-----------------------------------------|---|---|---|---|---|
| 2. | Walking on a level at my own pace 0 | 1 | 2 | 3 | 4 | 5 |
| 3. | Walking on a level with others my age 0 | 1 | 2 | 3 | 4 | 5 |
| 4. | Walking up a hill0 | 1 | 2 | 3 | 4 | 5 |
| 5. | Walking up stairs | 1 | 2 | 3 | 4 | 5 |
| 6. | While eating 0 | 1 | 2 | 3 | 4 | 5 |
| 7. | Standing up from a chair | 1 | 2 | 3 | 4 | 5 |
| 8. | Brushing my teeth | 1 | 2 | 3 | 4 | 5 |
| 9. | Shaving and/or brushing my hair0 | 1 | 2 | 3 | 4 | 5 |

Pirfenidone — F. Hoffmann-La Roche Ltd

| 10. | Showering/bathing 0 | 1 | 2 | 3 | 4 | 5 |
|-----|---------------------|---|---|---|---|---|
|-----|---------------------|---|---|---|---|---|

When I do, or if I were to do, the following tasks, I would rate my breathlessness as:

0 None at all
1
2
3
4 Severe
5 Maximum or unable to do because of breathlessness

| 11. Dressing 0 | 1 | 2 | 3 | 4 | 5 |
|-----------------------------------------------|---|---|---|---|---|
| 12. Picking things up and tidying up a room 0 | 1 | 2 | 3 | 4 | 5 |
| 13. Doing the dishes | 1 | 2 | 3 | 4 | 5 |
| 14. Sweeping/vacuuming0 | 1 | 2 | 3 | 4 | 5 |
| 15. Making the bed | 1 | 2 | 3 | 4 | 5 |
| 16. Shopping 0 | 1 | 2 | 3 | 4 | 5 |
| 17. Doing laundry 0 | 1 | 2 | 3 | 4 | 5 |
| 18. Washing the car | 1 | 2 | 3 | 4 | 5 |
| 19. Mowing the lawn 0 | 1 | 2 | 3 | 4 | 5 |
| 20. Watering the lawn | 1 | 2 | 3 | 4 | 5 |
| 21. Sexual activities | 1 | 2 | 3 | 4 | 5 |

Pirfenidone — F. Hoffmann-La Roche Ltd

0 None at all

1

2

- 4 Severe
- 5 Maximum or unable to do because of breathlessness

#### How much do the following limit you in your daily life?

| 22. | Shortness of breath | 0 | 1 | 2 | 3 | 4 | 5 |
|-----|------------------------------------------|----|---|---|---|---|---|
| 23. | Fear of "hurting myself" by overexertion | .0 | 1 | 2 | 3 | 4 | 5 |
| 24. | Fear of shortness of breath | .0 | 1 | 2 | 3 | 4 | 5 |

#### **Scoring**

Twenty one items assess the severity of shortness of breath during specific activities associated with daily living if patients do not routinely perform the activity, they are asked to estimate the degree of shortness of breath anticipated. Three additional items ask about limitations due to: shortness of breath, fear of harm from overexertion and fear of shortness of breath.

Each of the 24 activities are rated on how dyspnea affects the activity on a 6-point scale: 0 = None at all to 5 = Maximal or unable to do because of breathlessness

The scores from all 24 questions are totalled to provide a score in the range 0 - 120.

Pirfenidone — F. Hoffmann-La Roche Ltd

#### **SGRQ**

The St. George's Respiratory Questionnaire (SGRQ) is an index designed to measure and quantify health-related health status in patients with chronic airflow limitations.

### ST. GEORGE'S RESPIRATORY QUESTIONNAIRE ENGLISH FOR THE UNITED STATES

#### ST. GEORGE'S RESPIRATORY QUESTIONNAIRE (SGRQ)

This questionnaire is designed to help us learn much more about how your breathing is troubling you and how it affects your life. We are using it to find out which aspests of your illness cause you the most problems, rather than what the doctors and nurses think your problems are.

Please read the instructions carefully and ask if you do not understand anything.

Do not spend too long deciding about your answers.

| Before completing the rest of the questionnaire: | | | | | |
|---|---|---|---|---|---|
| Please sheek one box to show how you describe<br>your current health: | Very good | Good | Fair | Poor | Very poor |

Copyright reserved P.W. Jones, PhD FRCP Professor of Respiratory Medicine, St. George's University of London, Jenner Wing, Crammer Terrace, London SW17 ORE, UK.

USA / English version «Past three months» version Tel. +44 (0) 20 9725 5371 Fax +44 (0) 20 8725 5955

continued...

Pirfenidone — F. Hoffmann-La Roche Ltd

### St. George's Respiratory Questionnaire PART 1

| Please describe how often your respiratory problems have affected you over the past 3 months. | | | | | | |
|---|---|---|---|---|---|---|
| estion: | x for each qu | (√) one bo | se check | Plea | | |
| not<br>at<br>all | only with<br>respiratory<br>infections | a few<br>days<br>a month | several<br>days<br>a week | almost<br>every<br>day | | |
| | | | | | . Over the past 3 months, I have coughed: | 1. |
| | | | | | <ul> <li>Over the past 3 months, I have brought up<br/>phiegm (sputum):</li> </ul> | 2. |
| | | | | | <ul> <li>Over the past 3 months, I have had shortness<br/>of breath;</li> </ul> | 3. |
| | | | | | <ul> <li>Over the past 3 months, I have had wheezing attacks:</li> </ul> | 4. |
| | | | ered from | you suffe | How many times during the past 3 months have<br>severe or very unpleasant respiratory attacks? | 5. |
| one: | _ ` ' | | more | | | |
| | | 3 time | more | | | |
| | s 🗆 | 2 time | | | | |
| | e 🗆 | 1 tim | | | | |
| | e 🗌 | e of the tim | none | | | |
| | | | | attack) | . How long did the worst respiratory attack last?<br>(Go to Question 7 if you did not have a severe a | 6. |
| one: | _ ` ' | | | | | |
| | _ = | | | | | |
| | | 1 or 2 day | | | | |
| | y 🗆 | s than a da | les | | | |
| | | | d days | many goo | Over the past 3 months, in a typical week, how<br>(with few respiratory problems) have you had? | 7. |
| one: | _ ` ' | | | | | |
| | _ | 4 good day | | | | |
| | d 🗆 | ay was goo | ly every da | near | | |
| | d 🗆 | ay was goo | every da | | | |
| | | | ? | e morning | . If you wheeze, is it worse when you get up in th | 8. |
| me: | e check (🗸) | | | | | |
| on | e check (*) e check (*) e check (*) f c check (*) | than 3 time 3 time 2 time 1 tim e of the tim Pleasek or more r more day 1 or 2 day s than a da Pleas o good day 2 good day 4 good day ay was goo ay was goo | none a w 3 o less od days Ni 1 or: 3 or- dy every da | many goo | How long did the worst respiratory attacks? How long did the worst respiratory attack last? (Go to Question 7 if you did not have a severe a Over the past 3 months, in a typical week, how (with few respiratory problems) have you had? | 6. |

Pirfenidone — F. Hoffmann-La Roche Ltd

## St. George's Respiratory Questionnaire PART 2

| Section 1 | | | |
|---|---|---|---|
| How would you describe your respiratory condition | 1? | | |
| | | Please | check (🗸) one: |
| The mo | st impor | tant problem I have | |
| Cause | s me qui | te a lot of problems | |
| | Causes | me a few problems | |
| | C | auses no problems | |
| If you have ever held a job: | | | |
| | | Please | check (✔) one: |
| My respiratory problems made | me stop | working altogether | |
| My respiratory problems interfere with my job | or made | me change my job | |
| My respiratory pr | oblems | do not affect my job | |
| Section 2 | | | |
| These are questions about what activities usually ma | ake you | ieei snort or breau | triese days. |
| | | ment please check | |
| (- | | x that applies | |
| | _ | hese days: | |
| | True | False | |
| 5101 | | | |
| Sitting or lying still | | H | |
| Washing or dressing yourself | | | |
| Washing or dressing yourself<br>Walking around the house | | | |
| Washing or dressing yourself | | | |
| Washing or dressing yourself<br>Walking around the house | | | |
| Washing or dressing yourself<br>Walking around the house<br>Walking outside on level ground | | | |

### St. George's Respiratory Questionnaire

| PART 2 | | | | |
|---|---|---|---|---|
| Section 3 | | | | |
| These are more questions about your cough and sh | ortness | of breath <u>th</u> | ese day | <u>s</u> . |
| Fore | ach state | ment please | check | |
| | | x that appli | | |
| | _ | hese days: | | |
| Coughing hurts | True | False | | |
| Coughing makes me fired | H | H | | |
| Lam short of breath when I tak | H | H | | |
| I am short of breath when I bend over | H | H | | |
| My coughing or breathing disturbs my sleep | Ħ | $\overline{\Box}$ | | |
| I get exhausted easily | H | | | |
| i get exhausted easily | _ | | | |
| Section 4 | | | | |
| The second secon | | | | |
| These are questions about other effects that your redays. | espirator | y problems | may ha | re on you <u>the</u> |
| _ | | _ | | |
| | | | | ment, please<br>e box that |
| | | | | these days: |
| | | | True | False |
| My cough or breathing is emb | arrassing | in public | Ш | Ц |
| My respiratory problems are a nuisance to my family, fr | iends or r | eighbors | | |
| I get afraid or panic when I cann | ot catch n | ny breath | | |
| I feel that I am not in control of my re | spiratory | problems | $\perp$ | Ц |
| I do not expect my respiratory problem | s to get a | ny better | Ш | Ц |
| I have become frail or an invalid because of my re | spiratory | problems | Ш | |
| Exercise | is not sa | fe for me | | |
| Everything seems to | much of | an effort | Ш | |
| Section 5 | | | | |
| These are questions about your respiratory treatme section 6. | nt. If you | are not re | ceiving | treatment go i |
| Fo | r each sta | stement, ple | ase | |
| che | | box that ap | plies | |
| | True | hese days:<br>False | | |
| My treatment does not help me very much | | raise | | |
| | H | | | |
| I get embarrassed using my medication in public | | | | |
| have unpleasant side effects from my medication | | | | |
| My treatment interferes with my life a lot | | | | |
| SA / US English version 4 | | | | |

Pirfenidone — F. Hoffmann-La Roche Ltd

Statistical Analysis Plan MA39189, Version 2.0, 29-Oct-2018

continued...

#### St. George's Respiratory Questionnaire PART 2

| Section 6 | | | | |
|---|---|---|---|---|
| These are questions about how your activities might | be affected | by your | espirator | y problem |
| | tř | ne box tha | t apples t<br>respirator | y problem |
| I take a long time to ge | | | True | False |
| I cannot take a bath or shower, or I tak | | | H | H |
| walk slower than other people my | • | | | $\equiv$ |
| Jobs such as household chores take a long time, or | | | | |
| If I walk up one flight of stairs, I have | | • | | |
| If I hurry or walk fast, I have | | | | |
| My breathing makes it difficult to do things such as walk<br>up stairs, light gardening such | | , dance, | | |
| My breathing makes it difficult to do things such a<br>dig in the garden or shovel snow, jog or walk briskl | | | | |
| My breathing makes it difficult to do things<br>manual work, ride a<br>or pla | | | | |
| Section 7 We would like to know how your respiratory problem | is usually al | Tect your | daily life | |
| The would like to know how your respiratory problem | io doddiry di | reor your | duny inc. | |
| the box the | tatement, ple<br>at applies to<br>respiratory p | you becau | se of | |
| | True | False | | |
| I cannot play sports or do other physical activities | | $\vdash$ | | |
| I cannot go out for entertainment or recreation | | H | | |
| I cannot go out for entertainment or recreation<br>eannot go out of the house to do the shopping | | | | |
| I cannot go out for entertainment or recreation | | | | |

Pirfenidone — F. Hoffmann-La Roche Ltd

#### St. George's Respiratory Questionnaire

| | a list of other activities that your respiratory problems may prevent you from doing. (You have to check these, they are just to remind you of ways your shortness of breath may you): |
|---|---|
| G | oing for walks or walking the dog |
| Do | oing activities or chores at home or in the garden |
| Se | exual intercourse |
| G | oing to a place of worship, or a place of entertainment |
| G | oing out in bad weather or into smoky rooms |
| Vis | siting family or friends or playing with children |
| | ease write in any other important activities that your respiratory problems may stop you from |
| | ow please check the box (one only) that you think best describes how your respiratory problems fect you: |
| | It does not stop me from doing anything I would like to do |
| | It stops me from doing one or two things I would like to do |
| | It stops me from doing most of the things I would like to do |
| | It stops me from doing everything I would like to do |
| | you for completing this questionnaire. Before you finish would you please make sure that you have<br>ed all the questions. |

#### STRUCTURE OF SGRQ

The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction.

**Part 1 (Questions 1-8)** addresses the frequency of respiratory symptoms. It is not designed to be a precise epidemiological tool, but to assess the patient's perception of their recent respiratory problems.

Part 2 (Sections 9-16) addresses the patient's current state (i.e. how they are these days).

The Activity score measures disturbances to daily physical activity. The Impacts score covers a range of disturbances of psycho-social function. Validation studies for the original SGRQ showed that this component relates in part to respiratory symptoms, but it also correlates quite

Pirfenidone — F. Hoffmann-La Roche Ltd

strongly with exercise performance (6-minute walk test), breathlessness in daily life (MRC breathlessness score) and disturbances of mood (anxiety and depression). The Impacts score is, therefore, the broadest component of the questionnaires, covering the whole range of disturbances that respiratory patients experience in their lives.

Three component scores are calculated for the SGRQ

**Symptoms** – concerned with the effect of respiratory symptoms their frequency and severity

Activity concerned with activities that cause or are limited by breathlessness

**Impacts** covers a range of aspects concerned with social functioning and psychological disturbances resulting from airway disease.

**Total score** summaries the impact of disease on overall health status. Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status.

#### SGRQ SCORES IN HEALTHY SUBJECTS

Means (95% confidence intervals) for SGRQ scores in normal subjects with no history of respiratory disease

| N | Age-years | FEV1 as<br>%<br>predicted | Symptoms score | Activity score | Impacts<br>Score | Total<br>Score |
|---|---|---|---|---|---|---|
| 72 | 46 (17 - 80) | 95 (91-<br>99) | 12 (9-15) | 9 (7-12) | 2 (1-3) | 6 (5-7) |

Pirfenidone — F. Hoffmann-La Roche Ltd

#### **Scoring**

Questions 1-7 The eCRF screens should be set up so that where a patient has ticked a box, a value of 1 is entered for the appropriate question. By default, the empty boxes are entered as 0. Where a patient has missed a question the cells on the spreadsheet are left blank. Example: Response = 1c, 'Over the last year I have coughed a few days a month'. A value of 1 is entered for 1c and a value of 0 is entered for 1a, 1b, 1d and 1e. If no tick was present for question 1 then 1a to 1e would be left blank.

Question 8 Where a patient has ticked 'Yes' to having a worse wheeze in the morning, a value of 1 is entered for the appropriate question. All other responses are entered as 0. Example: Do you have a wheeze? = 'Yes' and Worse in the morning = 'Yes'. then response to question 8 = 1. Do you have a wheeze? = 'Yes' and Worse in the morning = 'No'. Or, Do you have a wheeze? = 'No'. then response to question 8=0.

Questions 9, 10 & 17 Where a patient has ticked a box, a value of 1 is entered for the appropriate question. The empty boxes are entered as 0. Where a patient has missed the question the cells on the spreadsheet are left blank. Example: Response = 10a, 'My chest trouble made me stop work'. A value of 1 is entered for 10a and a value of 0 is entered for 10b and 10c. If no tick was present for question 10, then 10a to 10c would be left blank.

Questions 11 - 16 Where a patient has ticked 'True' a value of 1 is entered for the appropriate question and where a patient has ticked 'False' a value of 0 is entered. Where a patient has missed a question the cell on the spreadsheet is left blank.

Example: 15a = 'True' then 15a = 1.

14c = 'False' then 14c = 0.

13h = missing then 13h is left blank

In response to question 14, if a patient is not receiving medication, enter the responses as zero, otherwise the calculator will read the values as missing.

Missing Questions

There should not be any missing items in the questionnaire, but the SGRQ can have up to 24% of missing items in the questionnaire. If more than 24% of items are missing the scores will be missing.

Pirfenidone — F. Hoffmann-La Roche Ltd

#### ITEM WEIGHTS

Once the questions have been answered the following weights are applied to the individual responses

#### PART 1

Over the past 3 months, I have coughed:

| Most<br>days/week | Several days/<br>week | A few days a month | Only with chest infections | Not at all |
|---|---|---|---|---|
| 80.6 | 63.2 | 29.3 | 28.1 | 0.0 |

Over the past 3 months, I have brought up phlegm (sputum):

| Most<br>days/week | Several days/<br>week | A few days a month | Only with chest infections | Not at all |
|---|---|---|---|---|
| 76.8 | 60.0 | 34.0 | 30.2 | 0.0 |

3) Over the past 3 months, I have had shortness of breath:

| Most<br>days/week | Several days/<br>week | A few days a month | Only with chest infections | Not at all |
|---|---|---|---|---|
| 87.2 | 71.4 | 43.7 | 35.7 | 0.0 |

4) Over the past 3 months, I have had attacks of wheezing:

| Most<br>days/week | Several days/<br>week | A few days a month | Only with chest infections | Not at all |
|---|---|---|---|---|
| 86.2 | 71.40 | 45.6 | 36.4 | 0.0 |

Pirfenidone — F. Hoffmann-La Roche Ltd

5) During the past 3 months, how many severe or very bad unpleasant attacks of chest trouble have you had?

| More than three | 3 attacks | 2 attacks | 1 attack | None |
|-----------------|-----------|-----------|----------|------|
| 86.7 | 73.5 | 60.3 | 44.2 | 0.0 |

6) How long did the worst attack of chest trouble last?

| a week or more | 3 or more days | 1 or 2 days | Less than a day | None |
|----------------|----------------|-------------|-----------------|------|
| 89.7 | 73.5 | 58.8 | 41.9 | 0.0 |

Pirfenidone — F. Hoffmann-La Roche Ltd

7) Over the past 3 months, in an average week, how many good days (with little chest trouble) have you had?

| No good days | 1 or 2 good<br>days | 3 or 4 good<br>days | Nearly every day | Every day |
|---|---|---|---|---|
| 93.3 | 76.6 | 61.5 | 15.4 | 0.0 |

8) If you have a wheeze, is it worse in the morning?

| No | Yes |
|-----|------|
| 0.0 | 62.0 |

#### PART 2

The weights in Part 2 are also applied to the individual responses to each question. The worse the impact the higher the weight. This means that weights are not applied sequentially in the order that the response is given.

9) How would you describe your chest condition?

| The most important problem I have | 83 .2 |
|-----------------------------------|-------|
| Causes me quite a lot of problems | 82.5 |
| Causes me a few problems | 34.6 |
| Causes no problem | 0.0 |

10) If you have ever had paid employment?

My chest trouble made me stop work 88.9

Pirfenidone — F. Hoffmann-La Roche Ltd

| My chest trouble interferes with my work or made me change my work | 77.6 |
|-----------------------------------------------------------------------|------|
| My chest trouble does not affect my work | 0.0 |
| 11) Questions about what activities usually make you feel breathless. | |
| Sitting or lying still | 90.6 |
| Getting washed or dressed | 82.8 |
| Walking around the home | 80.2 |
| Walking outside on the level | 81.4 |
| Walking up a flight of stairs | 76.1 |
| Walking up hills | 75.1 |
| Playing sports or games | 72.1 |

| 12) | More | questions | about | your | cough | and | breathlessness |
|-----|------|-----------|-------|------|-------|-----|----------------|

| My cough hurts | 81.1 |
|-----------------------------------------------------------------------|------|
| My cough makes me tired | 79.1 |
| I get breathless when I talk | 84.5 |
| I get breathless when I bend over | 76.8 |
| My cough or breathing disturbs my sleep | 87.9 |
| I get exhausted easily | 84.0 |
| 13) Questions about other effects your chest trouble may have on you. | |
| My cough or breathing is embarrassing in public | 74.1 |
| My chest trouble is a nuisance to my family, friends or neighbours | 79.1 |
| I get afraid or panic when I cannot get my breath | 87.7 |
| I feel that I am not in control of my chest problem | 90.1 |
| I do not expect my chest to get any better | 82.3 |
| I have become frail or an invalid because of my chest | 89.9 |
| Exercise is not safe for me | 75.7 |
| Everything seems too much of an effort | 84.5 |
| 14) Questions about your medication. | |
| My medication does not help me very much | 88.2 |
| Pirfenidone — F. Hoffmann-La Roche Ltd | |
| Statistical Analysis Plan MA39189, Version 2.0, 29-Oct-2018 | |

| | I get embarrassed using my medication in public | 53.9 |
|---|---|---|
| | I have unpleasant side effects from my medication | 81.1 |
| | My medication interferes with my life a lot | 70.3 |
| 15) | Questions about how activities may be affected by your breathing. | |
| | I take a long time to get washed or dressed | 74.2 |
| | I cannot take a bath or shower, or I take a long time | 81.0 |
| | I walk more slowly than other people, or I stop for rests | 71.7 |
| | Jobs such as housework take a long time, or I have to stop for rests | 70.6 |
| | If I walk up one flight of stairs, I have to go slowly or stop | 71.6 |
| | If I hurry or walk fast, I have to stop or slow down | 72.3 |
| | My breathing makes it difficult to do things such as walk up hills, carry things up stairs, light gardening such as weeding, dance, play bowls or play golf | 74.5 |
| | My breathing makes it difficult to do things such as carry heavy loads, dig the garden or shovel snow, jog or walk at 5 miles per hour, play tennis or swim | 71.4 |
| | My breathing makes it difficult to do things such as very heavy manual work, run, cycle, swim fast or play competitive sports | 63.5 |

Pirfenidone — F. Hoffmann-La Roche Ltd

16) We would like to know how your chest trouble usually affects your daily life.

| I cannot play sports or games | 64.8 |
|-------------------------------------------------|------|
| I cannot go out for entertainment or recreation | 79.8 |
| I cannot go out of the house to do the shopping | 81.0 |
| I cannot do housework | 79.1 |
| I cannot move far from my bed or chair | 94.0 |

17) Tick the statement which you think best describes how your chest affects you.

| It does not stop me doing anything I would like to do | 0.0 |
|---------------------------------------------------------|------|
| It stops me doing one or two things I would like to do | 42.0 |
| It stops me doing most of the things I would like to do | 84.2 |
| It stops me doing everything I would like to do | 96.7 |

#### SCORING ALGORITHM

Three component scores are calculated: Symptoms; Activity; Impacts

One **Total** score is also calculated.

#### PRINCIPLE OF CALCULATION

Each questionnaire response has a unique empirically derived 'weight'. The lowest possible weight is zero and the highest is 100.

Pirfenidone — F. Hoffmann-La Roche Ltd

Each component of the questionnaire is scored separately in three steps:

i. The weights for all items with a positive response are summed.

ii The weights for missed items are deducted from the maximum possible weight for

each component. The weights for all missed items are deducted from the maximum

possible weight for the Total score.

iii. The score is calculated by dividing the summed weights by the adjusted maximum

possible weight for that component and expressing the result as a percentage :

Score = 100 x Summed weights from positive items in that component

Sum of weights for all items in that component

The Total score is calculated in similar way:

Score =  $100 \times \text{Summed}$  weights from positive items in the questionnaire

Sum of weights for all items in the questionnaire

Sum of maximum possible weights for each component and Total:

Symptoms 662.5

Activity 1209.1

Impacts 2117.8

Total 3989.4

(Note: these are the maximum possible weights that could be obtained for the worst possible state of the patient).

Pirfenidone — F. Hoffmann-La Roche Ltd

It will be noted that the questionnaire requests a single response to questions 1-7, 9-10 and 17. If multiple responses are given to one of these questions then averaging the weights for the positive responses for that question are acceptable

#### SYMPTOMS COMPONENT

This is calculated from the summed weights for the positive responses to questions 1-8.

#### **ACTIVITY COMPONENT**

This is calculated from the summed weights for the positive responses to questions 11 and 15.

#### **IMPACTS COMPONENT**

This is calculated from the summed weights for the positive responses to questions 9-10, 12-14 and 16-17.

#### **TOTAL SCORE**

The Total score is calculated by summing all positive responses in the questionnaire and expressing the result as a percentage of the total weight for the questionnaire

#### HANDLING MISSED ITEMS

There should not be any missed items but if there are missing items the scores should be calculated using the following rules:

following should be used: The following method is recommended for missing items:

#### **Symptoms**

Pirfenidone — F. Hoffmann-La Roche Ltd

| The Symptoms component will tolerate a maximum of 2 missed items. The weight for the misse item is subtracted from the total possible weight for the Symptoms component (662.5) and from the Total weight (3989.4). | ed<br> |
|---|---|
| Pirfenidone — F. Hoffmann-La Roche Ltd | |
| Statistical Analysis Plan MA39189, Version 2.0, 29-Oct-2018 | |
| 8 | 6 |

#### **Activity**

The Activity component will tolerate a maximum of 4 missed items. The weight for the

missed item is subtracted from the total possible weight for the Activity component (1209.1) and from the Total weight (3989.4).

#### **Impacts**

The Impacts component will tolerate a maximum of 6 missed items. The weight for the missed item is subtracted from the total possible weight for the Impacts component (2117.8) and from the Total weight (3989.4).

This visual analogue scale is designed to help us learn about the severity of your cough. This scale is 100mm (10cm) in length.

During the last week, how do you rate the severity of your cough; 0mm representing no cough and 100mm representing the worst cough ever? Please indicate the severity of your cough by placing an **X** on the line.

#### **Cough Visual Analogue Scale (VAS)**

During the last week, how do you rate the severity of your cough; 0 mm representing no cough and 100 mm representing the worst cough ever? Please indicate the severity of your cough by placing an  $\mathbf{X}$  on the line.

### Worst Cough ever (100mm)



Pirfenidone — F. Hoffmann-La Roche Ltd